Replication of Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes (CANVAS Trial)

NCT03936010

May 27, 2021

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes (CANVAS trial)

#### 1.2 <u>Intended aim(s)</u>

To compare canagliflozin to placebo on cardiovascular (CV) events including CV death, heart attack, and stroke in patients with type 2 diabetes mellitus (T2DM), whose diabetes is not well controlled at the beginning of the study and who have a history of CV events or have a high risk for CV events.

#### 1.3 Primary endpoint for replication and RCT finding

Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial Infarction (MI), and Nonfatal Stroke

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

With 688 cardiovascular safety events recorded across the trials, there would be at least 90% power, at an alpha level of 0.05, to exclude an upper margin of the 95% confidence interval for the hazard ratio of 1.3.

### 1.5 Primary trial estimate targeted for replication

HR = 0.86 (95% CI 0.75–0.97) comparing canagliflozin to placebo (Neal et al., 2017)

### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

### 3. Data Source(s)

United/Optum, MarketScan, Medicare

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

### **Design Diagram – CANVAS TRIAL REPLICATION**



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing canagliflozin to the DPP-4 inhibitor (DPP4i) antidiabetic class. DPP4is serve as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The comparison against DPP4 inhibitors is the **primary comparison**. Initiators of 2nd generation sulfonylureas are used as a secondary comparator group. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of canagliflozin or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.

#### 5.2 Important steps for cohort formation

#### 5.2.1 Eligible cohort entry dates

Market availability of canagliflozin in the U.S. started on March 29, 2013.

- For Marketscan and Medicare: April 1, 2013-Dec 31, 2017 (end of data availability).
- For Optum: April 1, 2013-March 31, 2019 (end of data availability).

### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

For canagliflozin vs. DPP4i

| | Optum | | Mark | Marketscan M | | icare* |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 74,864,884 | | 191,990,035 | | 23,466,175 |

| Patients who used exposure or a reference between April 1, 2013 to Dec 2017 (for Marketscan/Medicare)/March 2019 (for Optum) | -74,192,962 | 671,922 | -<br>191,172,811 | 817,224 | -21,718,863 | 1,747,312 |
|---|---|---|---|---|---|---|
| Patients who have continuous 6 months registration in the database | -89,308 | 582,614 | -69,496 | 747,728 | -466,595 | 1,280,717 |
| Patients without prior use of reference | -339,732 | 242,882 | -464,089 | 283,639 | -810,370 | 470,347 |
| Patients without prior use of exposure | -75,001 | 167,881 | -89,428 | 194,211 | -71,119 | 399,228 |
| Excluded because patient qualified in >1 exposure category | -236 | 167,645 | -312 | 193,899 | -301 | 398,927 |
| Excluded based on Age | -7 | 167,638 | 0 | 193,899 | 0 | 398,927 |
| Excluded based on Gender | -8 | 167,630 | 0 | 193,899 | 0 | 398,927 |
| Excluded based on Inclusion 1- DM Type 2 with ICD-10 | -5,385 | 162,245 | -9,472 | 184,427 | -4,090 | 394,837 |
| Excluded based on Inclusion 2- History or high risk of cardiovascular disease (with 180 day lookback) | -25,130 | 137,115 | -39,753 | 144,674 | -20,833 | 374,004 |
| Excluded based on Inclusion 3- Include all males OR Female postmenopausal- >45 years of age OR use of contraceptives | -7 | 137,108 | -9 | 144,665 | 0 | 374,004 |
| Excluded based on Exclusion 1- DM Type I + Secondary DM + Diabetic ketoacidosis with ICD10 CODES | -4,572 | 132,536 | -3,939 | 140,726 | -16,980 | 357,024 |
| Excluded based on Exclusion 4- History of one or more severe hypoglycemic episode- Severe hypoglycemia (Inpatient, primary) | -109 | 132,427 | -47 | 140,679 | -472 | 356,552 |
| Excluded based on Exclusion 5- Glucose-galactose malabsorption/Primary Renal glucosuria | -37 | 132,390 | -30 | 140,649 | -173 | 356,379 |
| Excluded based on Exclusion #7- Renal disease that requires treatment with immunosuppresive therapy | -1,512 | 130,878 | -662 | 139,987 | -6,367 | 350,012 |
| Excluded based on Exclusion 8- MI, unstable angina, revascularization procedure, or cerebrovascular accident within 3 months | -2,345 | 128,533 | -1,604 | 138,383 | -8,548 | 341,464 |
| Excluded based on Exclusion 9- Cardiac conduction disorder(inpatient)/Other cardiac dysrhythmia (inpatient) | -167 | 128,366 | -71 | 138,312 | -517 | 340,947 |
| Excluded based on Exclusion 10- Liver disease | -2,303 | 126,063 | -1,695 | 136,617 | -6,089 | 334,858 |
| Excluded based on Exclusion 11- Any history of or planned bariatric surgery (prior 5 years) | -22 | 126,041 | -95 | 136,522 | -12 | 334,846 |
| Excluded based on Exclusion 14- History of Malignant Neoplasm (prior 5 years) | -4,554 | 121,487 | -3,985 | 132,537 | -19,311 | 315,535 |
| Excluded based on Exclusion 15- HIV/AIDS (dx and meds) -prior 5 years | -64 | 121,423 | -56 | 132,481 | -127 | 315,408 |
| Excluded based on Exclusion 16- Hematological disorder | -1,540 | 119,883 | -1,633 | 130,848 | -7,624 | 307,784 |
| Excluded based on Exclusion 17- CCI (180 days) >=10 | -177 | 119,706 | -50 | 130,798 | -696 | 307,088 |
| · | | | | | | |

| Excluded based on Exclusion 18 - Major Surgery (90 days prior) | -191 | 119,515 | -212 | 130,586 | -674 | 306,414 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion 20- Use of SGLT2i (prior 6 months) | -833 | 118,682 | -892 | 129,694 | -817 | 305,597 |
| Excluded based on Exclusion 22- use of a corticosteroid medication or immunosuppressive agent | -3,235 | 115,447 | -3,085 | 126,609 | -8,985 | 296,612 |
| Excluded based on Exclusion 23- Use of cana in prior 3 months (although this is already applied as part of cohort creation) | 0 | 115,447 | 0 | 126,609 | 0 | 296,612 |
| Excluded based on Exclusion 24- Alcohol or Drug abuse (prior 3 years) and Exclusion 25- Pregnancy | -972 | 114,475 | -532 | 126,077 | -1,766 | 294,846 |
| Final cohort | | 114,475 | | 126,077 | | 294,846 |

<sup>\*</sup> Medicare database includes only patients with at least one diagnosis for diabetes, heart failure, or cerebrovascular disease.

For canagliflozin vs. 2<sup>nd</sup> generation SUs

| | Optum | | Mark | etscan | Med | dicare* |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 74,864,884 | | 191,990,035 | | 23,466,175 |
| Patients who used exposure or a reference between April 1, 2013 to Dec 2017 (for Marketscan/Medicare)/March 2019 (for Optum) | -<br>73,662,096 | 1,202,788 | -<br>190,768,942 | 1,221,093 | -<br>20,351,733 | 3,114,442 |
| Patients who have continuous 6 months registration in the database | -165,247 | 1,037,541 | -115,162 | 1,105,931 | -861,454 | 2,252,988 |
| Patients without prior use of reference | -710,706 | 326,835 | -759,153 | 346,778 | -1,627,827 | 625,161 |
| Patients without prior use of exposure | -70,933 | 255,902 | -88,833 | 257,945 | -68,783 | 556,378 |
| Excluded because patient qualified in >1 exposure category | -168 | 255,734 | -149 | 257,796 | -118 | 556,260 |
| Excluded based on Age | -10 | 255,724 | 0 | 257,796 | 0 | 556,260 |
| Excluded based on Gender | -17 | 255,707 | 0 | 257,796 | 0 | 556,260 |
| Excluded based on Inclusion 1- DM Type 2 with ICD-10 | -14,479 | 241,228 | -23,583 | 234,213 | -8,608 | 547,652 |
| Excluded based on Inclusion 2- History or high risk of cardiovascular disease (with 180 day lookback) | -38,807 | 202,421 | -54,172 | 180,041 | -30,020 | 517,632 |
| Excluded based on Inclusion 3- Include all males OR Female postmenopausal- >45 years of age OR use of contraceptives | -21 | 202,400 | -36 | 180,005 | 0 | 517,632 |

<sup>\*\*</sup>Exclusion 24 and 25 collapsed to adhere to CMS cell suppression guidelines.

| Excluded based on Exclusion 1- DM Type I + Secondary DM + Diabetic ketoacidosis with ICD10 CODES | -5,426 | 196,974 | -4,290 | 175,715 | -19,804 | 497,828 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion 4- History of one or more severe hypoglycemic episode- Severe hypoglycemia (Inpatient, primary) | -76 | 196,898 | -37 | 175,678 | -332 | 497,496 |
| Excluded based on Exclusion 5- Glucose-galactose malabsorption/Primary Renal glucosuria | -53 | 196,845 | -55 | 175,623 | -221 | 497,275 |
| Excluded based on Exclusion #7- Renal disease that requires treatment with immunosuppresive therapy | -2,276 | 194,569 | -976 | 174,647 | -9,763 | 487,512 |
| Excluded based on Exclusion 8- MI, unstable angina, revascularization procedure, or cerebrovascular accident within 3 months | -3,178 | 191,391 | -2,244 | 172,403 | -11,210 | 476,302 |
| Excluded based on Exclusion 9- Cardiac conduction disorder(inpatient)/Other cardiac dysrhythmia (inpatient) | -240 | 191,151 | -121 | 172,282 | -837 | 475,465 |
| Excluded based on Exclusion 10- Liver disease | -3,273 | 187,878 | -2,251 | 170,031 | -8,410 | 467,055 |
| Excluded based on Exclusion 11- Any history of or planned bariatric surgery (prior 5 years) | -27 | 187,851 | -109 | 169,922 | -16 | 467,039 |
| Excluded based on Exclusion 14- History of Malignant Neoplasm (prior 5 years) | -6,172 | 181,679 | -5,306 | 164,616 | -25,472 | 441,567 |
| Excluded based on Exclusion 15- HIV/AIDS (dx and meds) -prior 5 years | -112 | 181,567 | -72 | 164,544 | -198 | 441,369 |
| Excluded based on Exclusion 16- Hematological disorder | -1,925 | 179,642 | -1,989 | 162,555 | -9,438 | 431,931 |
| Excluded based on Exclusion 17- CCI (180 days) >=10 | -287 | 179,355 | -50 | 162,505 | -993 | 430,938 |
| Excluded based on Exclusion 18 - Major Surgery (90 days prior) | -317 | 179,038 | -291 | 162,214 | -856 | 430,082 |
| Excluded based on Exclusion 20- Use of SGLT2i (prior 6 months) | -904 | 178,134 | -984 | 161,230 | -874 | 429,208 |
| Excluded based on Exclusion 22- use of a corticosteroid medication or immunosuppressive agent | -4,334 | 173,800 | -3,909 | 157,321 | -10,920 | 418,288 |
| Excluded based on Exclusion 23- Use of cana in prior 3 months (although this is already applied as part of cohort creation) | 0 | 173,800 | 0 | 157,321 | 0 | 418,288 |
| Excluded based on Exclusion 24- Alcohol or Drug abuse (prior 3 years) and Exclusion 25- Pregnancy | -1566 | 172,234 | -777 | 156,544 | -2,592 | 415,696 |
| Final cohort | | 172,234 | | 156,544 | | 415,696 |

<sup>\*</sup> Medicare database includes only patients with at least one diagnosis for diabetes, heart failure, or cerebrovascular disease.

### 6. Variables

# 6.1 Exposure-related variables:

<sup>\*\*</sup> Exclusion 24 and 25 collapsed to adhere to CMS cell suppression guidelines.

#### Study drug:

The study exposure of interest is initiation of canagliflozin. Initiation will be defined by no use of any SGLT-2 inhibitor or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents:

- Initiators of canagliflozin will be compared to initiators of
  - o DPP4i (primary)
  - o 2nd generation sulfonylureas

Because canagliflozin and comparators are frequently used as second or third line treatments of T2DM, we expect it to be unlikely that canagliflozin and comparators are initiated in patients with substantially different baseline risk for proposed outcomes.

#### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B). These covariates are based on those used by Patorno et al. (2019).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- Secondary outcomes: Individual components:
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - o Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases
    - Information on CV mortality through data linkage with the National Death Index (NDI) will only become available at a later date for Medicare and will be used in secondary analyses.

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

- 1. Diabetes Ketoacidosis (we expect to see a positive association; Neal et al., 2017)
- 2. Heart failure (we expect to see a protective effect; Neal et al., 2017)

#### **Control outcome definitions**

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| Diabetic Ketoacidosis | Inpatient ICD-9 diagnosis: 250.1x | Note- The corresponding ICD-10 codes will also be used |
| Heart Failure | Inpatient ICD-9 diagnosis (primary diagnosis): 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 | Note- The corresponding ICD-10 codes will also be used |

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of canagliflozin and comparator and will continue until the earliest date of the following events:

• The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,

- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (canagliflozin and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator or any other agent in the comparator class and vice versa (e.g. switching from saxagliptin to linagliptin would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - An added treatment that is not part of the exposure or comparator group does not fulfill this criterion (e.g. if a canagliflozin user adds insulin, he or she does not get censored at the time of insulin augmentation)

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

## 7. Initial Feasibility Analysis

#### Aetion report name:

For canagliflozin vs. DPP4i

Optum- <a href="https://bwh-dope.aetion.com/#/projects/details/660/results/26056/result/0">https://bwh-dope.aetion.com/#/projects/details/660/results/26056/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/#/projects/details/661/results/26055/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/26057/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/26055/result/0">https://bwh-dope.aetion.com/#/projects/details/662/results/26055/result/0</a>

For canagliflozin vs. 2<sup>nd</sup> generation SUs

Optum- <a href="https://bwh-dope.aetion.com/#/projects/details/660/results/26064/result/0">https://bwh-dope.aetion.com/#/projects/details/660/results/26064/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/26066/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/26065/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/26066/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/26065/result/0</a>

#### Date conducted: 09/30/2018

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report name:

• For canagliflozin vs. DPP4i

Optum- <a href="https://bwh-dope.aetion.com/#/projects/details/660/results/26064/result/0">https://bwh-dope.aetion.com/#/projects/details/660/results/26064/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/26066/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/26066/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/26066/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/26066/result/0</a>

• For canagliflozin vs. 2<sup>nd</sup> generation Sus

Optum- https://bwh-dope.aetion.com/#/projects/details/660/results/26067/result/0 Marketscan- https://bwh-dope.aetion.com/#/projects/details/661/results/26068/result/0 Medicare- https://bwh-dope.aetion.com/#/projects/details/662/results/26069/result/0

Date conducted: 09/30/2018

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica M. Franklin | Date reviewed: | 10/26/18 |
|-------------------------|---------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/11/18 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment after PS matching

#### Aetion report name:

### For canagliflozin vs. DPP4i

- o Optum- https://bwh-dope.aetion.com/projects/details/660/results/44837/result/0
- o Marketscan- https://bwh-dope.aetion.com/projects/details/661/results/44838/result/0
- o Medicare- https://bwh-dope.aetion.com/projects/details/662/results/44839/result/0

## For canagliflozin vs. 2nd generation SUs

- o Optum- https://bwh-dope.aetion.com/projects/details/660/results/44834/result/0
- o Marketscan- https://bwh-dope.aetion.com/projects/details/661/results/44835/result/0
- o Medicare- https://bwh-dope.aetion.com/projects/details/662/results/44836/result/0

#### Date conducted: 11/18/2019

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to **Appendix B**.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

o For canagliflozin vs. DPP4i

| <u> </u> | | | |
|---|---|---|---|
| | Overall | Referent | Exposure |
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 589 (0.39%) | 374 (0.49%) | 215 (0.28%) |
| Start of an additional exposure | 6,913 (4.54%) | 2,413 (3.17%) | 4,500 (5.91%) |
| End of index exposure | 98,215 (64.53%) | 47,931 (62.98%) | 50,284 (66.08%) |
| Specified date reached | 22,353 (14.69%) | 12,162 (15.98%) | 10,191 (13.39%) |
| End of patient enrollment | 19,170 (12.60%) | 9,407 (12.36%) | 9,763 (12.83%) |
| Switch to other DPP4i (for censoring) + nursing home admission | 4,962 (3.26%) | 3,814 (5.01%) | 1,148 (1.51%) |

o For canagliflozin vs. 2nd generation SUs

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 548 (0.40%) | 364 (0.53%) | 184 (0.27%) |
| Start of an additional exposure | 6,001 (4.36%) | 1,842 (2.68%) | 4,159 (6.04%) |
| End of index exposure | 85,900 (62.38%) | 41,024 (59.58%) | 44,876 (65.18%) |
| Specified date reached | 22,281 (16.18%) | 12,957 (18.82%) | 9,324 (13.54%) |
| End of patient enrollment | 18,853 (13.69%) | 9,660 (14.03%) | 9,193 (13.35%) |
| Switch to other SUs (for censoring) + nursing home admission | 4,117 (2.99%) | 3,003 (4.36%) | 1,114 (1.62%) |

- Report follow-up time by treatment group.
  - o For canagliflozin vs. DPP4i

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Marketscan Medicare | | | |
| Overall Patient Population | 127 [58-306] | 149 [72-341] | 147 [81-318] |

| Referent | 121 [58-297] | 153 [87-327] | 153 [87-327] |
|----------|--------------|--------------|--------------|
| Exposure | 134 [58-318] | 142 [58-310] | 142 [58-310] |

#### o For canagliflozin vs. 2nd generation SUs

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group | Optum | Marketscan | Medicare |
| Overall Patient Population | 141 [63-336] | 159 [83-358] | 172 [90-373] |
| Referent | 140 [75-330] | 200 [118-414] | 200 [118-414] |
| Exposure | 141 [58-341] | 144 [62-327] | 144 [62-327] |

## • Report risk per 1,000 patients

#### Aetion report name:

## • For canagliflozin vs. DPP4i

Optum-<a href="https://bwh-dope.aetion.com/#/projects/details/660/results/34590/result/0">https://bwh-dope.aetion.com/#/projects/details/660/results/34590/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/34592/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/34591/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/34592/result/0">https://bwh-dope.aetion.com/#/projects/details/662/results/34592/result/0</a>

## • For canagliflozin vs. 2<sup>nd</sup> generation SUs

Optum- <a href="https://bwh-dope.aetion.com/#/projects/details/660/results/34596/result/0">https://bwh-dope.aetion.com/#/projects/details/660/results/34596/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/#/projects/details/661/results/34597/result/0">https://bwh-dope.aetion.com/#/projects/details/661/results/34597/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/#/projects/details/662/results/34598/result/0">https://bwh-dope.aetion.com/#/projects/details/662/results/34598/result/0</a>

## <u>Date conducted:</u> 04/25/2019 For canagliflozin vs. DPP4i

 Optum
 Marketscan
 Medicare

 Risk per 1,000 patients
 7.58
 7.81
 22.56

## For canagliflozin vs. 2<sup>nd</sup> generation SUs

| | Optum | Marketscan | Medicare |
|-------------------------|-------|------------|----------|
| Risk per 1,000 patients | 9.71 | 9.39 | 27.67 |

#### 10. Final Power Assessment

Date conducted: 12/01/2019

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).

#### o For canagliflozin vs. DPP4i

#### Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 76,101 | Reference | 76,101 |
| Exposed | 76,101 | Exposed | 76,101 |
| Risk per 1,000 patients | 12.65 | Risk per 1,000 patients | 12.65 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1925.3553 | Number of events expected | 1925.3553 |
| Power | 0.911332398 | Power | 0.999926523 |

Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 19,532 | Reference | 19,532 |
| Exposed | 19,532 | Exposed | 19,532 |
| Risk per 1,000 patients | 7.58 | Risk per 1,000 patients | 7.58 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 296.10512 | Number of events expected | 296.10512 |
| Power | 0.254449294 | Power | 0.616911596 |

# Marketscan

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 23,168 | Reference | 23,168 |
| Exposed | 23,168 | Exposed | 23,168 |
| Risk per 1,000 patients | 7.58 | Risk per 1,000 patients | 7.58 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 351.22688 | Number of events expected | 351.22688 |
| Power | 0.292672624 | Power | 0.690943556 |

# Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 33,401 | Reference | 33,401 |
| Exposed | 33,401 | Exposed | 33,401 |
| Risk per 1,000 patients | 22.56 | Risk per 1,000 patients | 22.56 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1507.05312 | Number of events expected | 1507.05312 |
| Power | 0.833370249 | Power | 0.999133759 |

# o For canagliflozin vs. 2nd generation SUs

# Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 68,850 | Reference | 68,850 |
| Exposed | 68,850 | Exposed | 68,850 |
| Risk per 1,000 patients | 15.59 | Risk per 1,000 patients | 15.59 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 2146.743 | Number of events expected | 2146.743 |
| Power | 0.937493971 | Power | 0.999980899 |

## ■ <u>Optum</u>

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 16,740 | Reference | 16,740 |
| Exposed | 16,740 | Exposed | 16,740 |
| Risk per 1,000 patients | 9.71 | Risk per 1,000 patients | 9.71 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 325.0908 | Number of events expected | 325.0908 |
| Power | 0.274612159 | Power | 0.657366306 |

## ■ <u>Marketscan</u>

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 23,265 | Reference | 23,265 |
| Exposed | 23,265 | Exposed | 23,265 |
| Risk per 1,000 patients | 9.39 | Risk per 1,000 patients | 9.39 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 436.9167 | Number of events expected | 436.9167 |
| Power | 0.350813593 | Power | 0.782915462 |

## ■ <u>Medicare</u>

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 28,845 | Reference | 28,845 |
| Exposed | 28,845 | Exposed | 28,845 |
| Risk per 1,000 patients | 27.67 | Risk per 1,000 patients | 9.39 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1596.2823 | Number of events expected | 541.7091 |
| Power | 0.853826925 | Power | 0.86285876 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/9/19 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/20/19 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 12/20/19

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <a href="Google Form">Google Form</a>. This form also provides space for reviewers to list any concerns that they feel may

contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

#### Aetion report name:

Date conducted:

#### 13.1 For **primary analysis**:

• In the PS-matched cohort of <u>canagliflozin and DPP4i</u> initiators from Section 9, calculate the HR for each outcome for canagliflozin versus referent patients using a Cox proportional hazards model.

### 13.2 For secondary analyses:

- In the PS-matched cohort of <u>canagliflozin and 2<sup>nd</sup> generation SU</u> initiators from Section 9, calculate the HR for canagliflozin versus referent patients using a Cox proportional hazards model.
- In both pre-matched cohorts, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for canagliflozin versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

#### 14. Requested Results

### 14.1 Results from primary and secondary analyses:

Separately for each endpoint and each comparator group:

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |
| ••• | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 15. References

American Diabetes Association. 8. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018;41(Suppl 1):S73-S85. doi:10.2337/dc18-S008.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. **page** 177

Neal B, Perkovic V, Mahaffey KW, De Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR. Canagliflozin and cardiovascular and renal events in type 2 diabetes. New England Journal of Medicine. 2017; 377(7):644-57.

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019; in press. (https://www.ahajournals.org/doi/pdf/10.1161/CIRCULATIONAHA.118.039177)

Effectiveness research with Real World Data to support FDA's regulatory decision making

| # | CANVAS trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | Trial details- Secondary indication, 4a- unintended super | iority with label change | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/open?id=1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV | Criteria |
| | EXPOSURE vs. COMPARISON | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-9 to ICD-10 mapping: <a href="https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk.general-equivalence-mapping.html">https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk.general-equivalence-mapping.html</a> . | Adequate mapping in claims |
| | Canagliflozin vs. placebo | Canagliflozin vs. DPP4 inhibitors (primary comparison) or vs. 2nd generation sulfonylureas (secondary) | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | , | Poor mapping or cannot be measured in claims |
| | Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial Infarction (MI), and Nonfatal Stroke HR = <b>0.86 (95% CI 0.75–0.97)</b> | Measured 1 days after drug initiation in diagnosis position specified below and inpatient care setting: Inpatient mortality/MI/Stroke - For MI Any diagnosis position in inpatient care setting ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) For stroke Primary diagnosis position in inpatient care setting ICD-9 discharge diagnosis: ICD-9 discharge diagnosis: ICD-9 discharge diagnosis: ICD-9 discharge diagnosis: INTAGENERATION OF THE PROPRIET OF THE | For MI: →PPV 94% in Medicare claims data [Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Aworn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. American heart journal 2004;148/99-104.] →PPV 88.4% in commercially-insured population [Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacoepidemiology and Drug Safety 2010;19:596-603.] For stroke: PPV of 85% or higher for ischemic stroke PPV ranging from 80% to 93% for hemorrhagic stroke →[Andrade SE, Harrold LR, Tjia J, et al. Asystematic review of validated methods for identifying cerbrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiology and Drug Safety 2012;21 Suppl 1:100-28.] →[Tirschwell DL, Longstreth WT, ir. Validating administrative data in stroke research. Stroke, a journal of cerebral circulation 2002;33:2465-70.] →[Roumie CL, Mitche E, Gideon PS, Varsa-Leronoc, C-castelisague J, Griffin MR, Validation of ICD 9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Can't be measured in claims but not important for the analysis |
| | INCLUSION CRITERIA | | | |
| 1 | Man or woman with a diagnosis of type 2 diabetes with glycated hemoglobin level 27.0% to \$10.5% at screening and be either. | Patients with a diagnosis of <b>T2DM</b> (ICD-9 Dx code of 250.x0 or 250.x2) in the <b>180 days prior to drug</b> initiation in any diagnosis position and inpatient or outpatient care setting. | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCUATIONAHA118.039177 | |
| | o (1) not currently on antihyperglycemic agent (AHA) therapy or | | · | 1 |
| | o (2) on AHA monotherapy or combination therapy with any approved class of agents: e.g., sulfonylurea, metformin, peroxisome proliferator-activated receptor gamma (PPARy) agonist, ajpha-glucosidase inhibitor, glucagon-like peptide el (GLP-1) analogue, dipeptidyl peptidiase4 (GPP-4) inhibitor, or insulin. | Depending on the comparison group, we will require new-use (defined as no use 180 days prior to index date) of canagliflozin and a comparator drug | | |
| 2 | History or high risk of cardiovascular disease defined on the basis of either: | | | |
| | – Age ≥30 years with documented symptomatic atherosclerotic cardiovascular disease: | Age ≥30 years at drug initiation | | 1 |
| | o including stroke; | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting- Any stroke: ICD-9 Dx: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetti drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA-118.039177 | |
| | o or myocardial infarction (MI); | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting- Acute MI ICD-9 410.xx, Old MI: $412.xx$ | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. "Circulation. 2019 Apr 8. doi: 10.1161/circularionNoAHA118.039177 | |
| | o or hospital admission for unstable angina; | Measured 180 days prior to drug initiation in the Inpatient care setting with ICD-9 discharge diagnosis 411.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetti drugs: population based cohort study." BMJ 2018;360:k:119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 | |

| | o | | CABG: Measured 180 days prior to drug initiation in any diagnosis position and inpatient care setting - CPT-4: 33510 – 33536, 33545, 33572. OR – | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |
|---|---|---|---|---|
| 2a | | | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting -ICD-9 procedure: 36.1x, 36.2x | Patorno, Elisabetta et al. "Empagilflozin and the Risk of Heart Failure Hospitalization in<br>Routine Clinical Care: A First Analysis from the Empagilflozin Comparative Effectiveness and<br>Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi:<br>10.1161/CIRCULATIONAHA 118.039177 |
| | 0 | or percutaneous coronary intervention (PCI; with or without stenting); | PTCA: Measured 180 days prior to drug initiation in any procedure position and inpatient care setting - CPT-4: 92973, 92982, 92984, 92995, 92996, 92920 – 92921, 92924 – 92925, 92937, 92938, 92941, 92943, 92944 Measured 180 days prior to drug initiation in any procedure position and inpatient or outpatient care setting - ICD-9 procedure: 00.66, 36.01, 36.02, 36.03, 36.05, 36.09 Stenting: Measured 180 days prior to drug initiation in any procedure position and inpatient care setting- CPT-4: 92980, 92981, 92928 – 92929, 92933 - 92934 OR – Measured 180 days prior to drug initiation in any procedure position and inpatient care setting- ICD-9 procedure: 36.06, 36.07 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs; population based cohort study." BMI 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | o | or peripheral revascularization (angioplasty or surgery); | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting - ICD-9 39.25, 39.50, 39.99. | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs; population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS) SIUCy. "Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA118.039177 |
| | o | or symptomatic with documented hemodynamically-significant carotid or peripheral vascular disease; | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting - ICD9 diagnosis: 440.20 –440.24, 440.29 –440.32, 440.3, 440.4, 443.9 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin anticliabetic drugs; population based cohort study." BMI 2018;360:k131 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS Study." ("Cruciation. 2019 Apr 8. doi: |
| | o | or amputation secondary to vascular disease. | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. Lower extremity amputation ICD-9 diagnosis: V49.7x ICD-9 procedure: 84.10-84.18 CPT: 27590, 27591, 27592, 27880, 27881, 27882, 27884, 27886, 27888, 27889, 28800, 28805, 28810, 28820, 28825 | 10.1161/CIRCULATIONAHA 118.039177 Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/jmij.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. "Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA 118.039177 |
| | – A<br>vis | ge ≥50 years with 2 or more of the following risk factors determined at the screening<br>it: | Age 250 years at drug initiation | |
| | o | duration of type 2 diabetes of 10 years or more | N/A | We can't capture diabetes duration but will match on number of antidiabetic drugs during baseline |
| 2b | o | or systolic blood pressure >140 mmHg (average of 3 readings) recorded at the screening visit | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting -<br>Hypertension ICD-9 codes 401.x – 405.x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. "Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHOLATION. |
| | 0 | or while the subject is on at least one blood pressure-lowering treatment | Dispensing of at least one of the following medications in the 180 days prior to drug initiation: ACE inhibitor Benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril ARB ARISARTAN, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan Beta blocker Acebutolo, atenoloi, betaxoloi, bisoproloi, carteoloi, carvediloi, esmoloi, labetaloi, metoproloi tartrate, metoproloi succinate, propranoloi, penbutoloi, pindoloi, nadoloi, nebivoloi, sotaloi, timoloi Calcium channel blocker Dilitazem, miberadii, verapamil, amlodipine, clevidipine, bepridii, felodipine, isradipine, nicardipine, nifedipine, nimodipine, nisodipine Loop diurettis Furosemide, bumetanide, torsemide, ethacrynic acid Other diurettis Amiloride, eplerenone, spironolactone, triamterene Other hypertension drugs Doxazosin, eplerenone, prazosin, terazosin, clonidine, guanabenz, guanadrel, guanethidine, guanfacine, hydralazine, methyldopa, metyrosine, reserpine, minoxidii, aliskiren | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |

| _ | | | |
|---|---|---|---|
| | o or current daily cigarette smoker | Measured 180 days prior to drug initiation in any diagnosis/procedure position and inpatient or outpatient are setting- [CD-9 Codes V15.82 305.1x 984.84 [CPTCodes 99406, 99407, G0436, G0437, G9016, S9453, S4995, G9276, G9458, 1034F, 4004F, 4001F OR dispensing of at least one nicotine or varenicline prescription: nicotine, varenicline | Desai, Rishi J et al. "Identification of smoking using Medicare data—a validation study of claims-based algorithms." Pharmacoepidemiology and drug safety vol. 25,4 (2016): 472-5. doi:10.1002/pds.3953 |
| | o or documented microalbuminuria or macroalbuminuria | Measured 180 days prior to drug initiation in any diagnosis/procedure position and inpatient or outpatient care setting- Proteinuria ICD 9 DX 791.0 ICD10 DX R80.X Albumin abnormality ICD9 Dx-790.99 ICD10 Dx - R77.0 | |
| | o or documented high-density lipoprotein (HDL) cholesterol of <1 mmol/l (<39 mg/dl). | N/A | |
| | Women must be: -Postmenopausal, defined as -45 years of age with amenorrhea for at least 18 months, or -45 years of age with amenorrhea for at least 6 months and less than 18 months and a serum follicle shimulating hormone (FSH) level -40 IU/ml, | Women Age >45 years <b>at drug initiation</b> OR | |
| | or Surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation), or | N/A | |
| | otherwise be incapable of pregnancy, —or Heterosexually active and practicing a highly effective method of birth control, including | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. Encounter for contraceptive management ICD9: V25 OR Non-oral contraceptives (brand names)- Depo-subQ | |
| 3 | hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrie method e.g., condoms, diaphragm, or cevical cap with spermicidal foam, cream, or gel), or male partner sterilization, consistent with local regulations regarding use of birth control methods for subjects participating in clinical trials, for the duration of their participation in the study, | Prover a 104 Depo-Provera, generic Mirena Ortho Evra NuvaRing Implanon Oral contraceptives (generic names)- See "oral contraceptives - generic" sheet. Oral contraceptives (brand names)- See "oral contraceptives - generic" sheet. | Krumme, Alexis A, et. al. "Study protocol for the dabigatran, apixaban, rivaroxaban, edoxaban, warfarin comparative effectivenes research study." J. Comp. Eff. Res. (2018):7(1), 57–66. doi: 10.2217/cer-2017-0053. |
| | – or Not heterosexually active. Note: subjects who are not heterosexually active at screening must agree to utilize a highly effective method of birth control if they become heterosexually active during their participation in the study. | N/A | |
| 4 | Women of childbearing potential must have a negative urine β-human chorionic | N/A | One of the exclusion criteria is pregnancy, so this can be skipped. |
| 5 | gonadotropin (β-hCG) pregnancy test at screening and baseline (predose, Day 1). Willing and able to adhere to the prohibitions and restrictions specified in this protocol. | N/A | |
| 6 | Subjects must have signed an informed consent document indicators specified in an inspiration. Subjects must have signed an informed consent document indicators that they understand the purpose of and procedures required for the study and are willing to participate in the study. | N/A | |
| 7 | To participate in the optional pharmacogenomic component of this study, subjects must<br>have signed the informed consent form for pharmacogenomic research indicating<br>willingness to participate in the pharmacogenomic component of the study (where local<br>regulations permit). Refusal to give consent for this component does not exclude a subject<br>from participation in the clinical study. | N/A | |
| 8 | Subjects must have taken ≥80% of their single-blind placebo capsules during the 2-week | N/A | |
| $\vdash$ | run-in period at Day 1 to be eligible for randomization. | <u> </u> | |
| | EXCLUSION CRITERIA EXCLUSION CRITERIA | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting- DM type 1-At least 1 $(C9-9) \times code of 250.x1 $ or $250.x3$ or $(CD-10) \times code of E10.x$ Measured 180 days prior to drug initiation in any procedure position and inpatient or outpatient care setting- | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus |
| 1 | History of diabetic ketoacidosis, type 1 diabetes, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy. | setting. Secondary diabetes ICD-9 procedure: 249.xx Secondary diabetes Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. Ketoacidosis 250.1x Notes: We can't capture pancreas or beta-cell transplantation in claims datasets. | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagiliflorin versus other non-glifloria nartidiabette drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS ISUdy." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 2 | On an AHA and not on a stable regimen (i.e., agents and doses) for at least 8 weeks before<br>the screening visit and through the screening/run-in period. Note: a stable dose of insulin<br>is defined as no change in the insulin regimen (i.e., type[s] of insulin) and s15% change in<br>the total daily dose of insulin (averaged over 1 week to account for day-to-day variability). | N/A | |

| 3 | —For patients on a sulfonylurea agent or on insulin: fasting fingerstick glucose at site <10 mg/dl (-6 mmol/) at Baseline/Day 1. Note: at the investigator's discretion, based upon an assessment of recent self-monitored blood glucose (SMBG) values, subjects meeting either of these fingerstick glucose exclusion criteria may continue the single bilind placebo and return to the investigational site within 14 days and may be randomized if the repeat fasting fingerstick value no longer meets the exclusion criterion. Subjects with fingerstick glucose >270 mg/dl (>15 mmol/) may have their AHA regimen adjusted and be rescreened once on a stable regimen for at least 8 weeks. | N/A | |
|---|---|---|---|
| 4 | History of one or more severe hypoglycemic episode within 6 months before screening. Note: a severe hypoglycemic episode is defined as an event that requires the help of another person. | Measured 180 days prior to drug initiation in primary diagnosis position and inpatient care setting-<br>ICD-9 diagnosis:<br>251.0, 251.1x, 251.2x, or 250.8x.<br>If identified by 250.8x are not included if they co-occur with one of the following diagnoses:<br>259.8, 272.7, 681.xx, 682.xx, 686.9, 707.1x, 707.2x, 707.8, 707.9, 709.3, 730.0x, 730.1x, 730.2x,<br>731.8. | PPV 89% (ED component) – Ginde AA, Blanc PG, Lieberman RM, Camargo CA, Jr. Validation of ICD-9-CM coding algorithm for improved identification of hypoglycemia visits. BMC endocrine disorders 2008;8:4. PPV 78% (inpatient component) – Schelleman H, Bilker WB, Brensinger CM, Wan F, Hennessy S. Anti-infectives and the risk of severe hypoglycemia in users of glipizide or glyburide. Clinical pharmacology and therapeutics 2010;88:214-22. |
| 5 | History of hereditary glucose galactose malabsorption or primary renal glucosuria. | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. ICD-9 diagnosis codes: 271.3x, 271.4x | Elisabetta suggested these codes |
| 6 | Ongoing, inadequately controlled thyroid disorder. Note: subjects on thyroid hormone-replacement therapy must be on a stable dose for at least 6 weeks before Day 1. | N/A | |
| 7 | Renal disease that required treatment with immunosuppressive therapy or a history of dialysis or renal transplant. Note: subjects with a history of treated childhood renal disease, without sequelae, may participate. | Measured 180 days prior to drug initiation - 1. Acute renal diseases OR Chronic Renal Insufficiency in any diagnosis position and inpatient or outpatient care setting AND dispensing of an immunosuppressive agent: Acute Renal Disease 572.4x, 580.xx, 584.xx, 791.2x, 791.3x Chronic Renal Insufficiency 582.xx, 583.xx, 585.xx, 586.xx, 587.xx Immunosuppressive therapy: HCPCS codes "36514", "80420", "02526", "10702", "10704", "11020", "11030", "11040", "11094", "11095", "11095", "11303", "11706", "11700", "11700", "17500", "17504", "17504", "17624", "17637", "17638", "17683", "17684", "18540", "K0512", "K0513", "K0528", "50173" with immunosuppressive agents in next tab "immunosuppressive agents" OR 2. Dialysis in any diagnosis position and inpatient care setting OR Renal transplant in any diagnosis position and inpatient care setting Codes are in the sheet 'Dialysis and Renal Transplant' | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2013;360k:18 http://dx.doi.org/10.1136/bmj.kt19 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 8 | MI, unstable angina, revascularization procedure, or cerebrovascular accident within 3 months before screening, or a planned revascularization procedure, or history of New York Heart Association (NYHA) Class IV cardiac disease. | Measured 90 days prior to drug initiation in any diagnosis/procedure position and care setting defined below. Any of the following codes in inpatient or outpatient care setting: MI ICD-9 diagnosis 410.xx Unstable angina ICD-9 diagnosis 411.xx Left ventricular assist. CPT-4 33990-33993 Stroke ICD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.x1, 436.x Carotid bypass: ICD9 procedure: 39.28 TA 435.xx Peripheral arterial stenting or surgical revascularization ICD-9 39.25, 39.50, 39.99. PTCA: Inpatient CPT-4: 92973, 92982, 92984, 92995, 92996, 92920 –92921, 92924 –92925, 92937, 92938, 92941, 92943, 92944 OR Inpatient or outpatient -ICD-9 procedure: 00.66, 36.01, 36.02, 36.03, 36.05, 36.09 Stenting: Inpatient CPT-4: 9280, 92981, 92928 –92929, 92933 -92934 – OR – Inpatient or outpatient -ICD-9 procedure: 36.06, 36.07 CABG: Inpatient CPT-4: 33310 – 33536, 33536, 33572 – OR – Inpatient or outpatient -ICD-9 procedure: 36.1x, 36.2x Transmyocardial revascularization: Inpatient or Outpatient CPT-4: 33140, 33141 OR - Inpatient or outpatient ICD-9 procedure: 36.31-36.34 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagiiflozin versus other non-gilflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/pmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: AFirst Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Agr 8. doi: 10.1161/CIRCULATIONAHA-11.80-39317 Left Ventricular Assist Codes from-http://www.hcpro.com/HIM-289708-859/Tip-Note-new-codes-for-ventricular-assist-devices.html |
| 9 | Findings on 12-lead electrocardlogram (ECG) that would require urgent diagnostic evaluation or intervention (e.g., new clinically important arrhythmia or conduction disturbance). | Measured 180 days prior to drug initiation in primary diagnosis position and inpatient care setting-<br>Cardiac conduction disorders ICD 9: 425.xx.<br>Other cardiac dysrhythmia ICD 9: 427.xx., exclude 427.5x (cardiac arrest) and 427.3x<br>And, 427.6x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagifflozin versus other non-gilliozin antidiabetic drugs: population based cohort study." BMJ 2018;360-k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagifflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagifflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA1.118.039177 |

| 10 | History of hepatitis B surface antigen or hepatitis C antibody positive (unless associated with documented persistently stable/normal range aspartate aminotransferase [AST] and alanine aminotransferase [ALT] levels), or other clinically active liver disease. | Measured 180 days prior to drug initiation in any diagnosis/procedure position and inpatient or outpatient care setting-<br>Liver disease- ICD-9 diagnosis: 070.xx, 570.xx-573.xx 456.0x-456.Zx, 576.8x, 782.4x, 789.5x ICD-9 procedure codes: 39.1x, 42.91 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gillflozin alidabetic drugs; population based cohort study." BMJ 2018;360:119 http://dx.doi.org/10.1136/bmj.kt/p. Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
|---|---|---|---|
| 11 | Any history of or planned bariatric surgery. | Measured 1825 days prior to drug initiation in any procedure position and inpatient or outpatient care setting. CPT-Code-Abbreviation Procedure 43644 - LRYBG - Laparoscopic Roux-en-Ygastric bypass (Roux limb 150 cm or less) 43645 - LRYGBX- Laparoscopic gastric bypass with small intestine reconstruction to limit absorption 43770 - LAGB- Laparoscopic adjustable gastric band 43874 - CRYGBX- Open Roux-en-Ygastric bypass (Roux limb 150 cm or less) 43846 - GRYGB- Open Roux-en-Ygastric bypass (Roux limb 150 cm or less) 43847 - CRYGBX- Open gastric bypass with small intestine reconstruction to limit absorption | Hatoam, Ida J et al. "Clinical Factors Associated With Remission of Obesity-Related Comorbidities After Bariatric Surgery." JAMA Surg. 2016;151(2):130-137. doi:10.1001/jamasurg.2015.3231 |
| 12 | Estimated glomerular filtration rate (eGFR)<30 ml/min/1.73 m2 at screening (provided by the central laboratory) - For subjects taking metformin: at screening, serum creatinine ≥1.4 mg/dl (124 µmol/l) for men or ≥1.3 mg/dl (115 µmol/l) for women; no contraindication to the use of metformin (including eGFR) based on the label of the country of investigational site | N/A | |
| 13 | ALT levels > 2.0 times the upper limit of normal (ULN) or total bilirubin > 1.5 times the ULN at screening, unless in the opinion of the investigator and as agreed upon by the sponsor's medical officer, the findings are consistent with Gilbert's disease. | N/A | |
| 14 | History of malignancy within 5 years before screening (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the service with service and service with the sponsor's medical monitor, is considered cured with minimal risk of recurrence). | Measured 1825 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting-<br>History of malignant neoplasm 140.xx-208.xx (except 173.xx, non-melanoma skin cancer) | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gilliozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: AFirst Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.1180.303177 |
| 15 | History of human immunodeficiency virus (HIV) antibody positive. | Measured 1825 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. 402 Human immunodeficiency virus [HIV] disease 079.53 Human immunodeficiency virus, type 2 [HIV-2] V08 Asymptomatic human immunodeficiency virus [HIV] infection status OR filled prescription for HIV treatment: (Please see HIV Treatment sheet) | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRES) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 16 | Subject has a current clinically important hematological disorder (e.g., symptomatic anemia, proliferative bone marrow disorder, thrombocytopenia). | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. [CD-9 Diagnosis Codes: 238.4x, 289.83, 238.71, 280.x-285.x, 287.3x, 287.4x, 287.5x | Expert in this study area advised on the codes used for this inclusion/exclusion criteria. |
| 17 | Investigator's assessment that the subject's life expectancy is less than 1 year, or any condition that in the opinion of the investigator would make participation not in the best interest of the subject, or could prevent, limit, or confound the protocol-specified safety or efficacy assessments. | Measured 180 days prior to drug initiation-<br>CCI >=10 | Gagne, Josh J et. al. "A combined comorbidity score predicted mortality in elderly patients<br>better than existing scores." I Clin Epidemiol. 2011 Jul;64(7):749-59. doi:<br>10.1016/j.jclinpe.1201.0.10.004.<br>Sun, Jenny W et. al. "Validation of the Combined Comorbidity Index of Charlson and<br>Elixhauser to Predict 30-0ay Mortality Across ICD-9 and ICD-10." Med Care. 2018<br>Sep:56(9):812. doi: 10.1079/MR.000000000000954. |
| 18 | Major surgery (i.e., requiring general anesthesia) within 3 months of the screening visit or any surgery planned during the subject's expected participation in the study (except minor surgery; i.e., outpatient surgery under local anesthesia). | Measured 90 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting-<br>Major surgery selected from codes range 35.x-84.x | |
| 19 | Any condition that, in the opinion of the investigator, would compromise the well-being of<br>the subject or prevent the subject from meeting or performing study requirements. | N/A | |
| 20 | Current use of other sodium glucose co-transporter 2 (SGLT2) inhibitor. | Measured 180 days prior to drug initiation as a dispensing of one of the following drugs-<br>empagliflozin, dapagliflozin, ertugliflozin | |
| 21 | Known allergies, hypersensitivity, or intolerance to canagliflozin or its excipients. | N/A | |
| 22 | Current use of a corticosteroid medication or immunosuppressive agent, or likely to require treatment with a corticosteroid medication (for longer than 2 weeks in duration) or an immunosuppressive agent. Note: subjects using inhaled, intranasal, intra-articular, or topical corticosteroids, or corticosteroids in therapeutic replacement doses may participate. | Measured 180 days prior to drug initiation as a dispensing of one of the following drugs- Systemic corticosteroids (With Route of Administration is intravenous): Cortisone, hydrocortisone, prednisone, prednisone, methylprednisolone, triamcinolone, dexamethasone, betamethasone. immunosuppressive agents o RA, AS, and PS4: methotrexate, hydroxychloroquine, azathioprine, cyclosporine, lefunomide, minocycline, sulfasalazine. o SLE: hydroxychloroquine, azathioprine, mycophenolate mofetil. o IBD: azathioprine, mercaptopurine | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMU 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS tudy." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 Desai, Rishi et. al. "Risk of serious infections associated with use of immunosuppressive agents in pregnant women with autoimmune inflammatory conditions: cohort study" BMU 2017; 356 doi: https://doi.org/10.1136/bmj.j895 |
| 23 | Received an active investigational drug (including vaccines) or used an investigational medical device within 3 months before Day 1/baseline or received at least one dose of canagilflozin in a prior study. | Already applied based on the canagliflozin and comparator washout, but measured again <b>90 days prior to drug initiation</b> as a dispensing for <b>canagliflozin</b> | |

| 24 | History of drug or alcohol abuse within 3 years before screening. | Measured 1095 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting. Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study," BMJ 2013;360k:18 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA118.039177 |
|---|---|---|---|
| 25 | Pregnant or breastfeeding or planning to become pregnant or breastfeed during the study. | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care<br>settles. (Please see Pregnancy Sheet for code list) | |
| 26 | Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator. | N/A | |

| <u>Trial ID</u> | sNDA22 |
|---|---|
| Trial Name (with web links) | CANVAS |
| <u>NCT</u> | NCT01032629 |
| <u>Trial category</u> | Secondary indication |
| Therapeutic Area | Endocrinology |
| RCT Category | 4a- Unintended S with label change |
| <b>Brand Name</b> | Invokana |
| <b>Generic Name</b> | Canagliflozin |
| Sponsor | Janssen Research & Development, LLC |
| <u>Year</u> | 2017 |
| Measurable endpoint | Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial |
| <u>Ivieasurable enuponit</u> | Infarction (MI), and Nonfatal Stroke |
| <u>Exposure</u> | Canaglifloziin |
| <u>Comparator</u> | Placebo |
| <u>Population</u> | 50% on insulin, 47% using Sulfonylurea, 73% Metformin, 72% statin |
| <u>Trial finding</u> | HR = 0.86 (95% CI 0.75–0.97) |
| No. of Patients | 4330 |
| Non-inferiority margin | HR = 1.3 |
| Assay Sens. Endpoint | |
| Assay Sens. Finding | |
| | 0.90. With 688 cardiovascular safety events recorded across the trials, there would be at least 90% power, at an alpha level of 0.05, to |
| <u>Power</u> | exclude an upper margin of the 95% confidence interval for the hazard ratio of 1.3. |
| Blinding | |
| | Cardiovascular safety was to be shown if the upper boundary of the 95% confidence interval of the hazard ratio with canagliflozin as compared with |
| Statistical Method | placebo was less than 1.3, and superiority was to be shown if the upper<br>boundary was less than 1.0. |

### Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)

- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

### 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| drug_class | Brand Name |
|--------------------|---------------|
| oral contraceptive | Apri; |
| oral contraceptive | Desogen; |
| oral contraceptive | Ortho-Cept; |
| oral contraceptive | Reclipsen |
| oral contraceptive | Kariva; |
| oral contraceptive | Mircette |
| oral contraceptive | Cyclessa; |
| oral contraceptive | Velivet |
| oral contraceptive | Yasmin |
| oral contraceptive | Yaz |
| oral contraceptive | Demulen 1/35; |
| oral contraceptive | Kelnor; |
| oral contraceptive | Zovia 1/25 |
| oral contraceptive | Demulen 1/50; |
| oral contraceptive | Zovia 1/50 |
| oral contraceptive | Alesse; |
| oral contraceptive | Aviane; |
| oral contraceptive | Lessina; |
| oral contraceptive | Lutera |
| oral contraceptive | Nordette; |
| oral contraceptive | Portia; |
| oral contraceptive | Levora |
| oral contraceptive | Lybrel |
| oral contraceptive | Seasonale; |
| oral contraceptive | Quasense; |
| oral contraceptive | Jolessa |
| oral contraceptive | Seasonique |
| oral contraceptive | Empresse; |
| oral contraceptive | Triphasil; |
| oral contraceptive | Trivora |
| oral contraceptive | Ovcon 35 |
| oral contraceptive | Balziva; |

| oral contraceptive | Femcon Fe |
|--------------------|----------------------|
| oral contraceptive | Brevicon; |
| oral contraceptive | Nortrel 0.5/35; |
| oral contraceptive | Modicon; |
| oral contraceptive | Necon 0.5/35 |
| oral contraceptive | Norinyl 1/35; |
| oral contraceptive | Nortrel 1/35; |
| oral contraceptive | Ortho-Novum 1/35; |
| oral contraceptive | Necon 1/35 |
| oral contraceptive | Ovcon 50; |
| oral contraceptive | Necon 1/50 |
| oral contraceptive | Ortho-Novum 10/11 |
| oral contraceptive | Aranelle; |
| oral contraceptive | Tri-Norinyl |
| oral contraceptive | Ortho-Novum 7/7/7; |
| oral contraceptive | Necon |
| oral contraceptive | Micronor; |
| oral contraceptive | Nor-QD; |
| oral contraceptive | Camila; |
| oral contraceptive | Errin; |
| oral contraceptive | Jolivette |
| oral contraceptive | Junel 21 1/20; |
| oral contraceptive | Junel 21 Fe 1/20; |
| oral contraceptive | Loestrin 21 1/20; |
| oral contraceptive | Loestrin 21 Fe 1/20; |
| oral contraceptive | Loestrin 24 Fe; |
| oral contraceptive | Microgestin 1/20 |
| oral contraceptive | Microgestin Fe 1/20 |
| oral contraceptive | Junel 21 1.5/30; |
| oral contraceptive | Junel 21 Fe 1.5/30; |
| oral contraceptive | Loestrin 1.5/30; |
| oral contraceptive | Loestrin Fe 1.5/30 |
| oral contraceptive | Microgestin 1.5/30 |
| • | |

| oral contraceptive | Microgestin Fe 1.5/30 |
|--------------------|-----------------------|
| oral contraceptive | Estrostep Fe; |
| oral contraceptive | Tilia Fe; |
| oral contraceptive | TriLegest Fe |
| oral contraceptive | Ortho-Cyclen; |
| oral contraceptive | Sprintec; |
| oral contraceptive | MonoNessa; |
| oral contraceptive | Previfem |
| oral contraceptive | Ortho Tri-Cyclen Lo; |
| oral contraceptive | Tri-Previfem; |
| oral contraceptive | TriNessa |
| oral contraceptive | Ortho Tri-Cyclen; |
| oral contraceptive | Tri-Sprintec |
| oral contraceptive | Cryselle; |
| oral contraceptive | Lo/Ovral; |
| oral contraceptive | Low-Ogestrel |
| oral contraceptive | Ovral; |
| oral contraceptive | Ogestrel |
| oral contraceptive | Zovia 1/50 |
| oral contraceptive | Alesse; |
| oral contraceptive | Aviane; |
| oral contraceptive | Lessina; |
| oral contraceptive | Lutera |
| oral contraceptive | Nordette; |
| oral contraceptive | Portia; |
| oral contraceptive | Levora |
| oral contraceptive | Lybrel |
| oral contraceptive | Seasonale; |
| oral contraceptive | Quasense; |
| oral contraceptive | Jolessa |
| oral contraceptive | Seasonique |
| oral contraceptive | Empresse; |
| oral contraceptive | Triphasil; |

| oral contraceptive | Trivora |
|--------------------|----------------------|
| oral contraceptive | Ovcon 35 |
| oral contraceptive | Balziva; |
| oral contraceptive | Femcon Fe |
| oral contraceptive | Brevicon; |
| oral contraceptive | Nortrel 0.5/35; |
| oral contraceptive | Modicon; |
| oral contraceptive | Necon 0.5/35 |
| oral contraceptive | Norinyl 1/35; |
| oral contraceptive | Nortrel 1/35; |
| oral contraceptive | Ortho-Novum 1/35; |
| oral contraceptive | Necon 1/35 |
| oral contraceptive | Ovcon 50; |
| oral contraceptive | Necon 1/50 |
| oral contraceptive | Ortho-Novum 10/11 |
| oral contraceptive | Aranelle; |
| oral contraceptive | Tri-Norinyl |
| oral contraceptive | Ortho-Novum 7/7/7; |
| oral contraceptive | Necon |
| oral contraceptive | Micronor; |
| oral contraceptive | Nor-QD; |
| oral contraceptive | Camila; |
| oral contraceptive | Errin; |
| oral contraceptive | Jolivette |
| oral contraceptive | Junel 21 1/20; |
| oral contraceptive | Junel 21 Fe 1/20; |
| oral contraceptive | Loestrin 21 1/20; |
| oral contraceptive | Loestrin 21 Fe 1/20; |
| oral contraceptive | Loestrin 24 Fe; |
| oral contraceptive | Microgestin 1/20 |
| oral contraceptive | Microgestin Fe 1/20 |
| oral contraceptive | Junel 21 1.5/30; |
| oral contraceptive | Junel 21 Fe 1.5/30; |

| oral contraceptive | Loestrin 1.5/30; |
|--------------------|-----------------------|
| oral contraceptive | Loestrin Fe 1.5/30 |
| oral contraceptive | Microgestin 1.5/30 |
| oral contraceptive | Microgestin Fe 1.5/30 |
| oral contraceptive | Estrostep Fe; |
| oral contraceptive | Tilia Fe; |
| oral contraceptive | TriLegest Fe |
| oral contraceptive | Ortho-Cyclen; |
| oral contraceptive | Sprintec; |
| oral contraceptive | MonoNessa; |
| oral contraceptive | Previfem |
| oral contraceptive | Ortho Tri-Cyclen Lo; |
| oral contraceptive | Tri-Previfem; |
| oral contraceptive | TriNessa |
| oral contraceptive | Ortho Tri-Cyclen; |
| oral contraceptive | Tri-Sprintec |
| oral contraceptive | Cryselle; |
| oral contraceptive | Lo/Ovral; |
| oral contraceptive | Low-Ogestrel |
| oral contraceptive | Ovral; |
| oral contraceptive | Ogestrel |
| drug_class | generic | generic_ndc |
|---|---|---|
| oral contraceptive | estradiol | desogestrel-ethinyl estradiol |
| oral contraceptive | estradiol | desogestrel-ethinyl estradiol/ethinyl estradiol |
| oral contraceptive | estradiol | drospirenone/estradiol |
| oral contraceptive | estradiol | drospirenone/ethinyl estradiol/levomefolate calcium |
| oral contraceptive | estradiol | estradiol |
| oral contraceptive | estradiol | estradiol acetate |
| oral contraceptive | estradiol | estradiol benzoate |
| oral contraceptive | estradiol | estradiol cypionate |
| oral contraceptive | estradiol | estradiol cypionate/medroxyprogesterone acet |
| oral contraceptive | estradiol | estradiol hemihydrate, micronized |
| oral contraceptive | estradiol | estradiol micronized |
| oral contraceptive | estradiol | estradiol valerate |
| oral contraceptive | estradiol | estradiol valerate/dienogest |
| oral contraceptive | estradiol | estradiol valerate/sesame oil |
| oral contraceptive | estradiol | estradiol/estrone |
| oral contraceptive | estradiol | estradiol/estrone/vit b12 |
| oral contraceptive | estradiol | estradiol/levonorgestrel |
| oral contraceptive | estradiol | estradiol/norethindrone acetate |
| oral contraceptive | estradiol | estradiol/norgestimate |
| oral contraceptive | estradiol | estradiol/progesterone |
| oral contraceptive | estradiol | ethinyl estradiol |
| oral contraceptive | estradiol | ethinyl estradiol/drospirenone |
| oral contraceptive | estradiol | ethinyl estradiol/norethindrone acetate |
| oral contraceptive | estradiol | ethynodiol d-ethinyl estradiol |
| oral contraceptive | estradiol | ethynodiol diacetate-ethinyl estradiol |
| oral contraceptive | estradiol | etonogestrel/ethinyl estradiol |
| oral contraceptive | estradiol | levonorgestrel-ethinyl estradiol |
| oral contraceptive | estradiol | levonorgestrel/ethinyl estradiol and ethinyl estradiol |
| oral contraceptive | estradiol | me-testosterone/eth estradiol |
| oral contraceptive | estradiol | metttm/estradiol/multivits |
| oral contraceptive | estradiol | norelgestromin/ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone a-e estradiol |
| oral contraceptive | estradiol | norethindrone a-e estradiol/fe |

| oral contraceptive | estradiol | norethindrone a-e estradiol/ferrous fumarate |
|---|---|---|
| oral contraceptive | estradiol | norethindrone acetate-ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone acetate-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | estradiol | norethindrone-ethin estradiol |
| oral contraceptive | estradiol | norethindrone-ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | estradiol | norgestimate-ethinyl estradiol |
| oral contraceptive | estradiol | norgestrel-ethinyl estradiol |
| oral contraceptive | estradiol | testosterone cypionate/estradiol cypionate |
| oral contraceptive | estradiol | testosterone enanthate/estradiol valerate |
| oral contraceptive | estradiol | testosterone/estradiol |
| oral contraceptive | levonorgestrel | estradiol/levonorgestrel |
| oral contraceptive | levonorgestrel | levonorgestrel |
| oral contraceptive | levonorgestrel | levonorgestrel-eth estra |
| oral contraceptive | levonorgestrel | levonorgestrel-eth estra/pregnancy test kit |
| oral contraceptive | levonorgestrel | levonorgestrel-ethinyl estradiol |
| oral contraceptive | levonorgestrel | levonorgestrel/ethinyl estradiol and ethinyl estradiol |
| oral contraceptive | norethindrone | estradiol/norethindrone acetate |
| oral contraceptive | norethindrone | ethinyl estradiol/norethindrone acetate |
| oral contraceptive | norethindrone | leuprolide acetate/norethindrone acetate |
| oral contraceptive | norethindrone | norethindrone |
| oral contraceptive | norethindrone | norethindrone a-e estradiol |
| oral contraceptive | norethindrone | norethindrone a-e estradiol/fe |
| oral contraceptive | norethindrone | norethindrone a-e estradiol/ferrous fumarate |
| oral contraceptive | norethindrone | norethindrone acetate |
| oral contraceptive | norethindrone | norethindrone acetate-ethinyl estradiol |
| oral contraceptive | norethindrone | norethindrone acetate-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | norethindrone | norethindrone-ethin estradiol |
| oral contraceptive | norethindrone | norethindrone-ethinyl estrad |
| oral contraceptive | norethindrone | norethindrone-ethinyl estradiol |
| oral contraceptive | norethindrone | norethindrone-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | norethindrone | norethindrone-mestranol |

| oral contraceptive | norgestrel | norgestrel |
|--------------------|-------------------------|------------------------------|
| oral contraceptive | norgestrel | norgestrel-ethinyl estradiol |
| oral contraceptive | polyestradiol phosphate | polyestradiol phosphate |

| Antidiabetic class | Specific agent | Notes |
|---|---|---|
| | Canagliflozin | Approved 3/29/2013 |
| SGLT2-inhibitors | Dapagliflozin | |
| SGL 12-Infilotions | Empagliflozin | |
| | Ertugliflozin | Approved Dec 21, 2017 |
| | Glimepiride | |
| 2 <sup>nd</sup> generation sulfonylureas | Glipizide | |
| | Glyburide | |
| | Alogliptin | |
| DPP-4 inhibitors | Linagliptin | |
| DFF-4 lillionois | Saxagliptin | |
| | Sitagliptin | |
| | Exenatide | |
| | Liraglutide | |
| GLP-1 receptor agonist (GLP1-RA) | Albiglutide | Approved April 15, 2014 and discontinued July 26, 2017 |
| | Dulaglutide | Approved Sep 18, 2014 |
| | Lixisenatide | Approved July 28, 2016 |
| | Semaglutide | Approved Dec 5, 2017 |
| | Insulin Aspart | |
| | Insulin Aspart/Insulin Aspart Protamine | |
| | Insulin Degludec | |
| | Insulin Detemir | |
| | Insulin Glargine | |
| | Insulin Glulisine | |
| Insulin | Insulin human isophane (NPH) | |
| | Insulin human regular (search with NPH, | |
| | don't want bf-pk) | |
| | Insulin human regular/ Insulin human | |
| | isophane (NPH) | |
| | Insulin Lispro | |
| | Insulin Lispro/Insulin Lispro Protamine | |
| Glitazonas | Pioglitazone | |

| Uiitazuiies | Rosiglitazone |
|------------------------------------------|----------------|
| Maglitinidae | Nateglinide |
| Meglitinides | Repaglinide |
| Alpha-glucosidase inhibitors | Acarbose |
| Alpha-glucosidase inhibitors | Miglitol |
| Pramlintide | Pramlintide |
| | Acetohexamide |
| 1 st companding sulfamely mass | Chlorpropamide |
| 1 <sup>st</sup> generation sulfonylureas | Tolazamide |
| | Tolbutamide |

#### Immunosuppressive agents

**ALEMTUZUMAB** 

BETAMETHASONE

BETAMETHASONE ACETATE/BETAMETHASONE SODIUM PHOSPHATE

BETAMETHASONE DIPROPIONATE

BETAMETHASONE DIPROPIONATE/PROPYLENE GLYCOL

BETAMETHASONE SODIUM PHOSPHATE

BETAMETHASONE VALERATE

BUDESONIDE

BUDESONIDE. MICRONIZED

**CORTISONE ACETATE** 

DEXAMETHASONE

DEXAMETHASONE ACETATE

DEXAMETHASONE ACETATE. MICRONIZED

DEXAMETHASONE ISONICOTINATE

DEXAMETHASONE PHOSPHATE

DEXAMETHASONE SOD PHOSPHATE

DEXAMETHASONE SODIUM PHOSPHATE IN 0.9 % SODIUM CHLORIDE

DEXAMETHASONE SODIUM PHOSPHATE/PF

DEXAMETHASONE. MICRONIZED

**HYDROCORTISONE** 

HYDROCORTISONE ACETATE

HYDROCORTISONE CYPIONATE

HYDROCORTISONE SOD PHOSPHATE

HYDROCORTISONE SOD SUCCINATE

IMMUNE GLOBULIN, BOVINE/PLASMA PROTEIN FRACTION, BOVINE

IMMUNE GLOBULIN, GAMM (IGG)/GLYCINE/GLUCOSE/IGA 0 TO 50 MCG/ML

IMMUNE GLOBULIN, GAMM(IGG)/GLYCINE/IGA GREATER THAN 50 MCG/ML

IMMUNE GLOBULIN, GAMM(IGG)/MALTOSE/IGA GREATER THAN 50 MCG/ML

IMMUNE GLOBULIN.GAMM(IGG)/SORBITOL/GLYCIN/IGA 0 TO 50 MCG/ML

IMMUNE GLOBULIN, GAMM(IGG)/SUCROSE/IGA GREATER THAN 50 MCG/ML

IMMUNE GLOBULIN, GAMMA (IGG)/GLYCINE/IGA 0 TO 50 MCG/ML

IMMUNE GLOBULIN, GAMMA (IGG)/PROLINE/IGA 0 TO 50 MCG/ML

IMMUNE GLOBULIN,GAMMA (IGG)/SORBITOL/IGA 0 TO 50 MCG/ML LYMPHOCYTE IG, ANTITHYMOCYTE/THIMEROSAL LYMPHOCYTE IMMUNE GLOBULIN, ANTITHYMOCYTE (EQUINE) **METHYLPREDNISOLONE** METHYLPREDNISOLONE ACETATE METHYLPREDNISOLONE ACETATE. MICRONIZED METHYLPREDNISOLONE SODIUM SUCCINATE METHYLPREDNISOLONE SODIUM SUCCINATE/PF METHYLPREDNISOLONE, MICRONIZED **PREDNISOLONE** PREDNISOLONE ACETATE PREDNISOLONE ACETATE, MICRONIZED PREDNISOLONE SOD PHOSPHATE PREDNISOLONE, MICRONIZED **PREDNISONE** PREDNISONE MICRONIZED **RITUXIMAB** RITUXIMAB/HYALURONIDASE, HUMAN RECOMBINANT TRIAMCINOLONE TRIAMCINOLONE DIACETATE TRIAMCINOLONE HEXACETONIDE TRIAMCINOLONE HEXACETONIDE, MICRONIZED AZATHIOPRINE AZATHIOPRINE SODIUM CYCLOSPORINE CYCLOSPORINE, MODIFIED HYDROXYCHLOROQUINE SULFATE LEFLUNOMIDE MERCAPTOPURINE MINOCYCLINE HCL MINOCYCLINE HCL MICROSPHERES MINOCYCLINE HCL/EMOL COMB NO.16/SKIN CLNSR L4/TOP AGENT NO.3 MINOCYCLINE HCL/EYELID CLEANSER COMBINATION NO. 1 MINOCYCLINE HCL/WIPES WITH SKIN CLEANSER NO.4 MYCOPHENOLATE MOFETIL

MYCOPHENOLATE MOFETIL HCL

SULFASALAZINE

#### **HIV Treatment** Abacavir Amprenavir Atazanavir Darunavir Delavirdine Didanosine Efavirenz Emtricitabine Enfuvirtide Etravirine Fosamprenavir Indinavir Lamivudine-Zidovudine Maraviroc Nelfinavir Nevirapine Raltegravir Rilpivirine Ritonavir Ritonavir-Lopinavir Saquinavir Stavudine Tipranavir Zalcitabine Zidovudine

#### **Pregnancy** Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

#### **Dialysis codes**

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512. Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition. etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

-ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

-ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

- CPT4 codes:

50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy

50365, Renal allotransplantation, implantation, graft, w/ donor & recipient nephrectomy

#### Appendix B: Canagliflozin vs DPP4i



| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| ו | Optu | ım | Market | Scan | Medicare | | | POOLED | |
| Variable | Reference- DPP4i | Exposure-Canagliflozin | Reference- DPP4i | Exposure-Canagliflozin | Reference-DPP4i | Exposure-<br>Canagliflozin | Reference-DPP4i | Exposure- Canagliflozin | St. Diff. |
| Number of patients | 92,973 | 21,346 | 98,975 | 26,910 | 258,794 | 35,115 | 450,742 | 83,371 | |
| Age | | | | | | | | | |
| mean (sd) | 67.55 (9.32) | 62.19 (7.89) | 62.13 (8.88) | 59.26 (6.45) | 73.88 (6.99) | 70.94 (5.13) | 69.99 (7.96) | 64.93 (6.36) | 0.70 |
| median [IQR] | 68.00 [60.00, 74.00] | 61.00 [56.00, 68.00] | 61.00 [56.00, 66.00] | 59.00 [54.00, 63.00] | 72.00 [68.00, 78.00] ) | .00 [67.00, 74.00] | 68.76 (7.96) | 64.15 (6.36) | 0.64 |
| Age categories18 - 54; n (%) | 9,311 (10.0%) | 4,143 (19.4%) | 19,542 (19.7%) | 6,882 (25.6%) | 0 (0.0%) | 0 (0.0%) | 28,853 (6.4%) | 11,025 (13.2%) | -0.23 |
| 16 - 54, 11 (%)<br>55 - 64; n (%) | 23,950 (25.8%) | 9,021 (42.3%) | 50,842 (51.4%) | 15,706 (58.4%) | 3,273 (1.3%) | 396 (1.1%) | 78,065 (17.3%) | 25,123 (30.1%) | -0.30 |
| 65 - 74; n (%) | 38,089 (41.0%) | 6,682 (31.3%) | 17,664 (17.8%) | 3,566 (13.3%) | 152,505 (58.9%) | 27,352 (77.9%) | 208,258 (46.2%) | 37,600 (45.1%) | 0.02 |
| >= 75; n (%) | 21,623 (23.3%) | 1,500 (7.0%) | 10,927 (11.0%) | 756 (2.8%) | 103,016 (39.8%) | 7,367 (21.0%) | 135,566 (30.1%) | 9,623 (11.5%) | 0.47 |
| Gender | | | | | | | | | |
| Males; n (%) | 46,266 (49.8%) | 12,127 (56.8%) | 54,577 (55.1%) | 15,161 (56.3%) | 113,623 (43.9%) | 18,052 (51.4%) | 214,466 (47.6%) | 45,340 (54.4%) | -0.14 |
| Females; n (%) Race | 46,707 (50.2%) | 9,219 (43.2%) | 44,398 (44.9%) | 11,749 (43.7%) | 145,171 (56.1%) | 17,063 (48.6%) | 236,276 (52.4%) | 38,031 (45.6%) | 0.14 |
| White; n (%) | N/A | N/A | N/A | N/A | 191,721 (74.1%) | 28,985 (82.5%) | 191,721 (74.1%) | 28,985 (82.5%) | -0.20 |
| Black; n (%) | N/A | N/A | N/A | N/A | 30,531 (11.8%) | 2,789 (7.9%) | 30,531 (11.8%) | 2,789 (7.9%) | 0.13 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 12,516 (4.8%) | 906 (2.6%) | 12,516 (4.8%) | 906 (2.6%) | 0.12 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 12,026 (4.6%) | 951 (2.7%) | 12,026 (4.6%) | 951 (2.7%) | 0.10 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 1,608 (0.6%) | 130 (0.4%) | 1,608 (0.6%) | 130 (0.4%) | 0.03 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 10,392 (4.0%) | 1,354 (3.9%) | 10,392 (4.0%) | 1,354 (3.9%) | 0.01 |
| Region (lumping missing&other category with West) | | | | | | | | | |
| Northeast; n (%) | 11,368 (12.2%) | 1,714 (8.0%) | 19,209 (19.4%) | 4,647 (17.3%) | 49,085 (19.0%) | 5,891 (16.8%) | 79,662 (17.7%) | 12,252 (14.7%) | 0.08 |
| South; n (%) | 46,486 (50.0%) | 11,429 (53.5%) | 21,785 (22.0%) | 4,977 (18.5%) | 109,273 (42.2%) | 15,802 (45.0%) | 177,544 (39.4%) | 32,208 (38.6%) | 0.02 |
| Midwest; n (%) | 16,955 (18.2%) | 4,613 (21.6%) | 46,018 (46.5%) | 14,463 (53.7%) | 55,845 (21.6%) | 7,955 (22.7%) | 118,818 (26.4%) | 27,031 (32.4%) | -0.13 |
| West; n (%) | 18,164 (19.5%) | 3,590 (16.8%) | 10,722 (10.8%) | 2,533 (9.4%) | 44,591 (17.2%) | 5,467 (15.6%) | 73,477 (16.3%) | 11,590 (13.9%) | 0.07<br>0.02 |
| Unknown+missing; n (%) CV Covariates | N/A | N/A | 1,241 (1.3%) | 290 (1.1%) | N/A | N/A | 1,241 (1.3%) | 290 (1.1%) | 0.02 |
| Ischemic heart disease; n (%) | 17,210 (18.5%) | 3,092 (14.5%) | 13,876 (14.0%) | 3,306 (12.3%) | 67,253 (26.0%) | 8,851 (25.2%) | 98,339 (21.8%) | 15,249 (18.3%) | 0.09 |
| Acute MI; n (%) | 350 (0.4%) | 57 (0.3%) | 321 (0.3%) | 68 (0.3%) | 1,182 (0.5%) | 123 (0.4%) | 1,853 (0.4%) | 248 (0.3%) | 0.02 |
| ACS/unstable angina; n (%) | 438 (0.5%) | 95 (0.4%) | 398 (0.4%) | 103 (0.4%) | 1,445 (0.6%) | 184 (0.5%) | 2,281 (0.5%) | 382 (0.5%) | 0.00 |
| Old MI; n (%) | 2,139 (2.3%) | 367 (1.7%) | 995 (1.0%) | 200 (0.7%) | 7,156 (2.8%) | 875 (2.5%) | 10,290 (2.3%) | 1,442 (1.7%) | 0.04 |
| Stable angina; n (%) | 2,635 (2.8%) | 432 (2.0%) | 1,655 (1.7%) | 351 (1.3%) | 7,598 (2.9%) | 989 (2.8%) | 11,888 (2.6%) | 1,772 (2.1%) | 0.03 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 16,133 (17.4%) | 2,910 (13.6%) | 13,142 (13.3%) | 3,136 (11.7%) | 64,446 (24.9%) | 8,516 (24.3%) | 93,721 (20.8%) | 14,562 (17.5%) | 0.08 |
| Other atherosclerosis with ICD10; n (%) | 595 (0.6%) | 96 (0.4%) | 566 (0.6%) | 150 (0.6%) | 3,406 (1.3%) | 400 (1.1%) | 4,567 (1.0%) | 646 (0.8%) | 0.08 |
| other differences with rep 10 , in (10) | 333 (0.070) | 30 (0.170) | 300 (0.070) | 150 (0.070) | 3,100 (2.370) | 100 (1.170) | 1,507 (2.070) | 0.10 (0.070) | 0.02 |
| Previous cardiac procedure (CABG or PTCA or Stent); n (%) | 153 (0.2%) | 27 (0.1%) | 165 (0.2%) | 38 (0.1%) | 410 (0.2%) | 70 (0.2%) | #VALUE! | 135 (0.2%) | #VALUE! |
| History of CABG or PTCA; n (%) | 3,786 (4.1%) | 645 (3.0%) | 1,733 (1.8%) | 389 (1.4%) | 16,353 (6.3%) | 2,097 (6.0%) | 21,872 (4.9%) | 3,131 (3.8%) | 0.05 |
| Any stroke; n (%) | 3,557 (3.8%) | 526 (2.5%) | 2,842 (2.9%) | 511 (1.9%) | 15,686 (6.1%) | 1,822 (5.2%) | 22,085 (4.9%) | 2,859 (3.4%) | 0.08 |
| Ischemic stroke (w and w/o mention of cerebral infarction); n (%) | 3,535 (3.8%) | 524 (2.5%) | 2,824 (2.9%) | 508 (1.9%) | 15,576 (6.0%) | 1,817 (5.2%) | 21,935 (4.9%) | 2,849 (3.4%) | 0.08 |
| Hemorrhagic stroke; n (%) | 40 (0.0%) | 5 (0.0%) | 30 (0.0%) | 4 (0.0%) | 13,370 (0.0%) | 1,817 (3.2/6) | 21,535 (4.5%) | 2,043 (3.470) | ** |
| TIA; n (%) | 406 (0.4%) | 63 (0.3%) | 318 (0.3%) | 55 (0.2%) | 1,670 (0.6%) | 173 (0.5%) | 2,394 (0.5%) | 291 (0.3%) | 0.03 |
| Other cerebrovascular disease; n (%) | 974 (1.0%) | 135 (0.6%) | 632 (0.6%) | 97 (0.4%) | 4,269 (1.6%) | 353 (1.0%) | 5,875 (1.3%) | 585 (0.7%) | 0.06 |
| Late effects of cerebrovascular disease; n (%) | 950 (1.0%) | 98 (0.5%) | 398 (0.4%) | 67 (0.2%) | 3,602 (1.4%) | 261 (0.7%) | 4,950 (1.1%) | 426 (0.5%) | 0.07 |
| Cerebrovascular procedure; n (%) | 34 (0.0%) | 7 (0.0%) | 41 (0.0%) | 4 (0.0%) | 133 (0.1%) | 18 (0.1%) | 208 (0.0%) | 29 (0.0%) | #DIV/0! |
| Heart failure (CHF); n (%) | 6,529 (7.0%) | 824 (3.9%) | 3,776 (3.8%) | 566 (2.1%) | 25,130 (9.7%) | 2,306 (6.6%) | 35,435 (7.9%) | 3,696 (4.4%) | 0.15 |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n (%) | 6,053 (6.5%) | 924 (4.3%) | 3,642 (3.7%) | 717 (2.7%) | 25,306 (9.8%) | 2,686 (7.6%) | 35,001 (7.8%) | 4,327 (5.2%) | 0.11 |
| Atrial fibrillation; n (%) | 5,948 (6.4%) | 916 (4.3%) | 4,563 (4.6%) | 792 (2.9%) | 27,072 (10.5%) | 3,013 (8.6%) | 37,583 (8.3%) | 4,721 (5.7%) | 0.10 |
| Other cardiac dysrhythmia; n (%) | 7,501 (8.1%) | 1,129 (5.3%) | 5,013 (5.1%) | 865 (3.2%) | 29,407 (11.4%) | 3,368 (9.6%) | 41,921 (9.3%) | 5,362 (6.4%) | 0.11 |
| Cardiac conduction disorders; n (%) | 2,036 (2.2%) | 285 (1.3%) | 1,360 (1.4%) | 246 (0.9%) | 8,527 (3.3%) | 956 (2.7%) | 11,923 (2.6%) | 1,487 (1.8%) | 0.05 |
| Other CVD; n (%) | 8,272 (8.9%) | 1,281 (6.0%) | 6,502 (6.6%) | 1,292 (4.8%) | 33,542 (13.0%) | 3,782 (10.8%) | 48,316 (10.7%) | 6,355 (7.6%) | 0.11 |
| Diabetes-related complications | | | | | | 2 602 /= ==// | 20.000 10.000 | | |
| Diabetic retinopathy; n (%) | 6,055 (6.5%) | 1,287 (6.0%) | 3,395 (3.4%) | 1,172 (4.4%) | 17,502 (6.8%) | 2,693 (7.7%) | 26,952 (6.0%) | 5,152 (6.2%) | -0.01 |
| Diabetes with other ophthalmic manifestations; n (%) Retinal detachment, vitreous hemorrhage, vitrectomy; n | 808 (0.9%) | 139 (0.7%) | 2,103 (2.1%) | 739 (2.7%) | 6,484 (2.5%) | 992 (2.8%) | 9,395 (2.1%) | 1,870 (2.2%) | -0.01 |
| (%) | 350 (0.4%) | 80 (0.4%) | 288 (0.3%) | 77 (0.3%) | 908 (0.4%) | 149 (0.4%) | 1,546 (0.3%) | 306 (0.4%) | -0.02 |
| Retinal laser coagulation therapy; n (%) | 483 (0.5%) | 122 (0.6%) | 451 (0.5%) | 148 (0.5%) | 1,384 (0.5%) | 225 (0.6%) | 2,318 (0.5%) | 495 (0.6%) | -0.01 |
| Occurrence of Diabetic Neuropathy ; n (%) | 16,540 (17.8%) | 3,792 (17.8%) | 9,680 (9.8%) | 3,123 (11.6%) | 44,854 (17.3%) | 7,033 (20.0%) | 71,074 (15.8%) | 13,948 (16.7%) | -0.02 |

| Occurrence of diabetic nephropathy with ICD10; n (%) | 15,236 (16.4%) | 2,186 (10.2%) | 6,571 (6.6%) | 1,538 (5.7%) | 28,980 (11.2%) | 2,914 (8.3%) | 50,787 (11.3%) | 6,638 (8.0%) | 0.11 |
|---|---|---|---|---|---|---|---|---|---|
| Hypoglycemia ; n (%) | 1,930 (2.1%) | 459 (2.2%) | 1,787 (1.8%) | 678 (2.5%) | 6,000 (2.3%) | 829 (2.4%) | 9,717 (2.2%) | 1,966 (2.4%) | -0.01 |
| Hyperglycemia; n (%) | 3,471 (3.7%) | 661 (3.1%) | 2,989 (3.0%) | 672 (2.5%) | 10,518 (4.1%) | 1,135 (3.2%) | 16,978 (3.8%) | 2,468 (3.0%) | 0.04 |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 5,638 (6.1%) | 681 (3.2%) | 3,600 (3.6%) | 582 (2.2%) | 18,043 (7.0%) | 1,435 (4.1%) | 27,281 (6.1%) | 2,698 (3.2%) | 0.14 |
| Diabetic ketoacidosis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 00 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome | 0 (0.070) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 000 (0.070) | 00 (0.070) | #514/0: |
| (HONK); n (%) | 460 (0.5%) | 97 (0.5%) | 402 (0.4%) | 92 (0.3%) | 1,230 (0.5%) | 172 (0.5%) | 2,092 (0.5%) | 361 (0.4%) | 0.01 |
| Diabetes with peripheral circulatory disorders with ICD- | 100 (0.07-) | () | (0, | ( | _, (0.07.7) | | _,=== (=:=, | ( | |
| 10 ; n (%) | 6,454 (6.9%) | 1,015 (4.8%) | 2,805 (2.8%) | 698 (2.6%) | 17,985 (6.9%) | 2,091 (6.0%) | 27,244 (6.0%) | 3,804 (4.6%) | 0.06 |
| Diabetic Foot; n (%) | 1,580 (1.7%) | 286 (1.3%) | 1,274 (1.3%) | 345 (1.3%) | 5,641 (2.2%) | 715 (2.0%) | 8,495 (1.9%) | 1,346 (1.6%) | 0.02 |
| Gangrene ; n (%) | 133 (0.1%) | 20 (0.1%) | 74 (0.1%) | 10 (0.0%) | 347 (0.1%) | 28 (0.1%) | 554 (0.1%) | 58 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 492 (0.5%) | 63 (0.3%) | 134 (0.1%) | 32 (0.1%) | 1,170 (0.5%) | 109 (0.3%) | 1,796 (0.4%) | 204 (0.2%) | 0.04 |
| Osteomyelitis; n (%) | 356 (0.4%) | 53 (0.2%) | 266 (0.3%) | 67 (0.2%) | 910 (0.4%) | 98 (0.3%) | 1,532 (0.3%) | 218 (0.3%) | 0.00 |
| Skin infections ; n (%) | 4,261 (4.6%) | 989 (4.6%) | 4,253 (4.3%) | 1,163 (4.3%) | 14,883 (5.8%) | 1,984 (5.7%) | 23,397 (5.2%) | 4,136 (5.0%) | 0.01 |
| Erectile dysfunction; n (%) | 2,518 (2.7%) | 767 (3.6%) | 2,415 (2.4%) | 759 (2.8%) | 5,288 (2.0%) | 1,093 (3.1%) | 10,221 (2.3%) | 2,619 (3.1%) | -0.05 |
| Diabetes with unspecified complication; n (%) | 4,841 (5.2%) | 1,089 (5.1%) | 4,301 (4.3%) | 1,170 (4.3%) | 12,495 (4.8%) | 1,873 (5.3%) | 21,637 (4.8%) | 4,132 (5.0%) | -0.01 |
| Diabetes mellitus without mention of complications; n | | | | | | | | | |
| (%) | 79,354 (85.4%) | 18,017 (84.4%) | 90,348 (91.3%) | 24,734 (91.9%) | 239,419 (92.5%) | 32,095 (91.4%) | 409,121 (90.8%) | 74,846 (89.8%) | 0.03 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 86,092 (92.6%) | 19,597 (91.8%) | 85,616 (86.5%) | 23,560 (87.6%) | 247,659 (95.7%) | 33,591 (95.7%) | 419,367 (93.0%) | 76,748 (92.1%) | 0.03 |
| Hyperlipidemia ; n (%) | 69,860 (75.1%) | 16,586 (77.7%) | 70,415 (71.1%) | 20,473 (76.1%) | 205,187 (79.3%) | 28,928 (82.4%) | 345,462 (76.6%) | 65,987 (79.1%) | -0.06 |
| Edema; n (%) | 5,759 (6.2%) | 984 (4.6%) | 3,668 (3.7%) | 862 (3.2%) | 22,340 (8.6%) | 2,520 (7.2%) | 31,767 (7.0%) | 4,366 (5.2%) | 0.08 |
| Renal Dysfunction (non-diabetic) ; n (%) | 20,147 (21.7%) | 2,104 (9.9%) | 10,409 (10.5%) | 1,423 (5.3%) | 56,908 (22.0%) | 4,185 (11.9%) | 87,464 (19.4%) | 7,712 (9.3%) | 0.29 |
| Occurrence of acute renal disease ; n (%) | 2,464 (2.7%) | 173 (0.8%) | 1,510 (1.5%) | 132 (0.5%) | 7,853 (3.0%) | 371 (1.1%) | 11,827 (2.6%) | 676 (0.8%) | 0.14 |
| Occurrence of chronic renal insufficiency; n (%) | 17,268 (18.6%) | 1,743 (8.2%) | 7,789 (7.9%) | 1,056 (3.9%) | 48,344 (18.7%) | 3,461 (9.9%) | 73,401 (16.3%) | 6,260 (7.5%) | 0.27 |
| Chronic kidney disease ; n (%) | 16,746 (18.0%) | 1,620 (7.6%) | 7,378 (7.5%) | 898 (3.3%) | 46,107 (17.8%) | 3,184 (9.1%) | 70,231 (15.6%) | 5,702 (6.8%) | 0.28 |
| CKD Stage 3-4; n (%) | 11,687 (12.6%) | 834 (3.9%) | 4,947 (5.0%) | 451 (1.7%) | 32,580 (12.6%) | 1,859 (5.3%) | 49,214 (10.9%) | 3,144 (3.8%) | 0.27 |
| Occurrence of hypertensive nephropathy; n (%) | 7,429 (8.0%) | 682 (3.2%) | 3,128 (3.2%) | 368 (1.4%) | 19,295 (7.5%) | 1,185 (3.4%) | 29,852 (6.6%) | 2,235 (2.7%) | 0.19 |
| Occurrence of miscellaneous renal insufficiency; n (%) | 4,104 (4.4%) | 422 (2.0%) | 2,795 (2.8%) | 398 (1.5%) | 15,575 (6.0%) | 1,163 (3.3%) | 22,474 (5.0%) | 1,983 (2.4%) | 0.14 |
| Glaucoma or cataracts; n (%) | 18,671 (20.1%) | 3,608 (16.9%) | 14,922 (15.1%) | 3,666 (13.6%) | 68,628 (26.5%) | 9,616 (27.4%) | 102,221 (22.7%) | 16,890 (20.3%) | 0.06 |
| Cellulitis or abscess of toe; n (%) | 1,051 (1.1%) | 190 (0.9%) | 740 (0.7%) | 166 (0.6%) | 3,049 (1.2%) | 385 (1.1%) | 4,840 (1.1%) | 741 (0.9%) | 0.02 |
| Foot ulcer; n (%) | 1,516 (1.6%) | 268 (1.3%) | 1,254 (1.3%) | 347 (1.3%) | 5,567 (2.2%) | 708 (2.0%) | 8,337 (1.8%) | 1,323 (1.6%) | 0.02 |
| Bladder stones; n (%) | 99 (0.1%) | 12 (0.1%) | 86 (0.1%) | 12 (0.0%) | 343 (0.1%) | 50 (0.1%) | 528 (0.1%) | 74 (0.1%) | 0.00 |
| Kidney stones; n (%) | 1,802 (1.9%) | 330 (1.5%) | 1,911 (1.9%) | 471 (1.8%) | 5,922 (2.3%) | 763 (2.2%) | 9,635 (2.1%) | 1,564 (1.9%) | 0.01 |
| Urinary tract infections (UTIs); n (%) | 7,598 (8.2%) | 1,041 (4.9%) | 5,074 (5.1%) | 1,047 (3.9%) | 30,499 (11.8%) | 2,805 (8.0%) | 43,171 (9.6%) | 4,893 (5.9%) | 0.14 |
| Dipstick urinalysis; n (%) | 33,076 (35.6%) | 6,473 (30.3%) | 30,675 (31.0%) | 8,063 (30.0%) | 99,731 (38.5%) | 12,329 (35.1%) | 163,482 (36.3%) | 26,865 (32.2%) | 0.09 |
| Non-dipstick urinalysis; n (%) | 41,645 (44.8%) | 9,752 (45.7%) | 36,404 (36.8%) | 11,482 (42.7%) | 111,191 (43.0%) | 16,168 (46.0%) | 189,240 (42.0%) | 37,402 (44.9%) | -0.06 |
| Urine function test; n (%) | 1,859 (2.0%) | 275 (1.3%) | 1,802 (1.8%) | 345 (1.3%) | 7,703 (3.0%) | 906 (2.6%) | 11,364 (2.5%) | 1,526 (1.8%) | 0.05 |
| Cytology; n (%) | 537 (0.6%) | 88 (0.4%) | 639 (0.6%) | 126 (0.5%) | 2,033 (0.8%) | 220 (0.6%) | 3,209 (0.7%) | 434 (0.5%) | 0.03 |
| Cystos; n (%) | 820 (0.9%) | 135 (0.6%) | 855 (0.9%) | 185 (0.7%) | 2,921 (1.1%) | 335 (1.0%) | 4,596 (1.0%) | 655 (0.8%) | 0.02 |
| Other Covariates | 0 (0 00/) | 0 (0 00/) | 0 (0 00/) | 0 (0 00() | 0 (0.0%) | 0 (0 0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Liver disease; n (%) | 0 (0.0%)<br>11,742 (12.6%) | 0 (0.0%)<br>2,168 (10.2%) | 0 (0.0%)<br>7,946 (8.0%) | 0 (0.0%)<br>1,907 (7.1%) | 45,826 (17.7%) | 0 (0.0%)<br>5,609 (16.0%) | #VALUE!<br>65,514 (14.5%) | 9,684 (11.6%) | #VALUE!<br>0.09 |
| Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n | 11,742 (12.0%) | 2,100 (10.2%) | 7,940 (6.0%) | 1,907 (7.170) | 45,020 (17.7%) | 3,009 (10.0%) | 05,514 (14.5%) | 9,004 (11.0%) | 0.09 |
| (%) | 27,439 (29.5%) | 5,725 (26.8%) | 24,107 (24.4%) | 6,419 (23.9%) | 94,733 (36.6%) | 11,953 (34.0%) | 146,279 (32.5%) | 24,097 (28.9%) | 0.08 |
| Dorsopathies; n (%) | 16,535 (17.8%) | 3,757 (17.6%) | 14,621 (14.8%) | 4,093 (15.2%) | 55,400 (21.4%) | 7,711 (22.0%) | 86,556 (19.2%) | 15,561 (18.7%) | 0.01 |
| Fractures; n (%) | 2,037 (2.2%) | 322 (1.5%) | 1,777 (1.8%) | 385 (1.4%) | 7,550 (2.9%) | 772 (2.2%) | 11,364 (2.5%) | 1,479 (1.8%) | 0.05 |
| Falls; n (%) | 2,630 (2.8%) | 343 (1.6%) | 955 (1.0%) | 136 (0.5%) | 9,355 (3.6%) | 716 (2.0%) | 12,940 (2.9%) | 1,195 (1.4%) | 0.10 |
| Osteoporosis; n (%) | 4,528 (4.9%) | 507 (2.4%) | 1,890 (1.9%) | 297 (1.1%) | 19,484 (7.5%) | 1,793 (5.1%) | 25,902 (5.7%) | 2,597 (3.1%) | 0.13 |
| Hyperthyroidism; n (%) | 607 (0.7%) | 115 (0.5%) | 493 (0.5%) | 105 (0.4%) | 2,277 (0.9%) | 255 (0.7%) | 3,377 (0.7%) | 475 (0.6%) | 0.01 |
| Hypothyroidism ; n (%) | 14,093 (15.2%) | 3,015 (14.1%) | 11,014 (11.1%) | 3,225 (12.0%) | 31,705 (12.3%) | 4,238 (12.1%) | 56,812 (12.6%) | 10,478 (12.6%) | 0.00 |
| Other disorders of thyroid gland; n (%) | 3,204 (3.4%) | 782 (3.7%) | 2,893 (2.9%) | 984 (3.7%) | 9,716 (3.8%) | 1,454 (4.1%) | 15,813 (3.5%) | 3,220 (3.9%) | -0.02 |
| Depression; n (%) | 6,370 (6.9%) | 1,494 (7.0%) | 5,344 (5.4%) | 1,597 (5.9%) | 22,933 (8.9%) | 2,897 (8.3%) | 34,647 (7.7%) | 5,988 (7.2%) | 0.02 |
| Anxiety; n (%) | 6,068 (6.5%) | 1,357 (6.4%) | 4,637 (4.7%) | 1,230 (4.6%) | 18,829 (7.3%) | 2,345 (6.7%) | 29,534 (6.6%) | 4,932 (5.9%) | 0.03 |
| Sleep_Disorder; n (%) | 4,861 (5.2%) | 1,601 (7.5%) | 7,480 (7.6%) | 3,032 (11.3%) | 16,931 (6.5%) | 2,968 (8.5%) | 29,272 (6.5%) | 7,601 (9.1%) | -0.10 |
| Dementia; n (%) | 3,192 (3.4%) | 200 (0.9%) | 1,443 (1.5%) | 119 (0.4%) | 16,772 (6.5%) | 910 (2.6%) | 21,407 (4.7%) | 1,229 (1.5%) | 0.19 |
| Delirium; n (%) | 725 (0.8%) | 57 (0.3%) | 410 (0.4%) | 31 (0.1%) | 3,458 (1.3%) | 182 (0.5%) | 4,593 (1.0%) | 270 (0.3%) | 0.09 |
| Psychosis; n (%) | 831 (0.9%) | 88 (0.4%) | 440 (0.4%) | 52 (0.2%) | 4,373 (1.7%) | 258 (0.7%) | 5,644 (1.3%) | 398 (0.5%) | 0.08 |
| Obesity; n (%) | 18,832 (20.3%) | 5,799 (27.2%) | 14,581 (14.7%) | 5,276 (19.6%) | 34,677 (13.4%) | 6,927 (19.7%) | 68,090 (15.1%) | 18,002 (21.6%) | -0.17 |
| Overweight; n (%) | 5,629 (6.1%) | 1,083 (5.1%) | 2,441 (2.5%) | 593 (2.2%) | 9,232 (3.6%) | 1,237 (3.5%) | 17,302 (3.8%) | 2,913 (3.5%) | 0.02 |
| Smoking; n (%) | 8,487 (9.1%) | 1,743 (8.2%) | 5,746 (5.8%) | 1,323 (4.9%) | 28,073 (10.8%) | 3,758 (10.7%) | 42,306 (9.4%) | 6,824 (8.2%) | 0.04 |
| Alcohol abuse or dependence; n (%) | 16 (0.0%) | 2 (0.0%) | 22 (0.0%) | 5 (0.0%) | ** | ** | ** | ** | ** |
| Drug abuse or dependence; n (%) | 41 (0.0%) | 7 (0.0%) | 13 (0.0%) | 3 (0.0%) | | | | | |
| COPD; n (%) | 6,608 (7.1%) | 1,038 (4.9%) | 3,790 (3.8%) | 766 (2.8%) | 23,441 (9.1%) | 2,714 (7.7%) | 33,839 (7.5%) | 4,518 (5.4%) | 0.09 |

| Asthma; n (%) | 4,366 (4.7%) | 934 (4.4%) | 3,552 (3.6%) | 957 (3.6%) | 13,189 (5.1%) | 1,815 (5.2%) | 21,107 (4.7%) | 3,706 (4.4%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 7,604 (8.2%) | 2,530 (11.9%) | 8,904 (9.0%) | 3,255 (12.1%) | 15,485 (6.0%) | 3,345 (9.5%) | 31,993 (7.1%) | 9,130 (11.0%) | -0.14 |
| Pneumonia; n (%) | 1,613 (1.7%) | 234 (1.1%) | 1,356 (1.4%) | 241 (0.9%) | 6,178 (2.4%) | 541 (1.5%) | 9,147 (2.0%) | 1,016 (1.2%) | 0.06 |
| Imaging; n (%) | 34 (0.0%) | 6 (0.0%) | 21 (0.0%) | 2 (0.0%) | ** | ** | ** | ** | ** |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 513 (0.6%) | 116 (0.5%) | 358 (0.4%) | 99 (0.4%) | 1,637 (0.6%) | 273 (0.8%) | 2,508 (0.6%) | 488 (0.6%) | 0.00 |
| DM Medications - Glitazones; n (%) | 7,470 (8.0%) | 2,132 (10.0%) | 7,539 (7.6%) | 2,659 (9.9%) | 20,110 (7.8%) | 3,517 (10.0%) | 35,119 (7.8%) | 8,308 (10.0%) | -0.08 |
| | 15,209 (16.4%) | 5,869 (27.5%) | 13,275 (13.4%) | 8,133 (30.2%) | 44,262 (17.1%) | 11,188 (31.9%) | 72,746 (16.1%) | 25,190 (30.2%) | -0.34 |
| DM Medications - Insulin; n (%) | | | | | | | | | |
| DM Medications - Meglitinides; n (%) | 1,069 (1.1%) | 220 (1.0%) | 1,218 (1.2%) | 346 (1.3%) | 4,683 (1.8%) | 576 (1.6%) | 6,970 (1.5%) | 1,142 (1.4%) | 0.01 |
| DM Medications - Metformin; n (%) | 68,898 (74.1%) | 16,690 (78.2%) | 78,748 (79.6%) | 21,017 (78.1%) | 181,431 (70.1%) | 26,156 (74.5%) | 329,077 (73.0%) | 63,863 (76.6%) | -0.08 |
| Concomitant initiation or current use of 2nd Generation | | | | | | | | | |
| SUs; n (%) | 33,158 (35.7%) | 6,949 (32.6%) | 31,388 (31.7%) | 8,362 (31.1%) | 97,534 (37.7%) | 13,082 (37.3%) | 162,080 (36.0%) | 28,393 (34.1%) | 0.04 |
| Concomitant initiation or current use of AGIs; n (%) | 378 (0.4%) | 82 (0.4%) | 250 (0.3%) | 54 (0.2%) | 1,197 (0.5%) | 180 (0.5%) | 1,825 (0.4%) | 316 (0.4%) | 0.00 |
| Concomitant initiation or current use of Glitazones; n (%) | 5,771 (6.2%) | 1,613 (7.6%) | 5,925 (6.0%) | 2,013 (7.5%) | 15,535 (6.0%) | 2,693 (7.7%) | 27,231 (6.0%) | 6,319 (7.6%) | -0.06 |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 1,826 (2.0%) | 2,913 (13.6%) | 2,187 (2.2%) | 4,565 (17.0%) | 3,172 (1.2%) | 4,049 (11.5%) | 7,185 (1.6%) | 11,527 (13.8%) | -0.47 |
| | _,, | _,=== (=====, | _,, | ., (= , | -/ () | 1,0 10 (==10,1) | 1,200 (21011) | ,, | |
| Concomitant initiation or current use of Insulin; n (%) | 11,555 (12.4%) | 4,411 (20.7%) | 10,019 (10.1%) | 6,296 (23.4%) | 34,079 (13.2%) | 8,819 (25.1%) | 55,653 (12.3%) | 19,526 (23.4%) | -0.29 |
| | 11,555 (12.4%) | 4,411 (20.7%) | 10,019 (10.1%) | 0,290 (23.4%) | 34,079 (13.2%) | 0,019 (23.1%) | 33,033 (12.3%) | 19,320 (23.4%) | -0.29 |
| Concomitant initiation or current use of Meglitinides; n | 705 (0.00() | 1.12 (0.70) | 075 (0.00() | 222 (0.00() | 2 440 (4 20() | 402 (4 40() | 5 074 (4 40() | 766 (0.00() | 0.00 |
| (%) | 786 (0.8%) | 142 (0.7%) | 875 (0.9%) | 222 (0.8%) | 3,410 (1.3%) | 402 (1.1%) | 5,071 (1.1%) | 766 (0.9%) | 0.02 |
| Concomitant initiation or current use of Metformin; n (%) | 59,526 (64.0%) | 14,098 (66.0%) | 69,344 (70.1%) | 17,788 (66.1%) | 156,339 (60.4%) | 22,344 (63.6%) | 285,209 (63.3%) | 54,230 (65.0%) | -0.04 |
| Past use of 2nd Generation SUs ; n (%) | 6,990 (7.5%) | 1,805 (8.5%) | 7,050 (7.1%) | 2,003 (7.4%) | 19,774 (7.6%) | 2,765 (7.9%) | 33,814 (7.5%) | 6,573 (7.9%) | -0.02 |
| Past use of AGIs ; n (%) | 135 (0.1%) | 34 (0.2%) | 108 (0.1%) | 45 (0.2%) | 440 (0.2%) | 93 (0.3%) | 683 (0.2%) | 172 (0.2%) | 0.00 |
| Past use of Glitazones; n (%) | 1,699 (1.8%) | 519 (2.4%) | 1,614 (1.6%) | 646 (2.4%) | 4,575 (1.8%) | 824 (2.3%) | 7,888 (1.8%) | 1,989 (2.4%) | -0.04 |
| Past use of GLP-1 RA; n (%) | 1,513 (1.6%) | 1,248 (5.8%) | 1,750 (1.8%) | 1,865 (6.9%) | 2,968 (1.1%) | 1,792 (5.1%) | 6,231 (1.4%) | 4,905 (5.9%) | -0.24 |
| Past use of Insulin ; n (%) | 3,654 (3.9%) | 1,458 (6.8%) | 3,257 (3.3%) | 1,837 (6.8%) | 10,185 (3.9%) | 2,370 (6.7%) | 17,096 (3.8%) | 5,665 (6.8%) | -0.13 |
| Past use of Meglitinides ; n (%) | 283 (0.3%) | 78 (0.4%) | 343 (0.3%) | 124 (0.5%) | 1,273 (0.5%) | 174 (0.5%) | 1,899 (0.4%) | 376 (0.5%) | -0.01 |
| | | | | | | | | | -0.01 |
| Past use of metformin (final); n (%) | 9,372 (10.1%) | 2,592 (12.1%) | 9,405 (9.5%) | 3,229 (12.0%) | 25,092 (9.7%) | 3,812 (10.9%) | 43,869 (9.7%) | 9,633 (11.6%) | -0.06 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 48,661 (52.3%) | 11,586 (54.3%) | 52,091 (52.6%) | 14,264 (53.0%) | 126,600 (48.9%) | 17,572 (50.0%) | 227,352 (50.4%) | 43,422 (52.1%) | -0.03 |
| Use of ARBs; n (%) | 33,271 (35.8%) | 7,711 (36.1%) | 35,863 (36.2%) | 10,233 (38.0%) | 92,288 (35.7%) | 13,134 (37.4%) | 161,422 (35.8%) | 31,078 (37.3%) | -0.03 |
| Use of Loop Diuretics ; n (%) | 11,784 (12.7%) | 1,942 (9.1%) | 9,018 (9.1%) | 2,198 (8.2%) | 47,353 (18.3%) | 5,440 (15.5%) | 68,155 (15.1%) | 9,580 (11.5%) | 0.11 |
| Use of other diuretics; n (%) | 2,738 (2.9%) | 549 (2.6%) | 2,657 (2.7%) | 689 (2.6%) | 9,268 (3.6%) | 1,194 (3.4%) | 14,663 (3.3%) | 2,432 (2.9%) | 0.02 |
| Use of nitrates-United; n (%) | 4,319 (4.6%) | 759 (3.6%) | 3,623 (3.7%) | 874 (3.2%) | 18,544 (7.2%) | 2,233 (6.4%) | 26,486 (5.9%) | 3,866 (4.6%) | 0.06 |
| Use of other hypertension drugs; n (%) | 7,149 (7.7%) | 1,137 (5.3%) | 5,872 (5.9%) | 1,298 (4.8%) | 22,836 (8.8%) | 2,590 (7.4%) | 35,857 (8.0%) | 5,025 (6.0%) | 0.08 |
| | 1,454 (1.6%) | 242 (1.1%) | | 236 (0.9%) | 7,836 (3.0%) | 768 (2.2%) | 10,654 (2.4%) | 1,246 (1.5%) | 0.07 |
| Use of digoxin; n (%) | | | 1,364 (1.4%) | | | | | | |
| Use of Anti-arrhythmics; n (%) | 1,053 (1.1%) | 173 (0.8%) | 1,025 (1.0%) | 190 (0.7%) | 4,813 (1.9%) | 503 (1.4%) | 6,891 (1.5%) | 866 (1.0%) | 0.05 |
| Use of COPD/asthma meds; n (%) | 13,032 (14.0%) | 2,801 (13.1%) | 13,214 (13.4%) | 3,735 (13.9%) | 41,359 (16.0%) | 5,761 (16.4%) | 67,605 (15.0%) | 12,297 (14.7%) | 0.01 |
| Use of statins; n (%) | 67,725 (72.8%) | 15,590 (73.0%) | 67,262 (68.0%) | 18,843 (70.0%) | 190,375 (73.6%) | 26,610 (75.8%) | 325,362 (72.2%) | 61,043 (73.2%) | -0.02 |
| Use of other lipid-lowering drugs; n (%) | 10,744 (11.6%) | 2,824 (13.2%) | 13,362 (13.5%) | 4,298 (16.0%) | 33,537 (13.0%) | 5,264 (15.0%) | 57,643 (12.8%) | 12,386 (14.9%) | -0.06 |
| Use of antiplatelet agents; n (%) | 10,807 (11.6%) | 2,095 (9.8%) | 11,015 (11.1%) | 2,709 (10.1%) | 37,758 (14.6%) | 4,884 (13.9%) | 59,580 (13.2%) | 9,688 (11.6%) | 0.05 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | | | | |
| Apixaban, Warfarin); n (%) | 5,410 (5.8%) | 923 (4.3%) | 4,601 (4.6%) | 893 (3.3%) | 23,012 (8.9%) | 2,738 (7.8%) | 33,023 (7.3%) | 4,554 (5.5%) | 0.07 |
| Use of heparin and other low-molecular weight heparins; | | , , | , | , , | | , | | | |
| n (%) | 194 (0.2%) | 21 (0.1%) | 8 (0.0%) | 0 (0.0%) | 578 (0.2%) | 66 (0.2%) | 780 (0.2%) | 087 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 13,827 (14.9%) | 3,495 (16.4%) | 15,098 (15.3%) | 4,443 (16.5%) | 39,001 (15.1%) | 5,385 (15.3%) | 67,926 (15.1%) | 13,323 (16.0%) | -0.02 |
| Use of oral corticosteroids; n (%) | 11,453 (12.3%) | 2,456 (11.5%) | 11,415 (11.5%) | 2,993 (11.1%) | 36,129 (14.0%) | 4,819 (13.7%) | 58,997 (13.1%) | 10,268 (12.3%) | 0.02 |
| | | | | | | | | | 0.10 |
| Use of bisphosphonate (United); n (%) | 2,381 (2.6%) | 240 (1.1%) | 1,015 (1.0%) | 162 (0.6%) | 9,128 (3.5%) | 777 (2.2%) | 12,524 (2.8%) | 1,179 (1.4%) | -0.01 |
| Use of opioids; n (%) | 17,277 (18.6%) | 4,109 (19.2%) | 18,342 (18.5%) | 5,363 (19.9%) | 51,367 (19.8%) | 7,046 (20.1%) | 86,986 (19.3%) | 16,518 (19.8%) | |
| Use of antidepressants; n (%) | 19,561 (21.0%) | 4,900 (23.0%) | 18,887 (19.1%) | 6,026 (22.4%) | 59,621 (23.0%) | 8,616 (24.5%) | 98,069 (21.8%) | 19,542 (23.4%) | -0.04 |
| Use of antipsychotics; n (%) | 1,969 (2.1%) | 365 (1.7%) | 1,327 (1.3%) | 303 (1.1%) | 7,692 (3.0%) | 698 (2.0%) | 10,988 (2.4%) | 1,366 (1.6%) | 0.06 |
| Use of anticonvulsants; n (%) | 13,269 (14.3%) | 2,952 (13.8%) | 9,838 (9.9%) | 3,006 (11.2%) | 38,618 (14.9%) | 5,337 (15.2%) | 61,725 (13.7%) | 11,295 (13.5%) | 0.01 |
| Use of lithium; n (%) | 105 (0.1%) | 21 (0.1%) | 107 (0.1%) | 20 (0.1%) | 245 (0.1%) | 29 (0.1%) | 457 (0.1%) | 070 (0.1%) | 0.00 |
| Use of Benzos; n (%) | 8,001 (8.6%) | 1,860 (8.7%) | 7,927 (8.0%) | 2,274 (8.5%) | 26,120 (10.1%) | 3,388 (9.6%) | 42,048 (9.3%) | 7,522 (9.0%) | 0.01 |
| Use of anxiolytics/hypnotics; n (%) | 4,283 (4.6%) | 1,109 (5.2%) | 5,008 (5.1%) | 1,439 (5.3%) | 13,252 (5.1%) | 1,813 (5.2%) | 22,543 (5.0%) | 4,361 (5.2%) | -0.01 |
| Use of dementia meds; n (%) | 2,138 (2.3%) | 130 (0.6%) | 1,145 (1.2%) | 84 (0.3%) | 12,186 (4.7%) | 724 (2.1%) | 15,469 (3.4%) | 938 (1.1%) | 0.16 |
| Use of antiparkinsonian meds; n (%) | 1,865 (2.0%) | 401 (1.9%) | 1,487 (1.5%) | 438 (1.6%) | 7,223 (2.8%) | 996 (2.8%) | 10,575 (2.3%) | 1,835 (2.2%) | 0.01 |
| | | | 14 (0.0%) | | | | | | -0.04 |
| Any use of pramlintide; n (%) | 6 (0.0%) | 27 (0.1%) | , , | 51 (0.2%) | 26 (0.0%) | 36 (0.1%) | 046 (0.0%) | 114 (0.1%) | -0.04 |
| Any use of 1st generation sulfonylureas; n (%) | 6 (0.0%) | 0 (0.0%) | 11 (0.0%) | 0 (0.0%) | | ** | ** | ** | |
| Entresto (sacubitril/valsartan); n (%) | 133 (0.1%) | 14 (0.1%) | 40 (0.0%) | 4 (0.0%) | 153 (0.1%) | 13 (0.0%) | 326 (0.1%) | 031 (0.0%) | 0.00 |
| Initiation as monotherapy ; n (%) | 8,025 (8.6%) | 1,196 (5.6%) | 8,499 (8.6%) | 1,307 (4.9%) | 19,281 (7.5%) | 1,217 (3.5%) | 35,805 (7.9%) | 3,720 (4.5%) | 0.14 |
| Labs | | | | | | | 191,948 | 48,256 | |
| Lab values- HbA1c (%); n (%) | 39,394 (42.4%) | 9,243 (43.3%) | 6,873 (6.9%) | 1,671 (6.2%) | N/A | N/A | 46,267 (24.1%) | 10,914 (22.6%) | 0.04 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 31,798 (34.2%) | 7,578 (35.5%) | 5,566 (5.6%) | 1,424 (5.3%) | N/A | N/A | 37,364 (19.5%) | 9,002 (18.7%) | 0.02 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 39,394 (42.4%) | 9,243 (43.3%) | 6,873 (6.9%) | 1,671 (6.2%) | N/A | N/A | 46,267 (24.1%) | 10,914 (22.6%) | 0.04 |
| | | -, -(, | -, (, | ,. = \/ | ,/* | | -, (,-) | -,- (==/ | |

| Lab values- BNP; n (%) | 754 (0.8%) | 133 (0.6%) | 105 (0.1%) | 4 (0.0%) | N/A | N/A | 859 (0.4%) | 137 (0.3%) | 0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP (within 3 months); n (%) | 469 (0.5%) | 82 (0.4%) | 73 (0.1%) | 3 (0.0%) | N/A | N/A | 542 (0.3%) | 085 (0.2%) | 0.02 |
| Lab values- BNP (within 6 months); n (%) | 754 (0.8%) | 133 (0.6%) | 105 (0.1%) | 4 (0.0%) | N/A | N/A | 859 (0.4%) | 137 (0.3%) | 0.02 |
| Lab values- BUN (mg/dl); n (%) | 39,324 (42.3%) | 9,039 (42.3%) | 6,660 (6.7%) | 1,583 (5.9%) | N/A | N/A | 45,984 (24.0%) | 10,622 (22.0%) | 0.05 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 31,041 (33.4%) | 7,235 (33.9%) | 5,215 (5.3%) | 1,301 (4.8%) | N/A | N/A | 36,256 (18.9%) | 8,536 (17.7%) | 0.03 |
| | 39,324 (42.3%) | | | | N/A | N/A | 45,984 (24.0%) | 10,622 (22.0%) | 0.05 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | . , , | 9,039 (42.3%) | 6,660 (6.7%) | 1,583 (5.9%) | · · | | | | |
| Lab values- Creatinine (mg/dl); n (%) | 40,379 (43.4%) | 9,338 (43.7%) | 7,075 (7.1%) | 1,722 (6.4%) | N/A | N/A | 47,454 (24.7%) | 11,060 (22.9%) | 0.04 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 31,911 (34.3%) | 7,473 (35.0%) | 5,555 (5.6%) | 1,428 (5.3%) | N/A | N/A | 37,466 (19.5%) | 8,901 (18.4%) | 0.03 |
| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 40,379 (43.4%) | 9,338 (43.7%) | 7,075 (7.1%) | 1,722 (6.4%) | N/A | N/A | 47,454 (24.7%) | 11,060 (22.9%) | 0.04 |
| Lab values- HDL level (mg/dl); n (%) | 33,867 (36.4%) | 8,008 (37.5%) | 6,271 (6.3%) | 1,528 (5.7%) | N/A | N/A | 40,138 (20.9%) | 9,536 (19.8%) | 0.03 |
| , G , , , , | , . , | .,, | -, (, | , ( , | • | , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | .,, | |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 25,297 (27.2%) | 6,107 (28.6%) | 4,752 (4.8%) | 1,206 (4.5%) | N/A | N/A | 30,049 (15.7%) | 7,313 (15.2%) | 0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 33,867 (36.4%) | 8,008 (37.5%) | 6,271 (6.3%) | 1,528 (5.7%) | N/A | N/A | 40,138 (20.9%) | 9,536 (19.8%) | 0.03 |
| Lab values- LDL level (mg/dl); n (%) | 34,910 (37.5%) | 8,251 (38.7%) | 6,464 (6.5%) | 1,555 (5.8%) | N/A | N/A | 41,374 (21.6%) | 9,806 (20.3%) | 0.03 |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 26,067 (28.0%) | 6,315 (29.6%) | 4,889 (4.9%) | 1,231 (4.6%) | N/A | N/A | 30,956 (16.1%) | 7,546 (15.6%) | 0.01 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 34,910 (37.5%) | 8,251 (38.7%) | 6,464 (6.5%) | 1,555 (5.8%) | N/A | N/A | 41,374 (21.6%) | 9,806 (20.3%) | 0.03 |
| Lab values- NT-proBNP; n (%) | 109 (0.1%) | 12 (0.1%) | 17 (0.0%) | 0 (0.0%) | N/A | N/A | 126 (0.1%) | 12 (0.0%) | 0.04 |
| Lab values- NT-proBNP (within 3 months); n (%) | 65 (0.1%) | 7 (0.0%) | 12 (0.0%) | 0 (0.0%) | N/A | N/A | 77 (0.0%) | 7 (0.0%) | 0.01 |
| Lab values- NT-proBNP (within 6 months); n (%) | 109 (0.1%) | 12 (0.1%) | 17 (0.0%) | 0 (0.0%) | N/A | N/A | 126 (0.1%) | 12 (0.0%) | |
| Lab values- Total cholesterol (mg/dl); n (%) | 34,343 (36.9%) | 8,172 (38.3%) | 6,281 (6.3%) | 1,541 (5.7%) | N/A | N/A | 40,624 (21.2%) | 9,713 (20.1%) | 0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 months); n | | 6 257 (20 20) | 4.750 (4.00() | 4 222 (4 50() | 21/2 | | 20 452 (45 00() | 7 470 (45 50/) | 0.04 |
| (%) | 25,693 (27.6%) | 6,257 (29.3%) | 4,760 (4.8%) | 1,222 (4.5%) | N/A | N/A | 30,453 (15.9%) | 7,479 (15.5%) | 0.01 |
| Lab values- Total cholesterol (mg/dl) (within 6 months); n | 34,343 (36.9%) | 8,172 (38.3%) | 6,281 (6.3%) | 1,541 (5.7%) | N/A | N/A | 40,624 (21.2%) | 9,713 (20.1%) | 0.03 |
| (%) | | | | | | | | | |
| Lab values-Triglyceride level (mg/dl); n (%) | 34,067 (36.6%) | 8,123 (38.1%) | 6,220 (6.3%) | 1,515 (5.6%) | N/A | N/A | 40,287 (21.0%) | 9,638 (20.0%) | 0.02 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 25,487 (27.4%) | 6,217 (29.1%) | 4,718 (4.8%) | 1,205 (4.5%) | N/A | N/A | 30,205 (15.7%) | 7,422 (15.4%) | 0.01 |
| Lab values- Triglyceride level (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 34,067 (36.6%) | 8,123 (38.1%) | 6,220 (6.3%) | 1,515 (5.6%) | N/A | N/A | 40,287 (21.0%) | 9,638 (20.0%) | 0.02 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 39,196 | 9,185 | 6,611 | 1,615 | N/A | N/A | 45,807 | 10,800 | |
| mean (sd) | 8.25 (1.74) | 8.63 (1.75) | 8.43 (1.84) | 8.63 (1.70) | N/A | N/A | 8.28 (1.75) | 8.63 (1.74) | -0.20 |
| median [IQR] | 7.90 [7.10, 9.10] | 8.30 [7.40, 9.60] | 8.00 [7.10, 9.30] | 8.30 [7.40, 9.60] | N/A | N/A | 7.91 (1.75) | 8.30 (1.74) | -0.22 |
| Missing; n (%) | 53,777 (57.8%) | 12,161 (57.0%) | 92,364 (93.3%) | 25,295 (94.0%) | N/A | N/A | 146,141 (76.1%) | 37,456 (77.6%) | -0.04 |
| Lab result number- BNP mean | 754 | 133 | 105 | 4 | N/A | N/A | 859 | 137 | |
| mean (sd) | 155.94 (289.65) | 91.38 (156.35) | 3,194.66 (27,330.33) | 335.38 (447.47) | N/A | N/A | 527.38 (9530.18) | 98.50 (169.01) | 0.06 |
| median [IQR] | 66.30 [28.18, 168.20] | 42.60 [19.25, 88.20] | 103.50 [36.75, 363.17] | 192.50 [4.25, 809.38] | N/A | N/A | #VALUE! | 46.98 (169.01) | #VALUE! |
| Missing; n (%) | 92,219 (99.2%) | 21,213 (99.4%) | 98,870 (99.9%) | 26,906 (100.0%) | N/A | N/A | 191,089 (99.6%) | 48,119 (99.7%) | -0.02 |
| | . , , | | | | | | | 10.622 | -0.02 |
| Lab result number- BUN (mg/dl) mean | 39,324 | 9,039 | 6,660 | 1,583 | N/A | N/A | 45,984 | | |
| mean (sd) | 18.81 (7.90) | 16.88 (5.75) | 870.71 (12,029.05) | 2,719.95 (20,223.13) | N/A | N/A | 142.19 (4577.70) | 419.72 (7805.66) | -0.04 |
| median [IQR] | 17.00 [14.00, 22.00] | 16.00 [13.00, 19.50] | 16.00 [13.00, 20.00] | 16.00 [13.00, 20.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 53,649 (57.7%) | 12,307 (57.7%) | 92,315 (93.3%) | 25,327 (94.1%) | N/A | N/A | 145,964 (76.0%) | 37,634 (78.0%) | -0.05 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to | | | | | | | | | |
| 15 included) | 40,096 | 9,267 | 6,197 | 1,566 | N/A | N/A | 46,293 | 10,833 | |
| mean (sd) | 1.04 (0.39) | 0.92 (0.24) | 1.00 (0.38) | 0.93 (0.23) | N/A | N/A | 1.03 (0.39) | 0.92 (0.24) | 0.34 |
| median [IQR] | 0.96 [0.79, 1.19] | 0.89 [0.75, 1.04] | 0.95 [0.79, 1.09] | 0.90 [0.77, 1.05] | N/A | N/A | 0.96 (0.39) | 0.89 (0.24) | 0.22 |
| Missing; n (%) | 52,877 (56.9%) | 12,079 (56.6%) | 92,778 (93.7%) | 25,344 (94.2%) | N/A | N/A | 145,655 (75.9%) | 37,423 (77.6%) | -0.04 |
| Lab result number- HDL level (mg/dl) mean (only =<5000 | , (, | ,_, | , (, | | -4 | | = 12,000 (1 01011) | 21,122 (111212) | |
| included) | 33,867 | 8,008 | 6,237 | 1,506 | N/A | N/A | 40,104 | 9,514 | |
| mean (sd) | 46.39 (13.51) | 44.61 (12.78) | 44.36 (39.28) | 42.76 (13.63) | N/A | N/A | 46.07 (19.85) | 44.32 (12.92) | 0.10 |
| | | 43.00 [36.00, 52.00] | | | | N/A | | | 0.10 |
| median [IQR] | 44.00 [37.00, 53.50] | | 43.00 [35.50, 52.00] | 42.00 [35.00, 50.00] | N/A | | 43.84 (19.85) | 42.84 (12.92) | |
| Missing; n (%) | 59,106 (63.6%) | 13,338 (62.5%) | 92,738 (93.7%) | 25,404 (94.4%) | N/A | N/A | 151,844 (79.1%) | 38,742 (80.3%) | -0.03 |
| Lab result number- LDL level (mg/dl) mean (only =<5000 | 22 | 2 | | | | | | 2.22 | |
| included) | 34,168 | 8,115 | 5,889 | 1,378 | N/A | N/A | 40,057 | 9,493 | |
| mean (sd) | 85.70 (38.18) | 83.53 (38.95) | 87.52 (42.90) | 85.68 (40.86) | N/A | N/A | 85.97 (38.91) | 83.84 (39.23) | 0.05 |
| median [IQR] | 83.00 [62.00, 107.00] | 81.50 [60.50, 105.00] | 86.00 [64.00, 112.00] | 85.00 [62.00, 109.00] | N/A | N/A | 83.44 (38.91) | 82.01 (39.23) | 0.04 |
| Missing; n (%) | 58,805 (63.2%) | 13,231 (62.0%) | 93,086 (94.1%) | 25,532 (94.9%) | N/A | N/A | 151,891 (79.1%) | 38,763 (80.3%) | -0.03 |
| Lab result number-Total cholesterol (mg/dl) mean (only | | | | | | | | | |
| =<5000 included) | 34,315 | 8,162 | 6,246 | 1,518 | N/A | N/A | 40,561 | 9,680 | |
| mean (sd) | 171.23 (44.49) | 171.77 (46.18) | 171.78 (54.30) | 171.14 (48.01) | N/A | N/A | 171.31 (46.14) | 171.67 (46.47) | -0.01 |
| median [IQR] | 165.00 [141.00, 195.00] | 166.00 [141.00, 195.00] | 169.29 [143.50, 200.00] | 169.00 [143.00, 196.00] | N/A | N/A | 165.66 (46.14) | 166.47 (46.47) | -0.02 |
| Missing; n (%) | 58,658 (63.1%) | 13,184 (61.8%) | 92,729 (93.7%) | 25,392 (94.4%) | N/A | N/A | 151,387 (78.9%) | 38,576 (79.9%) | -0.02 |
| | _3,030 (03.170) | ,, (01.0/0) | ,, -5 (55.770) | ,(5 +/0) | | ,. | ,50. (, 5.570) | ,5.0(.5.5/0) | 0.02 |

| Lab result number-Triglyceride level (mg/dl) mean (only | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| =<5000 included) | 34,065 | 8,121 | 6,184 | 1,493 | N/A | N/A | 40,249 | 9,614 | |
| mean (sd) | 181.59 (137.93) | 200.66 (176.08) | 183.77 (164.61) | 203.24 (187.27) | N/A | N/A | 181.92 (142.36) | 201.06 (177.87) | -0.12 |
| median [IQR] | 151.00 [108.00, 214.00] | 161.00 [114.00, 232.00] | 148.00 [103.00, 217.50] | 162.50 [112.00, 237.00] | N/A | N/A | 150.54 (142.36) | 161.23 (177.87) | -0.07 |
| Missing; n (%) | 58,908 (63.4%) | 13,225 (62.0%) | 92,791 (93.8%) | 25,417 (94.5%) | N/A | N/A | 151,699 (79.0%) | 38,642 (80.1%) | -0.03 |
| | 20,222 (22:11-) | | , (, | , (=, | | .,, | | | |
| Lab result number-Hemoglobin mean (only >0 included) | 27,271 | 5,946 | 4,588 | 1,015 | N/A | N/A | 31,859 | 6,961 | |
| mean (sd) | 13.46 (1.61) | 14.01 (1.56) | 12,956.08 (338,258.30) | 2,982.84 (19,853.45) | N/A | N/A | 1877.32 (128356.31) | 446.90 (7579.01) | 0.02 |
| median [IQR] | 13.50 [12.40, 14.60] | 14.05 [12.90, 15.05] | 13.60 [12.50, 14.75] | 14.00 [12.90, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 65,702 (70.7%) | 15,400 (72.1%) | 94,387 (95.4%) | 25,895 (96.2%) | N/A | N/A | 160,089 (83.4%) | 41,295 (85.6%) | -0.06 |
| Lab result number- Serum sodium mean (only > 90 and < | | | | | | | | | |
| 190 included) | 39,270 | 9,104 | 6,401 | 1,563 | N/A | N/A | 45,671 | 10,667 | |
| mean (sd) | 139.43 (2.75) | 139.23 (2.68) | 138.97 (2.59) | 138.92 (2.40) | N/A | N/A | 139.37 (2.73) | 139.18 (2.64) | 0.07 |
| median [IQR] | 139.50 [138.00, 141.00] | 139.00 [138.00, 141.00] | 139.00 [137.00, 141.00] | 139.00 [137.50, 140.25] | N/A | N/A | 139.43 (2.73) | 139.00 (2.64) | 0.16 |
| Missing; n (%) | 53,703 (57.8%) | 12,242 (57.4%) | 92,574 (93.5%) | 25,347 (94.2%) | N/A | N/A | 146,277 (76.2%) | 37,589 (77.9%) | -0.04 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 36,671 | 8,549 | 5,603 | 1,329 | N/A | N/A | 42,274 | 9,878 | |
| mean (sd) | 4.26 (0.31) | 4.30 (0.30) | 4.09 (0.76) | 4.16 (0.66) | N/A | N/A | 4.24 (0.40) | 4.28 (0.37) | -0.10 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 4.20 [4.00, 4.40] | 4.25 [4.00, 4.50] | N/A | N/A | 4.29 (0.40) | 4.29 (0.37) | 0.00 |
| Missing; n (%) | 56,302 (60.6%) | 12,797 (60.0%) | 93,372 (94.3%) | 25,581 (95.1%) | N/A | N/A | 149,674 (78.0%) | 38,378 (79.5%) | -0.04 |
| Lab result number- Glucose (fasting or random) mean | . , , | . , , | . , , | . , , | · | • | . , , | . , , | |
| (only 10-1000 included) | 39,234 | 9,095 | 6,390 | 1,544 | N/A | N/A | 45,624 | 10,639 | |
| mean (sd) | 173.67 (69.39) | 181.41 (70.12) | 179.40 (72.02) | 180.71 (67.24) | N/A | N/A | 174.47 (69.77) | 181.31 (69.71) | -0.10 |
| median [IQR] | 158.00 [126.67, 203.00] | 166.50 [132.00, 216.00] | 162.00 [130.00, 211.50] | 167.00 [133.00, 216.00] | N/A | N/A | 158.56 (69.77) | 166.57 (69.71) | -0.11 |
| Missing; n (%) | 53,739 (57.8%) | 12,251 (57.4%) | 92,585 (93.5%) | 25,366 (94.3%) | N/A | N/A | 146,324 (76.2%) | 37,617 (78.0%) | -0.04 |
| O, (· / | , , | , - ( , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | .,, | • | , | .,. , . , | , | |
| Lab result number-Potassium mean (only 1-7 included) | 40,119 | 9,278 | 6,414 | 1,521 | N/A | N/A | 46,533 | 10,799 | |
| mean (sd) | 4.47 (0.44) | 4.45 (0.41) | 4.33 (0.46) | 4.36 (0.43) | N/A | N/A | 4.45 (0.44) | 4.44 (0.41) | 0.02 |
| median [IQR] | 4.45 [4.20, 4.70] | 4.40 [4.20, 4.70] | 4.30 [4.00, 4.60] | 4.37 [4.10, 4.60] | N/A | N/A | 4.43 (0.44) | 4.40 (0.41) | 0.07 |
| Missing; n (%) | 52,854 (56.8%) | 12,068 (56.5%) | 92,561 (93.5%) | 25,389 (94.3%) | N/A | N/A | 145,415 (75.8%) | 37,457 (77.6%) | -0.04 |
| Comorbidity Scores | . , , | , | | | · | • | | . , , | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.56 (1.72) | 2.09 (1.29) | 1.87 (1.28) | 1.67 (0.99) | 2.72 (1.83) | 2.35 (1.49) | 2.50 (1.70) | 2.06 (1.30) | 0.29 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | , , | 2.00 [1.00, 3.00] | 1.78 (1.70) | 1.68 (1.30) | 0.07 |
| Frailty Score: Qualitative Version 365 days as Categories, | , | | | | | (,) | • ( • ) | | |
| v1 | | | | | | | | | |
| 0; n (%) | 57,374 (61.7%) | 14,082 (66.0%) | 54,311 (54.9%) | 14,474 (53.8%) | 105,245 (40.7%) | 16,251 (46.3%) | 216,930 (48.1%) | 44,807 (53.7%) | -0.11 |
| 1 to 2; n (%) | 26,259 (28.2%) | 5,640 (26.4%) | 34,281 (34.6%) | 10,034 (37.3%) | 92,632 (35.8%) | 12,243 (34.9%) | 153,172 (34.0%) | 27,917 (33.5%) | 0.01 |
| 3 or more; n (%) | 9,340 (10.0%) | 1,624 (7.6%) | 10,383 (10.5%) | 2,402 (8.9%) | 60,917 (23.5%) | 6,621 (18.9%) | 80,640 (17.9%) | 10,647 (12.8%) | 0.14 |
| 5 61 11161-6, 11 (74) | 3,3 10 (20.070) | 1,021(7.0%) | 10,505 (10.5%) | 2,102 (0.5%) | 00,517 (25.570) | 0,021 (10.570) | 00,010 (27.5%) | 10,017 (12.070) | 0.11 |
| Frailty Score: Empirical Version 365 days as Categories, | | | | | | | | | |
| <0.12908; n (%) | 25,893 (27.9%) | 7,492 (35.1%) | 29,844 (30.2%) | 8,892 (33.0%) | 33,014 (12.8%) | 5,571 (15.9%) | 88,751 (19.7%) | 21,955 (26.3%) | -0.16 |
| 0.12908 - 0.1631167; n (%) | 32,822 (35.3%) | 8,051 (37.7%) | 37,569 (38.0%) | 10,669 (39.6%) | 72,707 (28.1%) | 11,082 (31.6%) | 143,098 (31.7%) | 29,802 (35.7%) | -0.08 |
| >= 0.1631167; n (%) | 34,258 (36.8%) | 5,803 (27.2%) | 31,562 (31.9%) | 7,349 (27.3%) | 153,073 (59.1%) | 18,462 (52.6%) | 218,893 (48.6%) | 31,614 (37.9%) | 0.22 |
| Non-Frailty; n (%) | 54,232 (58.3%) | 12,377 (58.0%) | 51,769 (52.3%) | 14,430 (53.6%) | 12,308 (4.8%) | 1,622 (4.6%) | 118,309 (26.2%) | 28,429 (34.1%) | -0.17 |
| ,,(-) | 0 1,202 (001011) | , (==:=:-, | | = 1, 100 (001011) | ,, | _,, (,, | | , (, | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 0.79 (1.40) | 0.64 (1.17) | 0.88 (1.36) | 0.83 (1.20) | 1.54 (1.93) | 1.25 (1.64) | 1.24 (1.72) | 0.96 (1.40) | 0.18 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | | 1.00 [0.00, 2.00] | 0.57 (1.72) | 0.42 (1.40) | 0.10 |
| Frailty Score (mean): Empirical Version 365 days, | (,, | (,, | (,, | (,, | | | () | ···= (=···+) | |
| mean (sd) | 0.16 (0.05) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.04) | 0.19 (0.06) | 0.18 (0.05) | 0.18 (0.05) | 0.16 (0.04) | 0.44 |
| median [IQR] | 0.15 [0.13, 0.18] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.16] | | 0.17 [0.14, 0.20] | 0.16 (0.05) | 0.15 (0.04) | 0.22 |
| Healthcare Utilization | (,, | 0.2. (0.2., 0.2.) | , | 0.2 (0.22, 0.20) | (,, | (,) | () | 0.20 (0.0.) | |
| Any hospitalization; n (%) | 4,363 (4.7%) | 515 (2.4%) | 4,045 (4.1%) | 559 (2.1%) | 17,460 (6.7%) | 1,265 (3.6%) | 25,868 (5.7%) | 2,339 (2.8%) | 0.14 |
| Any hospitalization, it (x) Any hospitalization within prior 30 days; n (%) | 1,461 (1.6%) | 85 (0.4%) | 1,226 (1.2%) | 80 (0.3%) | 5,637 (2.2%) | 209 (0.6%) | 8,324 (1.8%) | 374 (0.4%) | 0.13 |
| Any hospitalization within prior 30 days, it (%) Any hospitalization during prior 31-180 days; n (%) | 3,101 (3.3%) | 434 (2.0%) | 2,913 (2.9%) | 482 (1.8%) | 12,641 (4.9%) | 1,083 (3.1%) | 18,655 (4.1%) | 1,999 (2.4%) | 0.10 |
| Endocrinologist Visit; n (%) | 8,305 (8.9%) | 3,857 (18.1%) | 8,479 (8.6%) | 5,166 (19.2%) | 28,751 (11.1%) | 6,793 (19.3%) | 45,535 (10.1%) | 15,816 (19.0%) | -0.25 |
| Endocrinologist Visit, if (%) Endocrinologist Visit (30 days prior); n (%) | 5,443 (5.9%) | 2,835 (13.3%) | 5,738 (5.8%) | 4,064 (15.1%) | 18,611 (7.2%) | 4,820 (13.7%) | 29,792 (6.6%) | 11,719 (14.1%) | -0.25 |
| Endocrinologist Visit (30 days prior), if (%) Endocrinologist Visit (31 to 180 days prior); n (%) | 5,625 (6.1%) | 2,733 (12.8%) | 5,578 (5.6%) | 3,673 (13.6%) | 20,367 (7.9%) | 5,233 (14.9%) | 31,570 (7.0%) | 11,639 (14.0%) | -0.23 |
| | 77,583 (83.4%) | 2,733 (12.8%)<br>15,326 (71.8%) | 87,485 (88.4%) | 23,433 (87.1%) | 20,367 (7.9%) | 28,985 (82.5%) | 378,183 (83.9%) | 67,744 (81.3%) | 0.07 |
| Internal medicine/family medicine visits; n (%) | , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 13,320 (/1.8%) | 07,403 (00.4%) | 23,433 (07.1%) | 213,113 (02.3%) | 20,303 (02.370) | 310,103 (03.3%) | 07,744 (01.3%) | 0.07 |
| Internal medicine/family medicine visits (30 days prior);<br>n (%) | 59,224 (63.7%) | 11,193 (52.4%) | 66,816 (67.5%) | 17,732 (65.9%) | 155,670 (60.2%) | 21,013 (59.8%) | 281,710 (62.5%) | 49,938 (59.9%) | 0.05 |
| In (%) Internal medicine/family medicine visits (31 to 180 days | 33,224 (03.7%) | 11,133 (32.4%) | 00,010 (07.5%) | 11,132 (03.3%) | 133,070 (00.2%) | 21,013 (33.0%) | 201,/10(02.3%) | 42,230 (23.376) | 0.05 |
| prior); n (%) | 66,924 (72.0%) | 13,192 (61.8%) | 71,698 (72.4%) | 19,673 (73.1%) | 184,082 (71.1%) | 25,511 (72.6%) | 322,704 (71.6%) | 58,376 (70.0%) | 0.04 |
| Cardiologist visit; n (%) | 22,028 (23.7%) | 4,060 (19.0%) | 17,523 (17.7%) | 4,413 (16.4%) | 79,665 (30.8%) | 9,926 (28.3%) | 119,216 (26.4%) | 18,399 (22.1%) | 0.10 |
| Number of Cardiologist visits (30 days prior); n (%) | 7,462 (8.0%) | 1,253 (5.9%) | 5,922 (6.0%) | 1,343 (5.0%) | 27,234 (10.5%) | 3,020 (8.6%) | 40,618 (9.0%) | 5,616 (6.7%) | 0.10 |
| | 7,402 (0.070) | 1,233 (3.376) | 3,322 (0.0%) | 2,343 (3.070) | 2.,234 (10.3/0) | 5,520 (6.670) | .5,010 (5.0%) | 3,010 (0.770) | 0.03 |

| Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) | 18,520 (19.9%)<br>25,313 (27.2%)<br>3,407 (3.7%)<br>0 (0.0%) | 3,452 (16.2%)<br>4,791 (22.4%)<br>762 (3.6%)<br>0 (0.0%) | 14,636 (14.8%)<br>25,662 (25.9%)<br>3,506 (3.5%)<br>0 (0.0%) | 3,739 (13.9%)<br>6,067 (22.5%)<br>1,117 (4.2%)<br>0 (0.0%) | 68,179 (26.3%)<br>80,490 (31.1%)<br>8,264 (3.2%)<br>0 (0.0%) | 8,616 (24.5%)<br>9,794 (27.9%)<br>1,086 (3.1%)<br>0 (0.0%) | 101,335 (22.5%)<br>131,465 (29.2%)<br>15,177 (3.4%)<br>000 (0.0%) | 15,807 (19.0%)<br>20,652 (24.8%)<br>2,965 (3.6%)<br>000 (0.0%) | 0.09<br>0.10<br>-0.01<br>#DIV/0! |
|---|---|---|---|---|---|---|---|---|---|
| Naive new user v8 ; n (%) Nantidiabetic drugs at index date | 13,385 (14.4%) | 1,888 (8.8%) | 14,612 (14.8%) | 1,995 (7.4%) | 32,045 (12.4%) | 1,925 (5.5%) | 60,042 (13.3%) | 5,808 (7.0%) | 0.21 |
| mean (sd) | 2.23 (0.81) | 2.42 (0.92) | 2.23 (0.79) | 2.46 (0.96) | 2.21 (0.81) | 2.47 (0.91) | 2.22 (0.81) | 2.45 (0.93) | -0.26 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | | 2.00 [2.00, 3.00] | 2.00 (0.81) | 2.00 (0.93) | 0.00 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 10.02 (4.35) | 10.15 (4.34) | 9.12 (4.01) | 10.05 (4.19) | 9.97 (4.17) | 10.43 (4.16) | 9.79 (4.17) | 10.24 (4.22) | -0.11 |
| median [IQR] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 8.00 [6.00, 11.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | [0.00 [8.00, 13.00] | 8.78 (4.17) | 9.42 (4.22) | -0.15 |
| Number of Hospitalizations<br>mean (sd) | 0.05 (0.26) | 0.03 (0.17) | 0.04 (0.23) | 0.02 (0.16) | 0.08 (0.33) | 0.04 (0.22) | 0.07 (0.30) | 0.03 (0.19) | 0.16 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.02 (0.16) | , , | 0.00 [0.00, 0.00] | 0.07 (0.30) | 0.03 (0.19) | 0.00 |
| Number of hospital days | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.50) | 0.00 (0.13) | 0.00 |
| mean (sd) | 0.29 (2.21) | 0.12 (0.98) | 0.23 (1.60) | 0.10 (0.85) | 0.49 (2.90) | 0.21 (1.65) | 0.39 (2.53) | 0.15 (1.28) | 0.12 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , , | 0.00 [0.00, 0.00] | 0.00 (2.53) | 0.00 (1.28) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.31 (0.96) | 0.21 (0.75) | 0.09 (0.93) | 0.05 (0.78) | 0.42 (1.19) | 0.29 (1.02) | 0.32 (1.09) | 0.19 (0.88) | 0.13 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.09) | 0.00 (0.88) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 4.32 (3.26) | 4.23 (3.02) | 4.09 (3.12) | 4.26 (3.12) | 4.81 (3.63) | 4.99 (3.51) | 4.55 (3.45) | 4.56 (3.27) | 0.00 |
| median [IQR] | 4.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 6.00] | 4.00 [3.00, 7.00] | 3.78 (3.45) | 3.42 (3.27) | 0.11 |
| Number of Endocrinologist visits | 0.40(2.04) | 0.06 (3.30) | 0.20 (1.00) | 1.02 (2.44) | 0.61 (2.93) | 1 26 (4 60) | 0.52 (2.58) | 1.11 (3.94) | -0.18 |
| mean (sd)<br>median [IQR] | 0.40 (2.04)<br>0.00 [0.00, 0.00] | 0.96 (3.30)<br>0.00 [0.00, 0.00] | 0.38 (1.98)<br>0.00 [0.00, 0.00] | 1.03 (3.44)<br>0.00 [0.00, 0.00] | | 1.26 (4.60)<br>0.00 [0.00, 0.00] | 0.52 (2.58) | 0.00 (3.94) | 0.00 |
| Number of internal medicine/family medicine visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.38) | 0.00 (3.34) | 0.00 |
| mean (sd) | 8.97 (12.35) | 6.96 (10.66) | 6.59 (7.92) | 6.45 (7.85) | 7.38 (9.52) | 7.56 (9.83) | 7.53 (9.86) | 7.05 (9.47) | 0.05 |
| median [IQR] | 5.00 [2.00, 12.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 9.00] | 4.00 [2.00, 9.00] | 4.00 [2.00, 10.00] | | 4.21 (9.86) | 4.42 (9.47) | -0.02 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 1.01 (2.94) | 0.76 (2.48) | 0.70 (2.37) | 0.62 (2.13) | 1.49 (3.91) | 1.33 (3.64) | 1.22 (3.43) | 0.95 (2.94) | 0.08 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (3.43) | 0.00 (2.94) | 0.00 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd) | 0.47 (1.08) | 0.35 (0.85) | 0.42 (0.97) | 0.34 (0.79) | 0.57 (1.17) | 0.48 (1.04) | 0.52 (1.11) | 0.40 (0.92) | 0.12 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.11) | 0.00 (0.92) | 0.00 |
| Number of HbA1c tests ordered | 1.32 (0.89) | 1.37 (0.87) | 1 00 (0 07) | 1 20 (0 97) | 1.43 (0.84) | 1.57 (0.81) | 1.33 (0.86) | 1.43 (0.85) | -0.12 |
| mean (sd)<br>median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.08 (0.87)<br>1.00 [0.00, 2.00] | 1.30 (0.87)<br>1.00 [1.00, 2.00] | | 2.00 [1.00, 2.00] | 1.00 (0.86) | 1.42 (0.85) | -0.12 |
| Number of glucose tests ordered | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 (0.80) | 1.42 (0.83) | -0.49 |
| mean (sd) | 0.55 (3.99) | 0.43 (1.17) | 0.35 (1.05) | 0.42 (1.12) | 0.42 (1.04) | 0.45 (1.08) | 0.43 (2.04) | 0.44 (1.12) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (2.04) | 0.00 (1.12) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 1.03 (0.93) | 1.06 (0.95) | 0.91 (1.21) | 1.08 (1.23) | 1.03 (0.81) | 1.11 (0.82) | 1.00 (0.94) | 1.09 (1.00) | -0.09 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 (0.94) | 1.00 (1.00) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.04 (0.28) | 0.03 (0.22) | 0.04 (0.26) | 0.04 (0.24) | 0.07 (0.32) | 0.07 (0.33) | 0.06 (0.30) | 0.05 (0.28) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.30) | 0.00 (0.28) | 0.00 |
| Number of BUN tests orderedmean (sd) | 0.03 (0.22) | 0.02 (0.17) | 0.03 (0.21) | 0.02 (0.18) | 0.04 (0.26) | 0.04 (0.26) | 0.04 (0.24) | 0.03 (0.22) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , , | 0.00 [0.00, 0.00] | 0.00 (0.24) | 0.00 (0.22) | 0.00 |
| Number of tests for microalbuminuria | (,, | (,, | (,) | (,) | (,, | (,, | ( | 0.00 (0.22) | |
| mean (sd) | 0.85 (1.20) | 0.84 (1.16) | 0.64 (1.04) | 0.76 (1.11) | 0.50 (0.72) | 0.53 (0.72) | 0.60 (0.91) | 0.68 (0.98) | -0.08 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.91) | 0.00 (0.98) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level | | | | | | | | | |
| mean (sd) | 6.16 (6.85) | 5.46 (5.86) | 2.67 (4.07) | 2.01 (3.26) | 5.84 (7.61) | 5.73 (6.80) | 5.21 (6.82) | 4.46 (5.63) | 0.12 |
| median [IQR] | 5.00 [0.00, 9.00] | 5.00 [0.00, 8.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 3.33 (6.82) | 2.96 (5.63) | 0.06 |
| Use of thiazide; n (%) | 13,054 (14.0%) | 2,752 (12.9%) | 12,759 (12.9%) | 3,416 (12.7%) | 39,231 (15.2%) | 5,305 (15.1%) | 65,044 (14.4%) | 11,473 (13.8%) | 0.02 |
| Use of beta blockers; n (%) Use of calcium channel blockers; n (%) | 39,244 (42.2%)<br>32,362 (34.8%) | 7,904 (37.0%)<br>6,181 (29.0%) | 37,716 (38.1%)<br>31,378 (31.7%) | 9,582 (35.6%)<br>7,884 (29.3%) | 131,430 (50.8%)<br>97,784 (37.8%) | 17,160 (48.9%)<br>11,964 (34.1%) | 208,390 (46.2%)<br>161,524 (35.8%) | 34,646 (41.6%)<br>26,029 (31.2%) | 0.09<br>0.10 |
| osc or calcium channel blockers, II (70) | 32,302 (34.0%) | 0,101 (23.0%) | 31,370 (31.7%) | 7,004 (23.3%) | 31,104 (31.6%) | 11,304 (34.1%) | 101,324 (33.0%) | 20,023 (31.270) | 0.10 |

| | | | | PS-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optu | ım | Market | tScan | Medic | :are | | POOLED | |
| Variable | Reference-DPP4i | Exposure-Canagliflozin | Reference- DPP4i | Exposure-Canagliflozin | Reference- DPP4i | Exposure-Canagliflozin | Reference- DPP4i | Exposure- Canagliflozin | St. Diff |
| Number of patients | 19532 | 19532 | 23168 | 23168 | 33401 | 33401 | 76,101 | 76,101 | |
| Age | | | | | | | | | |
| mean (sd) | 62.47 (8.28) | 62.59 (7.93) | 59.39 (7.08) | 59.50 (6.58) | 71.02 (5.32) | 71.06 (5.19) | 65.28 (6.73) | 65.37 (6.41) | -0.01 |
| median [IQR] | 62.00 [55.00, 68.00] | 62.00 [56.00, 68.00] | 58.00 [54.00, 63.00] | 59.00 [55.00, 63.00] | 70.00 [67.00, 74.00] | 70.00 [67.00, 74.00] | 64.29 (6.73) | 64.60 (6.41) | -0.05 |
| Age categories | | a = | A | F = | ¥ ** *** | a | 40.40.41. | 0.000 (10.000 | _ |
| 18 - 54; n (%) | 4,084 (20.9%) | 3,519 (18.0%) | 6,340 (27.4%) | 5,719 (24.7%) | 0 (0.0%) | 0 (0.0%) | 10,424 (13.7%) | 9,238 (12.1%) | 0.05 |
| 55 - 64; n (%)<br>65 - 74; n (%) | 7,394 (37.9%)<br>6,444 (33.0%) | 8,104 (41.5%)<br>6,418 (32.9%) | 12,899 (55.7%)<br>2,941 (12.7%) | 13,461 (58.1%)<br>3,259 (14.1%) | 424 (1.3%)<br>25,613 (76.7%) | 370 (1.1%)<br>25,764 (77.1%) | 20,717 (27.2%)<br>34,998 (46.0%) | 21,935 (28.8%)<br>35,441 (46.6%) | -0.04<br>-0.01 |
| >=75; n (%) | 1,610 (8.2%) | 6,418 (32.9%)<br>1,491 (7.6%) | 2,941 (12.7%)<br>988 (4.3%) | 3,259 (14.1%)<br>729 (3.1%) | 7,364 (22.0%) | 7,267 (21.8%) | 34,998 (46.0%)<br>9,962 (13.1%) | 35,441 (46.6%)<br>9,487 (12.5%) | -0.01 |
| Gender | 1,010 (0.270) | 1,751 (7.070) | JUU (4.370) | , 25 (3.1/0) | .,507 (22.070) | .,20, (21.0/0) | 3,302 (13.1/0) | 5,.07 (12.370) | 0.02 |
| Males; n (%) | 10,959 (56.1%) | 10,973 (56.2%) | 12,925 (55.8%) | 12,966 (56.0%) | 16,977 (50.8%) | 17,007 (50.9%) | 40,861 (53.7%) | 40,946 (53.8%) | 0.00 |
| Females; n (%) | 8,573 (43.9%) | 8,559 (43.8%) | 10,243 (44.2%) | 10,202 (44.0%) | 16,424 (49.2%) | 16,394 (49.1%) | 35,240 (46.3%) | 35,155 (46.2%) | 0.00 |
| Race | , | , | • | , | , | • | , | | |
| White; n (%) | N/A | N/A | N/A | N/A | 27,463 (82.2%) | 27,436 (82.1%) | 27,463 (82.2%) | 27,436 (82.1%) | 0.00 |
| Black; n (%) | N/A | N/A | N/A | N/A | 2,664 (8.0%) | 2,721 (8.1%) | 2,664 (8.0%) | 2,721 (8.1%) | 0.00 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 905 (2.7%) | 893 (2.7%) | 905 (2.7%) | 893 (2.7%) | 0.00 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 970 (2.9%) | 935 (2.8%) | 970 (2.9%) | 935 (2.8%) | 0.01 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 118 (0.4%) | 125 (0.4%) | 118 (0.4%) | 125 (0.4%) | 0.00 |
| Other/Unknown; n (%) Region (lumping missing&other category with West) | N/A | N/A | N/A | N/A | 1,281 (3.8%) | 1,291 (3.9%) | 1,281 (3.8%) | 1,291 (3.9%) | -0.01 |
| Northeast; n (%) | 1,586 (8.1%) | 1,623 (8.3%) | 3,890 (16.8%) | 3,981 (17.2%) | 5,552 (16.6%) | 5,609 (16.8%) | 11,028 (14.5%) | 11,213 (14.7%) | -0.01 |
| South; n (%) | 10,537 (53.9%) | 10,459 (53.5%) | 4,391 (19.0%) | 4,343 (18.7%) | 15,091 (45.2%) | 15,024 (45.0%) | 30,019 (39.4%) | 29,826 (39.2%) | 0.00 |
| Midwest; n (%) | 4,118 (21.1%) | 4,140 (21.2%) | 12,382 (53.4%) | 12,389 (53.5%) | 7,584 (22.7%) | 7,572 (22.7%) | 24,084 (31.6%) | 24,101 (31.7%) | 0.00 |
| West; n (%) | 3,291 (16.8%) | 3,310 (16.9%) | 2,258 (9.7%) | 2,209 (9.5%) | 5,174 (15.5%) | 5,196 (15.6%) | 10,723 (14.1%) | 10,715 (14.1%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | 247 (1.1%) | 246 (1.1%) | N/A | N/A | 247 (1.1%) | 246 (1.1%) | 0.00 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 2,850 (14.6%) | 2,863 (14.7%) | 2,777 (12.0%) | 2,846 (12.3%) | 8,538 (25.6%) | 8,401 (25.2%) | 14,165 (18.6%) | 14,110 (18.5%) | 0.00 |
| Acute MI; n (%) | 49 (0.3%) | 53 (0.3%) | 65 (0.3%) | 60 (0.3%) | 116 (0.3%) | 118 (0.4%) | 230 (0.3%) | 231 (0.3%) | 0.00 |
| ACS/unstable angina; n (%) Old MI; n (%) | 93 (0.5%)<br>334 (1.7%) | 87 (0.4%)<br>331 (1.7%) | 96 (0.4%)<br>194 (0.8%) | 86 (0.4%)<br>182 (0.8%) | 170 (0.5%)<br>855 (2.6%) | 172 (0.5%)<br>839 (2.5%) | 359 (0.5%)<br>1,383 (1.8%) | 345 (0.5%)<br>1,352 (1.8%) | 0.00<br>0.00 |
| Old MI; n (%) Stable angina; n (%) | 334 (1.7%)<br>402 (2.1%) | 331 (1.7%)<br>407 (2.1%) | 194 (0.8%)<br>311 (1.3%) | 182 (0.8%)<br>310 (1.3%) | 855 (2.6%)<br>988 (3.0%) | 839 (2.5%)<br>954 (2.9%) | 1,383 (1.8%)<br>1,701 (2.2%) | 1,352 (1.8%)<br>1,671 (2.2%) | 0.00 |
| Coronary atherosclerosis and other forms of chronic | 402 (2.1%) | 407 (2.170) | 311 (1.370) | 310 (1.370) | 200 (2.0%) | JJ4 (2.370) | 1,/01 (2.270) | 1,0/1 (2.270) | 0.00 |
| ischemic heart disease; n (%) | 2,663 (13.6%) | 2,698 (13.8%) | 2,638 (11.4%) | 2,695 (11.6%) | 8,217 (24.6%) | 8,074 (24.2%) | 13,518 (17.8%) | 13,467 (17.7%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 88 (0.5%) | 85 (0.4%) | 113 (0.5%) | 130 (0.6%) | 339 (1.0%) | 384 (1.1%) | 540 (0.7%) | 599 (0.8%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent); | , 7 | ' | | | / | , | ,, | , | |
| n (%) | 25 (0.1%) | 25 (0.1%) | 37 (0.2%) | 32 (0.1%) | 40 (0.1%) | 67 (0.2%) | 102 (0.1%) | 124 (0.2%) | -0.03 |
| History of CABG or PTCA; n (%) | 596 (3.1%) | 600 (3.1%) | 352 (1.5%) | 340 (1.5%) | 2,019 (6.0%) | 1,992 (6.0%) | 2,967 (3.9%) | 2,932 (3.9%) | 0.00 |
| Any stroke; n (%) | 462 (2.4%) | 489 (2.5%) | 450 (1.9%) | 451 (1.9%) | 1,806 (5.4%) | 1,754 (5.3%) | 2,718 (3.6%) | 2,694 (3.5%) | 0.01 |
| Ischemic stroke (w and w/o mention of cerebral | 400 (0.10) | 407 (2 | **** | **** | 4 700 /5 | 4 740 /5 200 | 3 700 /5 55/ | 2 604 /2 ==0 | <u>.</u> |
| infarction); n (%)<br>Hemorrhagic stroke; n (%) | 460 (2.4%)<br>4 (0.0%) | 487 (2.5%)<br>5 (0.0%) | 448 (1.9%)<br>3 (0.0%) | 448 (1.9%)<br>4 (0.0%) | 1,798 (5.4%) | 1,749 (5.2%) | 2,706 (3.6%) | 2,684 (3.5%) | 0.01 |
| TIA; n (%) | 4 (0.0%)<br>48 (0.2%) | 5 (0.0%)<br>59 (0.3%) | 3 (0.0%)<br>46 (0.2%) | 4 (0.0%)<br>50 (0.2%) | 171 (0.5%) | 170 (0.5%) | 265 (0.3%) | 279 (0.4%) | -0.02 |
| Other cerebrovascular disease; n (%) | 138 (0.7%) | 130 (0.7%) | 46 (0.2%)<br>95 (0.4%) | 90 (0.4%) | 349 (1.0%) | 341 (1.0%) | 582 (0.8%) | 561 (0.7%) | -0.02 |
| Late effects of cerebrovascular disease; n (%) | 100 (0.5%) | 92 (0.5%) | 62 (0.3%) | 61 (0.3%) | 271 (0.8%) | 255 (0.8%) | 433 (0.6%) | 408 (0.5%) | 0.01 |
| Cerebrovascular procedure; n (%) | 3 (0.0%) | 6 (0.0%) | 6 (0.0%) | 3 (0.0%) | 13 (0.0%) | 17 (0.1%) | 022 (0.0%) | 026 (0.0%) | #DIV/0! |
| Heart failure (CHF); n (%) | 756 (3.9%) | 780 (4.0%) | 482 (2.1%) | 496 (2.1%) | 2,270 (6.8%) | 2,224 (6.7%) | 3,508 (4.6%) | 3,500 (4.6%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n | | | | | | | | | |
| (%) | 858 (4.4%) | 863 (4.4%) | 590 (2.5%) | 615 (2.7%) | 2,598 (7.8%) | 2,579 (7.7%) | 4,046 (5.3%) | 4,057 (5.3%) | 0.00 |
| Atrial fibrillation; n (%) | 854 (4.4%) | 843 (4.3%) | 704 (3.0%) | 711 (3.1%) | 2,914 (8.7%) | 2,860 (8.6%) | 4,472 (5.9%) | 4,414 (5.8%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 1,067 (5.5%) | 1,057 (5.4%) | 794 (3.4%) | 788 (3.4%) | 3,293 (9.9%) | 3,214 (9.6%) | 5,154 (6.8%) | 5,059 (6.6%) | 0.01 |
| Cardiac conduction disorders; n (%) | 270 (1.4%) | 270 (1.4%) | 227 (1.0%) | 220 (0.9%) | 864 (2.6%) | 912 (2.7%) | 1,361 (1.8%) | 1,402 (1.8%) | 0.00 |
| Other CVD; n (%) | 1,212 (6.2%) | 1,194 (6.1%) | 1,109 (4.8%) | 1,153 (5.0%) | 3,635 (10.9%) | 3,614 (10.8%) | 5,956 (7.8%) | 5,961 (7.8%) | 0.00 |
| Diabetes-related complications Diabetic retinopathy; n (%) | 1,161 (5.9%) | 1,147 (5.9%) | 909 (3.9%) | 935 (4.0%) | 2,514 (7.5%) | 2,514 (7.5%) | 4,584 (6.0%) | 4,596 (6.0%) | 0.00 |
| Diabetes with other ophthalmic manifestations; n (%) | 120 (0.6%) | 136 (0.7%) | 561 (2.4%) | 567 (2.4%) | 879 (2.6%) | 924 (2.8%) | 1 560 /2 00/3 | 1,627 (2.1%) | -0.01 |
| (%) Retinal detachment, vitreous hemorrhage, | 120 (0.6%) | 130 (U./%) | on1 (2.4%) | 307 (2.4%) | 0/9(2.0%) | 324 (2.8%) | 1,560 (2.0%) | 1,02/(2.1%) | -0.01 |
| vitrectomy; n (%) | 70 (0.4%) | 73 (0.4%) | 82 (0.4%) | 69 (0.3%) | 153 (0.5%) | 140 (0.4%) | 305 (0.4%) | 282 (0.4%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 115 (0.6%) | 103 (0.5%) | 145 (0.6%) | 122 (0.5%) | 222 (0.7%) | 209 (0.6%) | 482 (0.6%) | 434 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy ; n (%) | 3,305 (16.9%) | 3,391 (17.4%) | 2,498 (10.8%) | 2,503 (10.8%) | 6,540 (19.6%) | 6,535 (19.6%) | 12,343 (16.2%) | 12,429 (16.3%) | 0.00 |
| · | | | | | , . , . , . , . , . , | () | | / | |

| Occurrence of diabetic nephropathy with ICD10; n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (%) | 1,981 (10.1%) | 2,014 (10.3%) | 1,299 (5.6%) | 1,282 (5.5%) | 2,783 (8.3%) | 2,769 (8.3%) | 6,063 (8.0%) | 6,065 (8.0%) | 0.00 |
| Hypoglycemia ; n (%) | 403 (2.1%) | 414 (2.1%) | 517 (2.2%) | 518 (2.2%) | 736 (2.2%) | 769 (2.3%) | 1,656 (2.2%) | 1,701 (2.2%) | 0.00 |
| Hyperglycemia; n (%) | 650 (3.3%) | 631 (3.2%) | 659 (2.8%) | 626 (2.7%) | 1,112 (3.3%) | 1,107 (3.3%) | 2,421 (3.2%) | 2,364 (3.1%) | 0.01 |
| Disorders of fluid electrolyte and acid-base balance; n | | | | | | | | | |
| (%) | 653 (3.3%) | 647 (3.3%) | 501 (2.2%) | 511 (2.2%) | 1,420 (4.3%) | 1,381 (4.1%) | 2,574 (3.4%) | 2,539 (3.3%) | 0.01 |
| Diabetic ketoacidosis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome | | | | | | | | | |
| (HONK); n (%) | 86 (0.4%) | 88 (0.5%) | 80 (0.3%) | 81 (0.3%) | 163 (0.5%) | 158 (0.5%) | 329 (0.4%) | 327 (0.4%) | 0.00 |
| Diabetes with peripheral circulatory disorders with | | | | | | | | | |
| ICD-10 ; n (%) | 947 (4.8%) | 954 (4.9%) | 586 (2.5%) | 581 (2.5%) | 1,982 (5.9%) | 1,982 (5.9%) | 3,515 (4.6%) | 3,517 (4.6%) | 0.00 |
| Diabetic Foot; n (%) | 261 (1.3%) | 257 (1.3%) | 275 (1.2%) | 275 (1.2%) | 663 (2.0%) | 679 (2.0%) | 1,199 (1.6%) | 1,211 (1.6%) | 0.00 |
| Gangrene ; n (%) | 19 (0.1%) | 19 (0.1%) | 8 (0.0%) | 9 (0.0%) | 36 (0.1%) | 27 (0.1%) | 063 (0.1%) | 055 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 67 (0.3%) | 58 (0.3%) | 30 (0.1%) | 28 (0.1%) | 100 (0.3%) | 106 (0.3%) | 197 (0.3%) | 192 (0.3%) | 0.00 |
| Osteomyelitis; n (%) | 54 (0.3%) | 49 (0.3%) | 58 (0.3%) | 53 (0.2%) | 109 (0.3%) | 97 (0.3%) | 221 (0.3%) | 199 (0.3%) | 0.00 |
| Skin infections ; n (%) | 890 (4.6%) | 893 (4.6%) | 949 (4.1%) | 989 (4.3%) | 1,854 (5.6%) | 1,877 (5.6%) | 3,693 (4.9%) | 3,759 (4.9%) | 0.00 |
| Erectile dysfunction; n (%) | 689 (3.5%) | 695 (3.6%) | 617 (2.7%) | 635 (2.7%) | 1,022 (3.1%) | 1,015 (3.0%) | 2,328 (3.1%) | 2,345 (3.1%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 1,023 (5.2%) | 990 (5.1%) | 1,050 (4.5%) | 991 (4.3%) | 1,780 (5.3%) | 1,745 (5.2%) | 3,853 (5.1%) | 3,726 (4.9%) | 0.01 |
| Diabetes mellitus without mention of complications; | | | | | | | | | |
| n (%) | 16,531 (84.6%) | 16,497 (84.5%) | 21,189 (91.5%) | 21,263 (91.8%) | 30,549 (91.5%) | 30,535 (91.4%) | 68,269 (89.7%) | 68,295 (89.7%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims | | | | | | | | | |
| within 365 days; n (%) | 17,868 (91.5%) | 17,907 (91.7%) | 20,220 (87.3%) | 20,239 (87.4%) | 31,932 (95.6%) | 31,930 (95.6%) | 70,020 (92.0%) | 70,076 (92.1%) | 0.00 |
| Hyperlipidemia ; n (%) | 14,994 (76.8%) | 15,046 (77.0%) | 17,333 (74.8%) | 17,386 (75.0%) | 27,362 (81.9%) | 27,400 (82.0%) | 59,689 (78.4%) | 59,832 (78.6%) | 0.00 |
| Edema; n (%) | 914 (4.7%) | 894 (4.6%) | 739 (3.2%) | 756 (3.3%) | 2,395 (7.2%) | 2,412 (7.2%) | 4,048 (5.3%) | 4,062 (5.3%) | 0.00 |
| Renal Dysfunction (non-diabetic) ; n (%) | 1,939 (9.9%) | 2,024 (10.4%) | 1,275 (5.5%) | 1,284 (5.5%) | 4,135 (12.4%) | 4,083 (12.2%) | 7,349 (9.7%) | 7,391 (9.7%) | 0.00 |
| Occurrence of acute renal disease ; n (%) | 164 (0.8%) | 169 (0.9%) | 122 (0.5%) | 119 (0.5%) | 366 (1.1%) | 368 (1.1%) | 652 (0.9%) | 656 (0.9%) | 0.00 |
| Occurrence of chronic renal insufficiency; n (%) | 1,542 (7.9%) | 1,672 (8.6%) | 940 (4.1%) | 937 (4.0%) | 3,348 (10.0%) | 3,378 (10.1%) | 5,830 (7.7%) | 5,987 (7.9%) | -0.01 |
| Chronic kidney disease ; n (%) | 1,464 (7.5%) | 1,563 (8.0%) | 838 (3.6%) | 810 (3.5%) | 3,157 (9.5%) | 3,109 (9.3%) | 5,459 (7.2%) | 5,482 (7.2%) | 0.00 |
| CKD Stage 3-4; n (%) | 753 (3.9%) | 822 (4.2%) | 430 (1.9%) | 420 (1.8%) | 1,843 (5.5%) | 1,828 (5.5%) | 3,026 (4.0%) | 3,070 (4.0%) | 0.00 |
| Occurrence of hypertensive nephropathy; n (%) | 655 (3.4%) | 658 (3.4%) | 335 (1.4%) | 334 (1.4%) | 1,133 (3.4%) | 1,149 (3.4%) | 2,123 (2.8%) | 2,141 (2.8%) | 0.00 |
| Occurrence of miscellaneous renal insufficiency ; n | | | | | | | | | |
| (%) | 390 (2.0%) | 404 (2.1%) | 337 (1.5%) | 368 (1.6%) | 1,135 (3.4%) | 1,135 (3.4%) | 1,862 (2.4%) | 1,907 (2.5%) | -0.01 |
| Glaucoma or cataracts ; n (%) | 3,316 (17.0%) | 3,314 (17.0%) | 3,168 (13.7%) | 3,115 (13.4%) | 9,148 (27.4%) | 9,098 (27.2%) | 15,632 (20.5%) | 15,527 (20.4%) | 0.00 |
| Cellulitis or abscess of toe; n (%) | 197 (1.0%) | 179 (0.9%) | 146 (0.6%) | 144 (0.6%) | 346 (1.0%) | 367 (1.1%) | 689 (0.9%) | 690 (0.9%) | 0.00 |
| Foot ulcer; n (%) | 253 (1.3%) | 241 (1.2%) | 271 (1.2%) | 275 (1.2%) | 657 (2.0%) | 672 (2.0%) | 1,181 (1.6%) | 1,188 (1.6%) | 0.00 |
| Bladder stones; n (%) | 15 (0.1%) | 11 (0.1%) | 10 (0.0%) | 10 (0.0%) | 30 (0.1%) | 49 (0.1%) | 055 (0.1%) | 070 (0.1%) | 0.00 |
| Kidney stones; n (%) | 312 (1.6%) | 305 (1.6%) | 406 (1.8%) | 406 (1.8%) | 692 (2.1%) | 721 (2.2%) | 1,410 (1.9%) | 1,432 (1.9%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | 978 (5.0%) | 975 (5.0%) | 961 (4.1%) | 933 (4.0%) | 2,735 (8.2%) | 2,708 (8.1%) | 4,674 (6.1%) | 4,616 (6.1%) | 0.00 |
| Dipstick urinalysis; n (%) | 6,234 (31.9%) | 5,989 (30.7%) | 7,326 (31.6%) | 7,016 (30.3%) | 11,825 (35.4%) | 11,790 (35.3%) | 25,385 (33.4%) | 24,795 (32.6%) | 0.02 |
| Non-dipstick urinalysis; n (%) | 8,743 (44.8%) | 8,830 (45.2%) | 9,618 (41.5%) | 9,590 (41.4%) | 15,296 (45.8%) | 15,274 (45.7%) | 33,657 (44.2%) | 33,694 (44.3%) | 0.00 |
| Urine function test; n (%) | 279 (1.4%) | 256 (1.3%) | 339 (1.5%) | 306 (1.3%) | 1,002 (3.0%) | 850 (2.5%) | 1,620 (2.1%) | 1,412 (1.9%) | 0.01 |
| Cytology; n (%) | 79 (0.4%) | 80 (0.4%) | 129 (0.6%) | 116 (0.5%) | 229 (0.7%) | 206 (0.6%) | 437 (0.6%) | 402 (0.5%) | 0.01 |
| Cystos; n (%) | 127 (0.7%) | 123 (0.6%) | 151 (0.7%) | 164 (0.7%) | 356 (1.1%) | 317 (0.9%) | 634 (0.8%) | 604 (0.8%) | 0.00 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 1,991 (10.2%) | 2,018 (10.3%) | 1,579 (6.8%) | 1,656 (7.1%) | 5,413 (16.2%) | 5,337 (16.0%) | 8,983 (11.8%) | 9,011 (11.8%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | |
| pain; n (%) | 5,293 (27.1%) | 5,257 (26.9%) | 5,487 (23.7%) | 5,503 (23.8%) | 11,402 (34.1%) | 11,358 (34.0%) | 22,182 (29.1%) | 22,118 (29.1%) | 0.00 |
| Dorsopathies; n (%) | 3,513 (18.0%) | 3,473 (17.8%) | 3,457 (14.9%) | 3,478 (15.0%) | 7,367 (22.1%) | 7,314 (21.9%) | 14,337 (18.8%) | 14,265 (18.7%) | 0.00 |
| Fractures; n (%) | 313 (1.6%) | 304 (1.6%) | 351 (1.5%) | 323 (1.4%) | 758 (2.3%) | 740 (2.2%) | 1,422 (1.9%) | 1,367 (1.8%) | 0.01 |
| Falls; n (%) | 325 (1.7%) | 329 (1.7%) | 125 (0.5%) | 121 (0.5%) | 729 (2.2%) | 691 (2.1%) | 1,179 (1.5%) | 1,141 (1.5%) | 0.00 |
| Osteoporosis; n (%) | 484 (2.5%) | 496 (2.5%) | 262 (1.1%) | 266 (1.1%) | 1,735 (5.2%) | 1,739 (5.2%) | 2,481 (3.3%) | 2,501 (3.3%) | 0.00 |
| Hyperthyroidism; n (%) | 132 (0.7%) | 102 (0.5%) | 131 (0.6%) | 90 (0.4%) | 270 (0.8%) | 238 (0.7%) | 533 (0.7%) | 430 (0.6%) | 0.01 |
| Hypothyroidism ; n (%) | 2,755 (14.1%) | 2,732 (14.0%) | 2,713 (11.7%) | 2,686 (11.6%) | 4,012 (12.0%) | 3,970 (11.9%) | 9,480 (12.5%) | 9,388 (12.3%) | 0.01 |
| Other disorders of thyroid gland; n (%) | 735 (3.8%) | 666 (3.4%) | 780 (3.4%) | 775 (3.3%) | 1,483 (4.4%) | 1,324 (4.0%) | 2,998 (3.9%) | 2,765 (3.6%) | 0.02 |
| Depression; n (%) | 1,318 (6.7%) | 1,347 (6.9%) | 1,367 (5.9%) | 1,317 (5.7%) | 2,756 (8.3%) | 2,733 (8.2%) | 5,441 (7.1%) | 5,397 (7.1%) | 0.00 |
| Anxiety; n (%) | 1,279 (6.5%) | 1,247 (6.4%) | 1,075 (4.6%) | 1,056 (4.6%) | 2,282 (6.8%) | 2,256 (6.8%) | 4,636 (6.1%) | 4,559 (6.0%) | 0.00 |
| Sleep_Disorder; n (%) | 1,356 (6.9%) | 1,364 (7.0%) | 2,268 (9.8%) | 2,344 (10.1%) | 2,703 (8.1%) | 2,706 (8.1%) | 6,327 (8.3%) | 6,414 (8.4%) | 0.00 |
| Dementia; n (%) | 200 (1.0%) | 195 (1.0%) | 110 (0.5%) | 109 (0.5%) | 913 (2.7%) | 893 (2.7%) | 1,223 (1.6%) | 1,197 (1.6%) | 0.00 |
| Delirium; n (%) | 45 (0.2%) | 55 (0.3%) | 28 (0.1%) | 29 (0.1%) | 195 (0.6%) | 179 (0.5%) | 268 (0.4%) | 263 (0.3%) | 0.02 |
| Psychosis; n (%) | 89 (0.5%) | 87 (0.4%) | 44 (0.2%) | 47 (0.2%) | 255 (0.8%) | 255 (0.8%) | 388 (0.5%) | 389 (0.5%) | 0.00 |
| Obesity; n (%) | 5,168 (26.5%) | 5,115 (26.2%) | 4,206 (18.2%) | 4,246 (18.3%) | 6,410 (19.2%) | 6,322 (18.9%) | 15,784 (20.7%) | 15,683 (20.6%) | 0.00 |
| Overweight; n (%) | 1,026 (5.3%) | 1,024 (5.2%) | 576 (2.5%) | 522 (2.3%) | 1,239 (3.7%) | 1,189 (3.6%) | 2,841 (3.7%) | 2,735 (3.6%) | 0.01 |
| Smoking; n (%) | 1,624 (8.3%) | 1,622 (8.3%) | 1,219 (5.3%) | 1,174 (5.1%) | 3,528 (10.6%) | 3,585 (10.7%) | 6,371 (8.4%) | 6,381 (8.4%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 3 (0.0%) | 2 (0.0%) | 6 (0.0%) | 5 (0.0%) | ** | ** | ** | ** | ** |
| Drug abuse or dependence; n (%) | 6 (0.0%) | 7 (0.0%) | 2 (0.0%) | 2 (0.0%) | ** | ** | ** | ** | ** |
| COPD; n (%) | 983 (5.0%) | 998 (5.1%) | 693 (3.0%) | 666 (2.9%) | 2,671 (8.0%) | 2,602 (7.8%) | 4,347 (5.7%) | 4,266 (5.6%) | 0.00 |

| Asthma; n (%) | 870 (4.5%) | 847 (4.3%) | 804 (3.5%) | 802 (3.5%) | 1,756 (5.3%) | 1,728 (5.2%) | 3,430 (4.5%) | 3,377 (4.4%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 2,176 (11.1%) | 2,157 (11.0%) | 2,591 (11.2%) | 2,584 (11.2%) | 3,034 (9.1%) | 3,034 (9.1%) | 7,801 (10.3%) | 7,775 (10.2%) | 0.00 |
| Pneumonia; n (%) | 208 (1.1%) | 221 (1.1%) | 205 (0.9%) | 210 (0.9%) | 511 (1.5%) | 520 (1.6%) | 924 (1.2%) | 951 (1.2%) | 0.00 |
| Imaging; n (%) | 2 (0.0%) | 6 (0.0%) | 1 (0.0%) | 2 (0.0%) | ** | ** | ** | ** | ** |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 112 (0.6%) | 103 (0.5%) | 91 (0.4%) | 77 (0.3%) | 231 (0.7%) | 261 (0.8%) | 434 (0.6%) | 441 (0.6%) | 0.00 |
| DM Medications - Glitazones; n (%) | 1,856 (9.5%) | 1,876 (9.6%) | 2,142 (9.2%) | 2,148 (9.3%) | 3,295 (9.9%) | 3,279 (9.8%) | 7,293 (9.6%) | 7,303 (9.6%) | 0.00 |
| DM Medications - Insulin; n (%) | 4,810 (24.6%) | 4,865 (24.9%) | 5,930 (25.6%) | 5,958 (25.7%) | 10,126 (30.3%) | 10,087 (30.2%) | 20,866 (27.4%) | 20,910 (27.5%) | 0.00 |
| DM Medications - Meglitinides; n (%) | 203 (1.0%) | 194 (1.0%) | 294 (1.3%) | 272 (1.2%) | 583 (1.7%) | 542 (1.6%) | 1,080 (1.4%) | 1,008 (1.3%) | 0.01 |
| DM Medications - Metformin; n (%) | 15,366 (78.7%) | 15,269 (78.2%) | 18,243 (78.7%) | 18,260 (78.8%) | 24,894 (74.5%) | 24,848 (74.4%) | 58,503 (76.9%) | 58,377 (76.7%) | 0.00 |
| Concomitant initiation or current use of 2nd | | | | | | | | | |
| Generation SUs; n (%) | 6,481 (33.2%) | 6,440 (33.0%) | 7,299 (31.5%) | 7,328 (31.6%) | 12,787 (38.3%) | 12,548 (37.6%) | 26,567 (34.9%) | 26,316 (34.6%) | 0.01 |
| Concomitant initiation or current use of AGIs; n (%) | 50 (0.3%) | 77 (0.4%) | 33 (0.1%) | 50 (0.2%) | 154 (0.5%) | 175 (0.5%) | 237 (0.3%) | 302 (0.4%) | -0.02 |
| Concomitant initiation or current use of Glitazones; | | | | | | | | | |
| n (%) | 1,422 (7.3%) | 1,425 (7.3%) | 1,643 (7.1%) | 1,624 (7.0%) | 2,474 (7.4%) | 2,510 (7.5%) | 5,539 (7.3%) | 5,559 (7.3%) | 0.00 |
| Concomitant initiation or current use of GLP-1 RA; n | | | | | | | | | |
| (%) | 1,432 (7.3%) | 1,544 (7.9%) | 1,891 (8.2%) | 1,968 (8.5%) | 2,410 (7.2%) | 2,543 (7.6%) | 5,733 (7.5%) | 6,055 (8.0%) | -0.02 |
| Concomitant initiation or current use of Insulin; n | | | | | | | | | |
| (%) | 3,600 (18.4%) | 3,644 (18.7%) | 4,552 (19.6%) | 4,589 (19.8%) | 7,923 (23.7%) | 7,913 (23.7%) | 16,075 (21.1%) | 16,146 (21.2%) | 0.00 |
| Concomitant initiation or current use of | | | | | | | | | |
| Meglitinides; n (%) | 110 (0.6%) | 131 (0.7%) | 108 (0.5%) | 199 (0.9%) | 404 (1.2%) | 381 (1.1%) | 622 (0.8%) | 711 (0.9%) | -0.01 |
| Concomitant initiation or current use of Metformin; | | | | | | | | | |
| n (%) | 13,063 (66.9%) | 12,913 (66.1%) | 15,539 (67.1%) | 15,521 (67.0%) | 21,246 (63.6%) | 21,219 (63.5%) | 49,848 (65.5%) | 49,653 (65.2%) | 0.01 |
| Past use of 2nd Generation SUs; n (%) | 1,625 (8.3%) | 1,648 (8.4%) | 1,695 (7.3%) | 1,732 (7.5%) | 2,612 (7.8%) | 2,636 (7.9%) | 5,932 (7.8%) | 6,016 (7.9%) | 0.00 |
| Past use of AGIs; n (%) | 62 (0.3%) | 26 (0.1%) | 58 (0.3%) | 27 (0.1%) | 77 (0.2%) | 86 (0.3%) | 197 (0.3%) | 139 (0.2%) | 0.02 |
| Past use of Glitazones ; n (%) | 434 (2.2%) | 451 (2.3%) | 499 (2.2%) | 524 (2.3%) | 821 (2.5%) | 769 (2.3%) | 1,754 (2.3%) | 1,744 (2.3%) | 0.00 |
| Past use of GLP-1 RA; n (%) | 926 (4.7%) | 958 (4.9%) | 1,232 (5.3%) | 1,223 (5.3%) | 1,589 (4.8%) | 1,615 (4.8%) | 3,747 (4.9%) | 3,796 (5.0%) | 0.00 |
| Past use of Insulin ; n (%) | 1,210 (6.2%) | 1,221 (6.3%) | 1,379 (6.0%) | 1,369 (5.9%) | 2,204 (6.6%) | 2,175 (6.5%) | 4,793 (6.3%) | 4,765 (6.3%) | 0.00 |
| Past use of Meglitinides ; n (%) | 93 (0.5%) | 63 (0.3%) | 186 (0.8%) | 73 (0.3%) | 179 (0.5%) | 161 (0.5%) | 458 (0.6%) | 297 (0.4%) | 0.03 |
| Past use of metformin (final); n (%) | 2,303 (11.8%) | 2,356 (12.1%) | 2,705 (11.7%) | 2,739 (11.8%) | 3,648 (10.9%) | 3,629 (10.9%) | 8,656 (11.4%) | 8,724 (11.5%) | 0.00 |
| Other Medications | | . , , | | | , | , | | , | |
| Use of ACE inhibitors; n (%) | 10,585 (54.2%) | 10,617 (54.4%) | 12,359 (53.3%) | 12,301 (53.1%) | 16,705 (50.0%) | 16,765 (50.2%) | 39,649 (52.1%) | 39,683 (52.1%) | 0.00 |
| Use of ARBs; n (%) | 7,026 (36.0%) | 7,007 (35.9%) | 8,593 (37.1%) | 8,662 (37.4%) | 12,369 (37.0%) | 12,384 (37.1%) | 27,988 (36.8%) | 28,053 (36.9%) | 0.00 |
| Use of Loop Diuretics ; n (%) | 1,811 (9.3%) | 1,788 (9.2%) | 1,879 (8.1%) | 1,836 (7.9%) | 5,110 (15.3%) | 5,163 (15.5%) | 8,800 (11.6%) | 8,787 (11.5%) | 0.00 |
| Use of other diuretics; n (%) | 505 (2.6%) | 487 (2.5%) | 581 (2.5%) | 573 (2.5%) | 1,151 (3.4%) | 1,124 (3.4%) | 2,237 (2.9%) | 2,184 (2.9%) | 0.00 |
| Use of nitrates-United; n (%) | 696 (3.6%) | 705 (3.6%) | 742 (3.2%) | 742 (3.2%) | 2,191 (6.6%) | 2,134 (6.4%) | 3,629 (4.8%) | 3,581 (4.7%) | 0.00 |
| Use of other hypertension drugs; n (%) | 1,040 (5.3%) | 1,072 (5.5%) | 1,133 (4.9%) | 1,140 (4.9%) | 2,470 (7.4%) | 2,473 (7.4%) | 4,643 (6.1%) | 4,685 (6.2%) | 0.00 |
| Use of digoxin; n (%) | 234 (1.2%) | 218 (1.1%) | 189 (0.8%) | 217 (0.9%) | 754 (2.3%) | 737 (2.2%) | 1,177 (1.5%) | 1,172 (1.5%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 153 (0.8%) | 160 (0.8%) | 165 (0.7%) | 169 (0.7%) | 504 (1.5%) | 478 (1.4%) | 822 (1.1%) | 807 (1.1%) | 0.00 |
| Use of COPD/asthma meds; n (%) | 2,610 (13.4%) | 2,552 (13.1%) | 3,182 (13.7%) | 3,201 (13.8%) | 5,500 (16.5%) | 5,455 (16.3%) | 11,292 (14.8%) | 11,208 (14.7%) | 0.00 |
| Use of statins; n (%) | 14,115 (72.3%) | 14,168 (72.5%) | 15,879 (68.5%) | 16,013 (69.1%) | 25,077 (75.1%) | 25,241 (75.6%) | 55,071 (72.4%) | 55,422 (72.8%) | -0.01 |
| Use of other lipid-lowering drugs; n (%) | 2,443 (12.5%) | 2,510 (12.9%) | 3,546 (15.3%) | 3,536 (15.3%) | 5,010 (15.0%) | 4,896 (14.7%) | 10,999 (14.5%) | 10,942 (14.4%) | 0.00 |
| Use of antiplatelet agents; n (%) | 1,985 (10.2%) | 1,937 (9.9%) | 2,289 (9.9%) | 2,327 (10.0%) | 4,642 (13.9%) | 4,642 (13.9%) | 8,916 (11.7%) | 8,906 (11.7%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | 1,363 (10.276) | 1,537 (5.570) | 2,209 (9.970) | 2,327 (10.070) | 4,042 (13.576) | 4,042 (13.570) | 8,510 (11.776) | 8,500 (11.776) | 0.00 |
| Apixaban, Warfarin); n (%) | 833 (4.3%) | 855 (4.4%) | 799 (3.4%) | 791 (3.4%) | 2,604 (7.8%) | 2,590 (7.8%) | 4,236 (5.6%) | 4,236 (5.6%) | 0.00 |
| Use of heparin and other low-molecular weight | 033 (4.370) | 055 (4.470) | 755 (5.470) | 751 (5.470) | 2,004 (7.070) | 2,550 (7.670) | 4,230 (3.070) | 4,230 (3.070) | 0.00 |
| heparins; n (%) | 18 (0.1%) | 19 (0.1%) | 0 (0.0%) | 0 (0.0%) | 61 (0.2%) | 62 (0.2%) | 079 (0.1%) | 081 (0.1%) | 0.00 |
| Use of NSAIDs; n (%) | 3,256 (16.7%) | 3,211 (16.4%) | 3,774 (16.3%) | 3,788 (16.4%) | 5,117 (15.3%) | 5,126 (15.3%) | 12,147 (16.0%) | 12,125 (15.9%) | 0.00 |
| Use of oral corticosteroids; n (%) | 2,279 (11.7%) | 2,243 (11.5%) | 2,550 (11.0%) | 2,583 (11.1%) | 4,680 (14.0%) | 4,595 (13.8%) | 9,509 (12.5%) | 9,421 (12.4%) | 0.00 |
| Use of bisphosphonate (United); n (%) | 232 (1.2%) | 237 (1.2%) | 149 (0.6%) | 145 (0.6%) | 715 (2.1%) | 761 (2.3%) | 1,096 (1.4%) | 1,143 (1.5%) | -0.01 |
| Use of opioids; n (%) | 3,797 (19.4%) | 3,784 (19.4%) | 4,612 (19.9%) | 4,603 (19.9%) | 6,800 (20.4%) | 6,685 (20.0%) | 15,209 (20.0%) | 15,072 (19.8%) | 0.01 |
| Use of antidepressants; n (%) | 4,446 (22.8%) | 4,408 (22.6%) | 5,009 (21.6%) | 4,990 (21.5%) | 8,171 (24.5%) | 8,112 (24.3%) | 17,626 (23.2%) | 17,510 (23.0%) | 0.00 |
| Use of antipsychotics; n (%) | 347 (1.8%) | 337 (1.7%) | 272 (1.2%) | 250 (1.1%) | 668 (2.0%) | 682 (2.0%) | 1,287 (1.7%) | 1,269 (1.7%) | 0.00 |
| Use of anticonvulsants; n (%) | 2,716 (13.9%) | 2,697 (13.8%) | 2,509 (10.8%) | 2,513 (10.8%) | 5,149 (15.4%) | 5,060 (15.1%) | 10,374 (13.6%) | 10,270 (13.5%) | 0.00 |
| Use of lithium; n (%) | 29 (0.1%) | 18 (0.1%) | 27 (0.1%) | 14 (0.1%) | 48 (0.1%) | 29 (0.1%) | 104 (0.1%) | 061 (0.1%) | 0.00 |
| Use of Benzos; n (%) | 1,741 (8.9%) | 1,703 (8.7%) | 1,946 (8.4%) | 1,965 (8.5%) | 3,284 (9.8%) | 3,237 (9.7%) | 6,971 (9.2%) | 6,905 (9.1%) | 0.00 |
| Use of anxiolytics/hypnotics; n (%) | 1,016 (5.2%) | 1,001 (5.1%) | 1,247 (5.4%) | 1,234 (5.3%) | 1,747 (5.2%) | 1,718 (5.1%) | 4,010 (5.3%) | 3,953 (5.2%) | 0.00 |
| Use of dementia meds; n (%) | 126 (0.6%) | 129 (0.7%) | 79 (0.3%) | 80 (0.3%) | 747 (2.2%) | 705 (2.1%) | 952 (1.3%) | 914 (1.2%) | 0.01 |
| Use of antiparkinsonian meds; n (%) | 356 (1.8%) | 357 (1.8%) | 392 (1.7%) | 365 (1.6%) | 926 (2.8%) | 944 (2.8%) | 1,674 (2.2%) | 1,666 (2.2%) | 0.00 |
| Any use of pramlintide; n (%) | 3 (0.0%) | 24 (0.1%) | 6 (0.0%) | 43 (0.2%) | ** | ** | ** | ** | ** |
| Any use of 1st generation sulfonylureas; n (%) | 0 (0.0%) | 0 (0.0%) | 1 (0.0%) | 0 (0.0%) | ** | ** | ** | ** | ** |
| Entresto (sacubitril/valsartan); n (%) | 24 (0.1%) | 14 (0.1%) | 3 (0.0%) | 4 (0.0%) | 14 (0.0%) | 13 (0.0%) | 041 (0.1%) | 031 (0.0%) | 0.00 |
| Initiation as monotherapy ; n (%) | 1,207 (6.2%) | 1,196 (6.1%) | 1,314 (5.7%) | 1,306 (5.6%) | 1,176 (3.5%) | 1,217 (3.6%) | 3,697 (4.9%) | 3,719 (4.9%) | 0.00 |
| Labs | 1,207 (0.270) | 1,130 (0.176) | 1,314 (3.770) | 1,300 (3.0%) | 1,1/0 (3.3%) | 1,41/ (3.0%) | 3,697 (4.9%)<br>42,700 | 3,719 (4.9%) | 0.00 |
| Lab values- HbA1c (%) ; n (%) | 8,392 (43.0%) | 8,484 (43.4%) | 1,674 (7.2%) | 1,435 (6.2%) | N/A | N/A | 10,066 (23.6%) | 9,919 (23.2%) | 0.01 |
| Lab values- HbA1c (%) ; n (%)<br>Lab values- HbA1c (%) (within 3 months) ; n (%) | 6,836 (35.0%) | 6,971 (35.7%) | 1,874 (7.2%) | 1,435 (6.2%) | N/A<br>N/A | N/A<br>N/A | 8,206 (19.2%) | 8,195 (19.2%) | 0.00 |
| Lab values- HbA1c (%) (within 3 months); n (%) Lab values- HbA1c (%) (within 6 months); n (%) | 8,392 (43.0%) | 8,484 (43.4%) | 1,674 (7.2%) | 1,435 (6.2%) | N/A<br>N/A | N/A<br>N/A | 10,066 (23.6%) | 9,919 (23.2%) | 0.00 |
| Lab variacs TIDATE (/0) (WILLIIII O IIIOTILIIS), II (/0) | 0,332 (43.070) | 0,404 (43.470) | 1,074 (7.270) | 1,433 (0.270) | N/A | IN/A | 10,000 (23.076) | 3,313 (23.270) | 0.01 |

| Lab values- BNP; n (%) | 102 (0.5%) | 120 (0.6%) | 23 (0.1%) | 4 (0.0%) | N/A | N/A | 125 (0.3%) | 124 (0.3%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP (within 3 months); n (%) | 62 (0.3%) | 76 (0.4%) | 18 (0.1%) | 3 (0.0%) | N/A | N/A | 080 (0.2%) | 079 (0.2%) | 0.00 |
| Lab values- BNP (within 6 months); n (%) | 102 (0.5%) | 120 (0.6%) | 23 (0.1%) | 4 (0.0%) | N/A | N/A | 125 (0.3%) | 124 (0.3%) | 0.00 |
| Lab values- BUN (mg/dl); n (%) | 8,334 (42.7%) | 8,259 (42.3%) | 1,582 (6.8%) | 1,359 (5.9%) | N/A | N/A | 9,916 (23.2%) | 9,618 (22.5%) | 0.02 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 6,579 (33.7%) | 6,626 (33.9%) | 1,244 (5.4%) | 1,116 (4.8%) | N/A | N/A | 7,823 (18.3%) | 7,742 (18.1%) | 0.01 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 8,334 (42.7%) | 8,259 (42.3%) | 1,582 (6.8%) | 1,359 (5.9%) | N/A | N/A | 9,916 (23.2%) | 9,618 (22.5%) | 0.02 |
| Lab values- Creatinine (mg/dl); n (%) | 8,573 (43.9%) | 8,526 (43.7%) | 1,691 (7.3%) | 1,486 (6.4%) | N/A | N/A | 10,264 (24.0%) | 10,012 (23.4%) | 0.01 |
| Lab values- Creatinine (mg/dl) (within 3 months); n | 8,373 (43.5%) | 8,320 (43.7%) | 1,091 (7.3%) | 1,480 (0.4%) | N/A | 11// | 10,204 (24.070) | 10,012 (23.476) | 0.01 |
| | 6 700 (24 70) | 6 025 (25 00) | 4 227 (5 00/) | 4 222 (5 20() | 21/2 | 21/2 | 0.447 (40.00() | 0.007 (40.00() | 0.00 |
| (%) | 6,780 (34.7%) | 6,835 (35.0%) | 1,337 (5.8%) | 1,232 (5.3%) | N/A | N/A | 8,117 (19.0%) | 8,067 (18.9%) | 0.00 |
| Lab values- Creatinine (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 8,573 (43.9%) | 8,526 (43.7%) | 1,691 (7.3%) | 1,486 (6.4%) | N/A | N/A | 10,264 (24.0%) | 10,012 (23.4%) | 0.01 |
| Lab values- HDL level (mg/dl); n (%) | 7,438 (38.1%) | 7,329 (37.5%) | 1,535 (6.6%) | 1,315 (5.7%) | N/A | N/A | 8,973 (21.0%) | 8,644 (20.2%) | 0.02 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 5,579 (28.6%) | 5,616 (28.8%) | 1,181 (5.1%) | 1,045 (4.5%) | N/A | N/A | 6,760 (15.8%) | 6,661 (15.6%) | 0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 7,438 (38.1%) | 7,329 (37.5%) | 1,535 (6.6%) | 1,315 (5.7%) | N/A | N/A | 8,973 (21.0%) | 8,644 (20.2%) | 0.02 |
| Lab values- LDL level (mg/dl); n (%) | 7,633 (39.1%) | 7,557 (38.7%) | 1,599 (6.9%) | 1,341 (5.8%) | N/A | N/A | 9,232 (21.6%) | 8,898 (20.8%) | 0.02 |
| 3, 7, 7, 7, | ,, | , ( , | ,, | ,- ( , | • | • | -, - , - , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| Lab values-LDL level (mg/dl) (within 3 months); n (%) | 5,723 (29.3%) | 5,809 (29.7%) | 1,227 (5.3%) | 1,068 (4.6%) | N/A | N/A | 6,950 (16.3%) | 6,877 (16.1%) | 0.01 |
| zas values zsztievei (ing/ai/ (intiinis inontiis/) ii (/o/ | 3,723 (23.370) | 3,003 (23.770) | 1,227 (3.370) | 1,000 (1.0%) | , | .,,,, | 0,550 (10.570) | 0,077 (10.170) | 0.01 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 7,633 (39.1%) | 7,557 (38.7%) | 1,599 (6.9%) | 1,341 (5.8%) | N/A | N/A | 9,232 (21.6%) | 8,898 (20.8%) | 0.02 |
| | | | | | • | • | | | 0.02 |
| Lab values- NT-proBNP; n (%) | 14 (0.1%) | 12 (0.1%) | 3 (0.0%) | 0 (0.0%) | N/A | N/A | 17 (0.0%) | 0 (0.0%) | |
| Lab values- NT-proBNP (within 3 months); n (%) | 9 (0.0%) | 7 (0.0%) | 3 (0.0%) | 0 (0.0%) | N/A | N/A | 12 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 14 (0.1%) | 12 (0.1%) | 3 (0.0%) | 0 (0.0%) | N/A | N/A | 17 (0.0%) | 12 (0.0%) | - |
| Lab values-Total cholesterol (mg/dl); n (%) | 7,546 (38.6%) | 7,484 (38.3%) | 1,541 (6.7%) | 1,326 (5.7%) | N/A | N/A | 9,087 (21.3%) | 8,810 (20.6%) | 0.02 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 5,669 (29.0%) | 5,759 (29.5%) | 1,188 (5.1%) | 1,059 (4.6%) | N/A | N/A | 6,857 (16.1%) | 6,818 (16.0%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 7,546 (38.6%) | 7,484 (38.3%) | 1,541 (6.7%) | 1,326 (5.7%) | N/A | N/A | 9,087 (21.3%) | 8,810 (20.6%) | 0.02 |
| Lab values-Triglyceride level (mg/dl); n (%) | 7,490 (38.3%) | 7,438 (38.1%) | 1,519 (6.6%) | 1,304 (5.6%) | N/A | N/A | 9,009 (21.1%) | 8,742 (20.5%) | 0.01 |
| Lab values- Triglyceride level (mg/dl) (within 3 | ,,,,,,, | .,(, | _, | _,, | .,, | | -, (, | -,- := (, | |
| months); n (%) | 5,623 (28.8%) | 5,720 (29.3%) | 1,169 (5.0%) | 1,046 (4.5%) | N/A | N/A | 6,792 (15.9%) | 6,766 (15.8%) | 0.00 |
| | 3,023 (28.8%) | 3,720 (29.3%) | 1,169 (5.0%) | 1,046 (4.5%) | N/A | IN/A | 0,792 (13.9%) | 0,700 (13.6%) | 0.00 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 7,490 (38.3%) | 7,438 (38.1%) | 1,519 (6.6%) | 1,304 (5.6%) | N/A | N/A | 9,009 (21.1%) | 8,742 (20.5%) | 0.01 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 8,349 | 8,430 | 1,628 | 1,384 | N/A | N/A | 9,977 | 9,814 | |
| mean (sd) | 8.53 (1.83) | 8.61 (1.75) | 8.63 (1.88) | 8.63 (1.72) | N/A | N/A | 8.55 (1.84) | 8.61 (1.75) | -0.03 |
| median [IQR] | 8.10 [7.30, 9.45] | 8.30 [7.40, 9.60] | 8.20 [7.30, 9.50] | 8.30 [7.40, 9.59] | N/A | N/A | 8.12 (1.84) | 8.30 (1.75) | -0.10 |
| Missing; n (%) | 11,183 (57.3%) | 11,102 (56.8%) | 21,540 (93.0%) | 21,784 (94.0%) | N/A | N/A | 32,723 (76.6%) | 32,886 (77.0%) | -0.01 |
| Lab result number- BNP mean | 102 | 120 | 23 | 4 | N/A | N/A | 125 | 124 | |
| mean (sd) | 119.72 (204.33) | 95.52 (162.94) | 239.13 (519.14) | 335.38 (447.47) | N/A | N/A | 141.69 (288.38) | 103.26 (176.28) | 0.16 |
| median [IQR] | 48.55 [20.27, 141.98] | 44.35 [21.32, 88.78] | 49.00 [20.00, 214.00] | 192.50 [4.25, 809.38] | N/A | N/A | #VALUE! | 49.13 (176.28) | #VALUE! |
| | | | | | • | • | | | |
| Missing; n (%) | 19,430 (99.5%) | 19,412 (99.4%) | 23,145 (99.9%) | 23,164 (100.0%) | N/A | N/A | 42,575 (99.7%) | 42,576 (99.7%) | 0.00 |
| Lab result number- BUN (mg/dl) mean | 8,334 | 8,259 | 1,582 | 1,359 | N/A | N/A | 9,916 | 9,618 | |
| mean (sd) | 17.03 (6.43) | | 629.58 (9,120.88) | 3,069.88 (21,521.68) | N/A | N/A | 114.76 (3642.51) | 448.30 (8088.19) | -0.05 |
| median [IQR] | 16.00 [13.00, 20.00] | 16.00 [13.00, 19.50] | 15.50 [12.50, 19.00] | 16.00 [13.00, 20.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 11,198 (57.3%) | 11,273 (57.7%) | 21,586 (93.2%) | 21,809 (94.1%) | N/A | N/A | 32,784 (76.8%) | 33,082 (77.5%) | -0.02 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | |
| to 15 included) | 8,519 | 8,459 | 1,536 | 1,339 | N/A | N/A | 10,055 | 9,798 | |
| mean (sd) | 0.96 (0.31) | 0.92 (0.24) | 0.96 (0.30) | 0.93 (0.23) | N/A | N/A | 0.96 (0.31) | 0.92 (0.24) | 0.14 |
| median [IQR] | 0.90 [0.77, 1.09] | 0.89 [0.75, 1.04] | 0.92 [0.77, 1.07] | 0.90 [0.77, 1.06] | N/A | N/A | 0.90 (0.31) | 0.89 (0.24) | 0.04 |
| Missing; n (%) | 11,013 (56.4%) | 11,073 (56.7%) | 21,632 (93.4%) | 21,829 (94.2%) | N/A | N/A | 32,645 (76.5%) | 32,902 (77.1%) | -0.01 |
| Lab result number- HDL level (mg/dl) mean (only | 11,015 (50.476) | 11,075 (50.770) | 21,032 (33.470) | 21,025 (54.270) | 19/6 | N/A | 32,043 (70.370) | 32,302 (77.170) | 0.01 |
| | 7 420 | 7 220 | 1.520 | 1 204 | 21/2 | N/A | 8,966 | 8,623 | |
| =<5000 included) | 7,438 | 7,329 | 1,528 | 1,294 | N/A | • | | | |
| mean (sd) | 44.89 (13.09) | 44.78 (12.83) | 43.55 (14.91) | 43.02 (13.62) | N/A | N/A | 44.66 (13.42) | 44.52 (12.95) | 0.01 |
| median [IQR] | 43.00 [36.00, 51.50] | 43.00 [36.00, 52.00] | 42.83 [35.00, 51.00] | 42.00 [35.00, 50.00] | N/A | N/A | 42.97 (13.42) | 42.85 (12.95) | 0.01 |
| Missing; n (%) | 12,094 (61.9%) | 12,203 (62.5%) | 21,640 (93.4%) | 21,874 (94.4%) | N/A | N/A | 33,734 (79.0%) | 34,077 (79.8%) | -0.02 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | |
| =<5000 included) | 7,492 | 7,432 | 1,416 | 1,187 | N/A | N/A | 8,908 | 8,619 | |
| mean (sd) | 85.61 (39.60) | 84.29 (39.26) | 87.73 (41.40) | 87.33 (40.93) | N/A | N/A | 85.95 (39.89) | 84.71 (39.50) | 0.03 |
| median [IQR] | 83.00 [62.00, 109.00] | 82.00 [61.00, 106.00] | 87.00 [64.00, 113.00] | 88.00 [63.00, 112.00] | N/A | N/A | 83.64 (39.89) | 82.83 (39.50) | 0.02 |
| Missing; n (%) | 12,040 (61.6%) | 12,100 (61.9%) | 21,752 (93.9%) | 21,981 (94.9%) | N/A | N/A | 33,792 (79.1%) | 34,081 (79.8%) | -0.02 |
| Lab result number-Total cholesterol (mg/dl) mean | 12,0.0 (01.0/0) | 12,100 (01.570) | 21,752 (55.570) | 22,552 (5 7.570) | /^ | // | 33,732 (73.170) | 5 1,001 (7 5.070) | 3.02 |
| (only =<5000 included) | 7,541 | 7,474 | 1,534 | 1,304 | N/A | N/A | 9,075 | 8.778 | |
| | | | | | • | • | | -, | 2.25 |
| mean (sd) | 173.51 (47.47) | 172.60 (46.68) | 172.33 (52.31) | 173.37 (48.27) | N/A | N/A | 173.31 (48.32) | 172.71 (46.92) | 0.01 |
| median [IQR] | 167.00 [142.00, 198.25] | | 170.00 [143.38, 199.50] | 171.00 [147.00, 198.00] | N/A | N/A | 167.51 (48.32) | 167.59 (46.92) | 0.00 |
| Missing; n (%) | 11,991 (61.4%) | 12,058 (61.7%) | 21,634 (93.4%) | 21,864 (94.4%) | N/A | N/A | 33,625 (78.7%) | 33,922 (79.4%) | -0.02 |

| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only =<5000 included) | 7,489 | 7,436 | 1,511 | 1,283 | N/A | N/A | 9,000 | 8,719 | |
| mean (sd) | 197.03 (176.04) | 200.03 (177.75) | 188.47 (180.91) | 204.69 (194.45) | N/A | N/A | 195.59 (176.88) | 200.72 (180.31) | -0.03 |
| median [IQR] | 158.00 [112.00, 228.00] | 161.00 [114.00, 230.92] | 150.50 [104.50, 223.33] | 163.00 [113.00, 237.00] | N/A | N/A | 156.74 (176.88) | 161.29 (180.31) | -0.03 |
| Missing; n (%) | 12,043 (61.7%) | 12,096 (61.9%) | 21,657 (93.5%) | 21,885 (94.5%) | N/A | N/A | 33,700 (78.9%) | 33,981 (79.6%) | -0.02 |
| Lab result number- Hemoglobin mean (only >0 | E 576 | E 401 | 1.022 | 879 | N/A | NI/A | 6 600 | 6 360 | |
| included)<br>mean (sd) | 5,576<br>13.80 (1.57) | 5,481<br>14.00 (1.57) | 1,032<br>20,324.36 (440,120.87) | 3,301.14 (20,906.38) | N/A<br>N/A | N/A<br>N/A | 6,608<br>3185.79 (173886.11) | 6,360<br>468.31 (7769.62) | 0.02 |
| median [IQR] | 13.80 [12.71, 14.80] | 14.00 [12.90, 15.08] | 13.70 [12.70, 14.80] | 14.00 [12.90, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 13,956 (71.5%) | 14,051 (71.9%) | 22,136 (95.5%) | 22,289 (96.2%) | N/A | N/A | 36,092 (84.5%) | 36,340 (85.1%) | -0.02 |
| Lab result number- Serum sodium mean (only > 90 | | - 1,000 (1 -101-1) | ,, | | | | 00,000 (0) | , (, | ***- |
| and < 190 included) | 8,349 | 8,307 | 1,543 | 1,339 | N/A | N/A | 9,892 | 9,646 | |
| mean (sd) | 139.26 (2.68) | 139.23 (2.69) | 138.98 (2.54) | 138.92 (2.39) | N/A | N/A | 139.22 (2.66) | 139.19 (2.65) | 0.01 |
| median [IQR] | 139.33 [138.00, 141.00] | 139.00 [138.00, 141.00] | 139.00 [137.33, 140.62] | 139.00 [137.00, 140.33] | N/A | N/A | 139.28 (2.66) | 139.00 (2.65) | 0.11 |
| Missing; n (%) | 11,183 (57.3%) | 11,225 (57.5%) | 21,625 (93.3%) | 21,829 (94.2%) | N/A | N/A | 32,808 (76.8%) | 33,054 (77.4%) | -0.01 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 7,829 | 7,803 | 1,323 | 1,145 | N/A | N/A | 9,152 | 8,948 | |
| mean (sd) | 4.29 (0.31) | 4.30 (0.30) | 4.15 (0.71) | 4.17 (0.66) | N/A | N/A | 4.27 (0.39) | 4.28 (0.37) | -0.03 |
| median [IQR]<br>Missing; n (%) | 4.30 [4.10, 4.50]<br>11,703 (59.9%) | 4.30 [4.10, 4.50]<br>11,729 (60.1%) | 4.25 [4.00, 4.45]<br>21,845 (94.3%) | 4.25 [4.00, 4.50]<br>22,023 (95.1%) | N/A<br>N/A | N/A<br>N/A | 4.29 (0.39)<br>33,548 (78.6%) | 4.29 (0.37)<br>33,752 (79.0%) | 0.00<br>-0.01 |
| Lab result number- Glucose (fasting or random) mean | 11,705 (59.9%) | 11,729 (00.1%) | 21,045 (94.5%) | 22,023 (93.1%) | IN/A | IN/A | 33,346 (76.0%) | 33,732 (79.0%) | -0.01 |
| (only 10-1000 included) | 8,366 | 8,303 | 1,537 | 1,326 | N/A | N/A | 9,903 | 9,629 | |
| mean (sd) | 180.41 (72.14) | 181.43 (70.42) | 181.84 (71.36) | 182.28 (68.00) | N/A | N/A | 180.63 (72.02) | 181.55 (70.10) | -0.01 |
| median [IQR] | 163.50 [130.00, 214.00] | 166.50 [132.00, 216.00] | 165.00 [132.33, 215.75] | 168.25 [134.00, 217.12] | N/A | N/A | 163.73 (72.02) | 166.74 (70.10) | -0.04 |
| Missing; n (%) | 11,166 (57.2%) | 11,229 (57.5%) | 21,631 (93.4%) | 21,842 (94.3%) | N/A | N/A | 32,797 (76.8%) | 33,071 (77.4%) | -0.01 |
| Lab result number- Potassium mean (only 1-7 | | | | | | | | | |
| included) | 8,517 | 8,468 | 1,538 | 1,307 | N/A | N/A | 10,055 | 9,775 | |
| mean (sd) | 4.45 (0.42) | 4.45 (0.41) | 4.36 (0.44) | 4.36 (0.44) | N/A | N/A | 4.44 (0.42) | 4.44 (0.41) | 0.00 |
| median [IQR] | 4.40 [4.20, 4.70] | 4.40 [4.20, 4.70] | 4.35 [4.00, 4.60] | 4.40 [4.10, 4.60] | N/A | N/A | 4.39 (0.42) | 4.40 (0.41) | -0.02 |
| Missing; n (%) | 11,015 (56.4%) | 11,064 (56.6%) | 21,630 (93.4%) | 21,861 (94.4%) | N/A | N/A | 32,645 (76.5%) | 32,925 (77.1%) | -0.01 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10mean (sd) | 2.09 (1.28) | 2.10 (1.31) | 1.67 (1.00) | 1.67 (1.00) | 2.36 (1.50) | 2.35 (1.50) | 2.08 (1.31) | 2.08 (1.32) | 0.00 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.70 (1.31) | 1.70 (1.32) | 0.00 |
| Frailty Score: Qualitative Version 365 days as | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | 1.70 (1.51) | 1.70 (1.52) | 0.00 |
| Categories, v1 | | | | | | | | | |
| 0; n (%) | 13,009 (66.6%) | 12,920 (66.1%) | 12,672 (54.7%) | 12,648 (54.6%) | 15,535 (46.5%) | 15,495 (46.4%) | 41,216 (54.2%) | 41,063 (54.0%) | 0.00 |
| 1 to 2; n (%) | 5,078 (26.0%) | 5,112 (26.2%) | 8,472 (36.6%) | 8,480 (36.6%) | 11,515 (34.5%) | 11,612 (34.8%) | 25,065 (32.9%) | 25,204 (33.1%) | 0.00 |
| 3 or more; n (%) | 1,445 (7.4%) | 1,500 (7.7%) | 2,024 (8.7%) | 2,040 (8.8%) | 6,351 (19.0%) | 6,294 (18.8%) | 9,820 (12.9%) | 9,834 (12.9%) | 0.00 |
| Frailty Score: Empirical Version 365 days as | | | | | | | | | |
| Categories, | | | | | | | | | |
| <0.12908; n (%) | 6,873 (35.2%) | 6,844 (35.0%) | 7,705 (33.3%) | 7,732 (33.4%) | 5,501 (16.5%) | 5,302 (15.9%) | 20,079 (26.4%) | 19,878 (26.1%) | 0.01 |
| 0.12908 - 0.1631167; n (%)<br>>= 0.1631167; n (%) | 7,260 (37.2%)<br>5,399 (27.6%) | 7,324 (37.5%)<br>5,364 (27.5%) | 9,157 (39.5%)<br>6,306 (27.2%) | 9,149 (39.5%)<br>6,287 (27.1%) | 10,406 (31.2%)<br>17,494 (52.4%) | 10,542 (31.6%)<br>17,557 (52.6%) | 26,823 (35.2%)<br>29,199 (38.4%) | 27,015 (35.5%)<br>29,208 (38.4%) | -0.01<br>0.00 |
| >= 0.1031107, 11 (%)<br>Non-Frailty; n (%) | 11,171 (57.2%) | 11,285 (57.8%) | 12,238 (52.8%) | 12,310 (53.1%) | 1,723 (5.2%) | 1,549 (4.6%) | 25,132 (33.0%) | 25,144 (33.0%) | 0.00 |
| Non Trailey, 11 (70) | 11,171 (37.270) | 11,203 (37.070) | 12,230 (32.0%) | 12,310 (55.170) | 1,723 (3.270) | 1,545 (4.070) | 25,152 (55.070) | 23,144 (33.070) | 0.00 |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 0.63 (1.18) | 0.64 (1.18) | 0.81 (1.19) | 0.82 (1.20) | 1.26 (1.67) | 1.25 (1.64) | 0.96 (1.42) | 0.96 (1.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.44 (1.42) | 0.44 (1.41) | 0.00 |
| Frailty Score (mean): Empirical Version 365 days, | | | | | | | | | |
| mean (sd) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.04) | 0.14 (0.04) | 0.18 (0.05) | 0.18 (0.05) | 0.16 (0.04) | 0.16 (0.04) | 0.00 |
| median [IQR] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.16] | 0.14 [0.12, 0.16] | 0.17 [0.14, 0.20] | 0.17 [0.14, 0.20] | 0.15 (0.04) | 0.15 (0.04) | 0.00 |
| Healthcare Utilization | | | | | | | | | |
| Any hospitalization; n (%) | 451 (2.3%) | 488 (2.5%) | 496 (2.1%) | 517 (2.2%) | 1,265 (3.8%) | 1,237 (3.7%) | 2,212 (2.9%) | 2,242 (2.9%) | 0.00 |
| Any hospitalization within prior 30 days; n (%) | 62 (0.3%)<br>394 (2.0%) | 83 (0.4%)<br>409 (2.1%) | 64 (0.3%)<br>436 (1.9%) | 79 (0.3%)<br>441 (1.9%) | 198 (0.6%) | 207 (0.6%)<br>1,057 (3.2%) | 324 (0.4%)<br>1,924 (2.5%) | 369 (0.5%)<br>1,907 (2.5%) | -0.01<br>0.00 |
| Any hospitalization during prior 31-180 days; n (%)<br>Endocrinologist Visit; n (%) | 2,773 (14.2%) | 2,878 (14.7%) | 3,445 (14.9%) | 3,370 (14.5%) | 1,094 (3.3%)<br>5,826 (17.4%) | 5,874 (17.6%) | 12,044 (15.8%) | 1,907 (2.5%) | 0.00 |
| Endocrinologist Visit, IT(%) Endocrinologist Visit (30 days prior); n (%) | 1,974 (10.1%) | 2,042 (10.5%) | 2,569 (11.1%) | 2,555 (11.0%) | 4,001 (12.0%) | 4,092 (12.3%) | 8,544 (11.2%) | 8,689 (11.4%) | -0.01 |
| Endocrinologist Visit (30 days prior); n (%) | 1,939 (9.9%) | 1,992 (10.2%) | 2,311 (10.0%) | 2,302 (9.9%) | 4,404 (13.2%) | 4,479 (13.4%) | 8,654 (11.4%) | 8,773 (11.5%) | 0.00 |
| Internal medicine/family medicine visits; n (%) | 14,481 (74.1%) | 14,301 (73.2%) | 20,561 (88.7%) | 20,392 (88.0%) | 27,892 (83.5%) | 27,600 (82.6%) | 62,934 (82.7%) | 62,293 (81.9%) | 0.02 |
| Internal medicine/family medicine visits (30 days | , - , =, | , , . =/ | , (/ | | / | | | | |
| prior) ; n (%) | 10,679 (54.7%) | 10,582 (54.2%) | 15,756 (68.0%) | 15,756 (68.0%) | 20,325 (60.9%) | 20,166 (60.4%) | 46,760 (61.4%) | 46,504 (61.1%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | |
| days prior); n (%) | 12,286 (62.9%) | 12,278 (62.9%) | 16,906 (73.0%) | 16,939 (73.1%) | 24,413 (73.1%) | 24,255 (72.6%) | 53,605 (70.4%) | 53,472 (70.3%) | 0.00 |
| Cardiologist visit; n (%) | 3,671 (18.8%) | 3,733 (19.1%) | 3,785 (16.3%) | 3,767 (16.3%) | 9,403 (28.2%) | 9,408 (28.2%) | 16,859 (22.2%) | 16,908 (22.2%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 1,085 (5.6%) | 1,159 (5.9%) | 1,191 (5.1%) | 1,155 (5.0%) | 2,831 (8.5%) | 2,875 (8.6%) | 5,107 (6.7%) | 5,189 (6.8%) | 0.00 |

| Number of Cardiologist visits (31 to 180 days prior) | ): | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| n (%) | 3,120 (16.0%) | 3,172 (16.2%) | 3,152 (13.6%) | 3,189 (13.8%) | 8,218 (24.6%) | 8,170 (24.5%) | 14,490 (19.0%) | 14,531 (19.1%) | 0.00 |
| Electrocardiogram ; n (%) | 4,420 (22.6%) | 4,428 (22.7%) | 5,282 (22.8%) | 5,287 (22.8%) | 9,495 (28.4%) | 9,314 (27.9%) | 19,197 (25.2%) | 19,029 (25.0%) | 0.00 |
| Use of glucose test strips; n (%) | 684 (3.5%) | 679 (3.5%) | 913 (3.9%) | 898 (3.9%) | 981 (2.9%) | 1,014 (3.0%) | 2,578 (3.4%) | 2,591 (3.4%) | 0.00 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Naive new user v8 ; n (%) | 1,875 (9.6%) | 1,885 (9.7%) | 1,971 (8.5%) | 1,989 (8.6%) | 1,878 (5.6%) | 1,925 (5.8%) | 5,724 (7.5%) | 5,799 (7.6%) | 0.00 |
| N antidiabetic drugs at index date | | | | | | | | | |
| mean (sd) | 2.35 (0.86) | 2.35 (0.88) | 2.35 (0.87) | 2.35 (0.90) | 2.42 (0.86) | 2.42 (0.87) | 2.38 (0.86) | 2.38 (0.88) | 0.00 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 (0.86) | 2.00 (0.88) | 0.00 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 9.98 (4.40) | 9.99 (4.31) | 9.72 (4.22) | 9.71 (4.07) | 10.35 (4.25) | 10.32 (4.12) | 10.06 (4.28) | 10.05 (4.15) | 0.00 |
| median [IQR] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 10.00 [7.00, 13.00] | 10.00 [7.00, 13.00] | 9.44 (4.28) | 9.44 (4.15) | 0.00 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.03 (0.17) | 0.03 (0.18) | 0.02 (0.16) | 0.02 (0.16) | 0.04 (0.23) | 0.04 (0.23) | 0.03 (0.20) | 0.03 (0.20) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.20) | 0.00 (0.20) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 0.11 (1.04) | 0.12 (1.01) | 0.10 (0.84) | 0.11 (0.90) | 0.22 (1.39) | 0.22 (1.68) | 0.16 (1.16) | 0.16 (1.32) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.16) | 0.00 (1.32) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.21 (0.70) | 0.21 (0.77) | 0.05 (0.98) | 0.05 (0.79) | 0.30 (1.13) | 0.30 (1.03) | 0.20 (0.99) | 0.20 (0.90) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.99) | 0.00 (0.90) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 4.20 (3.19) | 4.18 (3.01) | 4.16 (3.17) | 4.15 (3.01) | 4.97 (3.57) | 4.95 (3.49) | 4.53 (3.36) | 4.51 (3.23) | 0.01 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 7.00] | 4.00 [3.00, 6.00] | 3.44 (3.36) | 3.44 (3.23) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.69 (2.71) | 0.74 (2.81) | 0.71 (2.77) | 0.75 (2.94) | 1.01 (3.82) | 1.13 (4.36) | 0.84 (3.26) | 0.91 (3.61) | -0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.26) | 0.00 (3.61) | 0.00 |
| Number of internal medicine/family medicine visits | s | | | | | | | | |
| mean (sd) | 7.21 (12.35) | 7.16 (10.75) | 6.39 (7.36) | 6.54 (7.69) | 7.45 (9.63) | 7.60 (9.85) | 7.07 (9.82) | 7.16 (9.50) | -0.01 |
| median [IQR] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 8.00] | 4.00 [2.00, 9.00] | 5.00 [2.00, 10.00] | 5.00 [2.00, 10.00] | 4.44 (9.82) | 4.44 (9.50) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 0.77 (2.66) | 0.76 (2.51) | 0.64 (2.39) | 0.62 (2.14) | 1.32 (3.64) | 1.33 (3.67) | 0.97 (3.06) | 0.97 (2.99) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (3.06) | 0.00 (2.99) | 0.00 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd) | 0.35 (0.83) | 0.35 (0.86) | 0.34 (0.82) | 0.34 (0.81) | 0.49 (1.03) | 0.48 (1.05) | 0.41 (0.92) | 0.40 (0.93) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.92) | 0.00 (0.93) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 1.35 (0.88) | 1.35 (0.86) | 1.26 (0.88) | 1.26 (0.86) | 1.56 (0.86) | 1.56 (0.80) | 1.41 (0.87) | 1.41 (0.83) | 0.00 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.44 (0.87) | 1.44 (0.83) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.42 (1.48) | 0.42 (1.17) | 0.39 (0.99) | 0.40 (1.12) | 0.43 (1.03) | 0.43 (1.07) | 0.42 (1.15) | 0.42 (1.11) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.15) | 0.00 (1.11) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 1.05 (0.93) | 1.05 (0.93) | 1.04 (1.21) | 1.04 (1.19) | 1.11 (0.84) | 1.10 (0.82) | 1.07 (0.99) | 1.07 (0.97) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (0.99) | 1.00 (0.97) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.03 (0.22) | 0.03 (0.22) | 0.04 (0.24) | 0.04 (0.24) | 0.06 (0.32) | 0.07 (0.33) | 0.05 (0.27) | 0.05 (0.28) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.27) | 0.00 (0.28) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.02 (0.16) | 0.02 (0.16) | 0.02 (0.18) | 0.02 (0.17) | 0.04 (0.25) | 0.04 (0.26) | 0.03 (0.21) | 0.03 (0.21) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.21) | 0.00 (0.21) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | |
| mean (sd) | 0.83 (1.17) | 0.83 (1.15) | 0.74 (1.09) | 0.73 (1.09) | 0.53 (0.72) | 0.53 (0.72) | 0.67 (0.97) | 0.67 (0.96) | 0.00 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.97) | 0.00 (0.96) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | |
| digit level | E EQ (E 22) | E E4 /E CC) | 2.40/2.201 | 2 42 (2 25) | E 02 (C 00) | E 7E (C 02) | 4.66 (5.76) | 4.50/5.72\ | 0.04 |
| mean (sd) | 5.59 (5.88) | 5.54 (5.90) | 2.18 (3.30) | 2.12 (3.35) | 5.83 (6.80) | 5.75 (6.82) | 4.66 (5.70) | 4.59 (5.72) | 0.01 |
| median [IQR] | 5.00 [0.00, 8.00] | 5.00 [0.00, 8.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 3.04 (5.70) | 3.04 (5.72) | 0.00 |
| Hea of this side on (9/) | 2 545 (12 09/) | 2 522 /12 00/\ 2 0 | 22 /12 79/\ | 2 040 /12 70/\ 5 / | 006 (15 00/) | E 034/1E 00/\ 10.4 | 04/12/00/\ | 10 505 (12 00/) | 0.00 |
| Use of thiazide; n (%) | 2,545 (13.0%) | 2,533 (13.0%) 2,9 | | 2,948 (12.7%) 5,0 | | 5,024 (15.0%) 10,4 | | 10,505 (13.8%) | 0.00 |
| Use of beta blockers; n (%) Use of calcium channel blockers; n (%) | 7,182 (36.8%)<br>5,692 (29.1%) | 7,314 (37.4%) 8,2<br>5,762 (29.5%) 6,7 | | 8,226 (35.5%) 16<br>6,841 (29.5%) 11 | | 16,300 (48.8%) 31,6<br>11,422 (34.2%) 23,7 | | 31,840 (41.8%)<br>24,025 (31.6%) | -0.01 |
| Ose of carcium channer brockers, if (76) | 3,032 (23.170) | 3,/02 (23.3%) 6,/ | 134 (23.370) | 0,041(23.3%) 11 | ,240 (33.7%) | 11,422 (34.2%) 23,7 | 32 (31.270) | 24,023 (31.0%) | -0.01 |

Appendix B: Canagliflozin vs 2nd Generation Sulfonylureas



| ĺ | Optu | m | Market | Scan | Medicare | | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| | Reference- 2nd | | Reference-2nd | | Reference-2nd | Exposure- | Reference-2nd | | |
| Variable | Generation SUs<br>154,886 | Exposure- Canagliflozin | Generation SUs<br>132,040 | Exposure-Canagliflozin | Generation SUs<br>385,432 | Canagliflozin<br>28,987 | Generation SUs<br>672,358 | Exposure- Canagliflozin<br>70,459 | St. Diff. |
| Number of patients Age | 154,886 | 17,154 | 132,040 | 24,318 | 385,432 | 28,987 | 672,358 | 70,459 | |
| mean (sd) | 67.76 (9.26) | 61.96 (7.84) | 62.52 (9.22) | 59.18 (6.40) | 73.86 (7.06) | 71.03 (5.27) | 70.23 (8.06) | 64.73 (6.37) | 0.76 |
| median [IQR] | 68.00 [61.00, 74.00] | 61.00 [56.00, 67.00] | 61.00 [56.00, 67.00] | 59.00 [54.00, 63.00] | 72.00 [68.00, 78.00] 0. | | 68.92 (8.06) | 64.01 (6.37) | 0.68 |
| Age categories | 00.00 [01.00, 74.00] | 01.00 [50.00, 07.00] | 01.00 [50.00, 07.00] | 33.00 [34.00, 03.00] | 72.00 [00.00, 70.00] 5. | 00 [07.00, 74.00] | 00.32 (0.00) | 04.01 (0.57) | 0.00 |
| 18 - 54; n (%) | 14,732 (9.5%) | 3,424 (20.0%) | 25,558 (19.4%) | 6,293 (25.9%) | 0 (0.0%) | 0 (0.0%) | 40,290 (6.0%) | 9,717 (13.8%) | -0.26 |
| 55 - 64; n (%) | 38,435 (24.8%) | 7,427 (43.3%) | 66,089 (50.1%) | 14,196 (58.4%) | 5,075 (1.3%) | 329 (1.1%) | 109,599 (16.3%) | 21,952 (31.2%) | -0.36 |
| 65 - 74; n (%) | 65,092 (42.0%) | 5,148 (30.0%) | 24,049 (18.2%) | 3,180 (13.1%) | 227,622 (59.1%) | 22,378 (77.2%) | 316,763 (47.1%) | 30,706 (43.6%) | 0.07 |
| >= 75; n (%) | 36,627 (23.6%) | 1,155 (6.7%) | 16,344 (12.4%) | 649 (2.7%) | 152,735 (39.6%) | 6,280 (21.7%) | 205,706 (30.6%) | 8,084 (11.5%) | 0.48 |
| Gender | | | | | | | | | |
| Males; n (%) | 80,936 (52.3%) | 9,575 (55.8%) | 74,065 (56.1%) | 13,608 (56.0%) | 176,834 (45.9%) | 14,378 (49.6%) | 331,835 (49.4%) | 37,561 (53.3%) | -0.08 |
| Females; n (%) | 73,950 (47.7%) | 7,579 (44.2%) | 57,975 (43.9%) | 10,710 (44.0%) | 208,598 (54.1%) | 14,609 (50.4%) | 340,523 (50.6%) | 32,898 (46.7%) | 0.08 |
| Race | 21/2 | N1/A | 21/2 | N1/A | 293,566 (76.2%) | 23,286 (80.3%) | 293,566 (76.2%) | 22 200 (00 20/) | -0.10 |
| White; n (%)<br>Black; n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | 46,063 (12.0%) | 2,353 (8.1%) | 46,063 (12.0%) | 23,286 (80.3%)<br>2,353 (8.1%) | 0.10 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 14,026 (3.6%) | 1,041 (3.6%) | 14,026 (3.6%) | 1,041 (3.6%) | 0.00 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 15,651 (4.1%) | 982 (3.4%) | 15,651 (4.1%) | 982 (3.4%) | 0.04 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 2,642 (0.7%) | 116 (0.4%) | 2,642 (0.7%) | 116 (0.4%) | 0.04 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 13,484 (3.5%) | 1,209 (4.2%) | 13,484 (3.5%) | 1,209 (4.2%) | -0.04 |
| | • | • | | • | | , | | | |
| Region (lumping missing&other category with West) | 16 655 (10 00/) | 1 460 (0 60/) | 24 642 (46 40/) | 4 500 (10 00/) | C2 475 (1C 50/) | E 472 (40 00/) | 101 772 (15 10/) | 11 540 (16 49/) | 0.04 |
| Northeast; n (%) | 16,655 (10.8%)<br>74,258 (47.9%) | 1,468 (8.6%)<br>9,215 (53.7%) | 21,643 (16.4%)<br>33,357 (25.3%) | 4,599 (18.9%)<br>4,231 (17.4%) | 63,475 (16.5%)<br>162,072 (42.0%) | 5,473 (18.9%)<br>12,619 (43.5%) | 101,773 (15.1%)<br>269,687 (40.1%) | 11,540 (16.4%)<br>26,065 (37.0%) | -0.04<br>0.06 |
| South; n (%)<br>Midwest; n (%) | 31,842 (20.6%) | 3,552 (20.7%) | 57,680 (43.7%) | 12,979 (53.4%) | 95,692 (24.8%) | 5,876 (20.3%) | 185,214 (27.5%) | 22,407 (31.8%) | -0.09 |
| West; n (%) | 32,131 (20.7%) | 2,919 (17.0%) | 17,703 (13.4%) | 2,224 (9.1%) | 64,193 (16.7%) | 5,019 (17.3%) | 114,027 (17.0%) | 10,162 (14.4%) | 0.03 |
| Unknown+missing; n (%) | N/A | N/A | 1,657 (1.3%) | 285 (1.2%) | N/A | N/A | 1,657 (1.3%) | 285 (1.2%) | 0.01 |
| CV Covariates | | .4 | _,, | | .4 | .,, | _,, | | |
| Ischemic heart disease; n (%) | 28,161 (18.2%) | 2,488 (14.5%) | 18,313 (13.9%) | 2,973 (12.2%) | 100,011 (25.9%) | 7,262 (25.1%) | 146,485 (21.8%) | 12,723 (18.1%) | 0.09 |
| Acute MI; n (%) | 644 (0.4%) | 39 (0.2%) | 444 (0.3%) | 58 (0.2%) | 1,926 (0.5%) | 101 (0.3%) | 3,014 (0.4%) | 198 (0.3%) | 0.02 |
| ACS/unstable angina; n (%) | 778 (0.5%) | 76 (0.4%) | 524 (0.4%) | 81 (0.3%) | 2,195 (0.6%) | 149 (0.5%) | 3,497 (0.5%) | 306 (0.4%) | 0.01 |
| Old MI; n (%) | 3,799 (2.5%) | 290 (1.7%) | 1,411 (1.1%) | 196 (0.8%) | 11,166 (2.9%) | 703 (2.4%) | 16,376 (2.4%) | 1,189 (1.7%) | 0.05 |
| Stable angina; n (%) | 4,163 (2.7%) | 350 (2.0%) | 2,056 (1.6%) | 318 (1.3%) | 10,964 (2.8%) | 864 (3.0%) | 17,183 (2.6%) | 1,532 (2.2%) | 0.03 |
| Coronary atherosclerosis and other forms of chronic | 26,304 (17.0%) | 2 255 (42 70/) | 17,287 (13.1%) | 2 011 (11 00/) | 06 007 (24 0%) | C 054 (24 00/) | 120 500 (20 00/) | 12 120 (17 20/) | 0.09 |
| ischemic heart disease; n (%) Other atherosclerosis with ICD10 Copy; n (%) | 26,304 (17.0%)<br>962 (0.6%) | 2,355 (13.7%)<br>74 (0.4%) | 670 (0.5%) | 2,811 (11.6%)<br>132 (0.5%) | 96,007 (24.9%)<br>4,672 (1.2%) | 6,954 (24.0%)<br>340 (1.2%) | 139,598 (20.8%)<br>6,304 (0.9%) | 12,120 (17.2%)<br>546 (0.8%) | 0.09 |
| Other atheroscierosis with 16010 Copy, 11 (76) | 302 (0.0%) | 74 (0.476) | 070 (0.3%) | 132 (0.3%) | 4,072 (1.270) | 340 (1.276) | 0,304 (0.376) | 340 (0.8%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent); n (%) | 256 (0.2%) | 18 (0.1%) | 227 (0.2%) | 32 (0.1%) | 734 (0.2%) | 53 (0.2%) | 1,217 (0.2%) | 103 (0.1%) | 0.03 |
| History of CABG or PTCA; n (%) | 6,458 (4.2%) | 505 (2.9%) | 2,302 (1.7%) | 345 (1.4%) | 24,925 (6.5%) | 1,676 (5.8%) | 33,685 (5.0%) | 2,526 (3.6%) | 0.07 |
| Any stroke; n (%) | 5,514 (3.6%) | 452 (2.6%) | 3,637 (2.8%) | 480 (2.0%) | 22,740 (5.9%) | 1,588 (5.5%) | 31,891 (4.7%) | 2,520 (3.6%) | 0.06 |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | |
| infarction); n (%) | 5,460 (3.5%) | 449 (2.6%) | 3,611 (2.7%) | 475 (2.0%) | 22,597 (5.9%) | 1,580 (5.5%) | 31,668 (4.7%) | 2,504 (3.6%) | 0.06 |
| Hemorrhagic stroke; n (%) | 72 (0.0%) | 5 (0.0%) | 44 (0.0%) | 6 (0.0%) | 231 (0.1%) | 11 (0.0%) | 347 (0.1%) | 22 (0.0%) | 0.04 |
| TIA; n (%) | 654 (0.4%) | 52 (0.3%) | 432 (0.3%) | 47 (0.2%) | 2,582 (0.7%) | 152 (0.5%) | 3,668 (0.5%) | 251 (0.4%) | 0.01<br>0.05 |
| Other cerebrovascular disease; n (%) Late effects of cerebrovascular disease; n (%) | 1,586 (1.0%)<br>1,489 (1.0%) | 109 (0.6%)<br>77 (0.4%) | 842 (0.6%)<br>610 (0.5%) | 98 (0.4%)<br>50 (0.2%) | 6,208 (1.6%)<br>5,373 (1.4%) | 332 (1.1%)<br>244 (0.8%) | 8,636 (1.3%)<br>7,472 (1.1%) | 539 (0.8%)<br>371 (0.5%) | 0.03 |
| Cerebrovascular procedure; n (%) | 71 (0.0%) | 5 (0.0%) | 44 (0.0%) | 4 (0.0%) | 239 (0.1%) | 17 (0.1%) | 354 (0.1%) | 26 (0.0%) | 0.04 |
| Heart failure (CHF); n (%) | 10,952 (7.1%) | 634 (3.7%) | 5,273 (4.0%) | 480 (2.0%) | 36,922 (9.6%) | 2,004 (6.9%) | 53,147 (7.9%) | 3,118 (4.4%) | 0.15 |
| , , , , | . , , | , , | . , , | , , | . , , | . , , | . , , | . , , | |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n (%) | 9,275 (6.0%) | 729 (4.2%) | 4,752 (3.6%) | 643 (2.6%) | 34,887 (9.1%) | 2,314 (8.0%) | 48,914 (7.3%) | 3,686 (5.2%) | 0.09 |
| Atrial fibrillation; n (%) | 10,323 (6.7%) | 740 (4.3%) | 6,297 (4.8%) | 765 (3.1%) | 41,954 (10.9%) | 2,419 (8.3%) | 58,574 (8.7%) | 3,924 (5.6%) | 0.12 |
| Other cardiac dysrhythmia; n (%) | 12,809 (8.3%) | 896 (5.2%) | 6,775 (5.1%) | 799 (3.3%) | 43,918 (11.4%) | 2,772 (9.6%) | 63,502 (9.4%) | 4,467 (6.3%) | 0.12 |
| Cardiac conduction disorders; n (%) | 3,451 (2.2%) | 225 (1.3%) | 1,828 (1.4%) | 211 (0.9%) | 12,984 (3.4%) | 758 (2.6%) | 18,263 (2.7%) | 1,194 (1.7%) | 0.07 |
| Other CVD; n (%) | 13,518 (8.7%) | 1,010 (5.9%) | 8,464 (6.4%) | 1,176 (4.8%) | 48,376 (12.6%) | 3,167 (10.9%) | 70,358 (10.5%) | 5,353 (7.6%) | 0.10 |
| Diabetes-related complications Diabetic retinopathy; n (%) | 8,707 (5.6%) | 978 (5.7%) | 4,265 (3.2%) | 1,010 (4.2%) | 22,583 (5.9%) | 2,188 (7.5%) | 35,555 (5.3%) | 4,176 (5.9%) | -0.03 |
| Diadetic retinopatity, it (/0) | (%0.5) / ۵٫/۵۸ | 3/0(3./%) | 4,203 (3.2%) | 1,010 (4.2%) | 22,303 (3.3%) | 2,100 (7.370) | 33,333 (3.3%) | 4,170 (3.3%) | -0.03 |
| Diabetes with other ophthalmic manifestations; n (%) | 1,194 (0.8%) | 100 (0.6%) | 2,603 (2.0%) | 618 (2.5%) | 8,498 (2.2%) | 828 (2.9%) | 12,295 (1.8%) | 1,546 (2.2%) | -0.03 |
| Retinal detachment, vitreous hemorrhage, vitrectomy; n | | | | | | | | | |
| (%) | 541 (0.3%) | 61 (0.4%) | 305 (0.2%) | 64 (0.3%) | 1,186 (0.3%) | 119 (0.4%) | 2,032 (0.3%) | 244 (0.3%) | 0.00 |
| Retinal laser coagulation therapy; n (%) Occurrence of Diabetic Neuropathy Copy; n (%) | 711 (0.5%)<br>25,944 (16.8%) | 104 (0.6%)<br>2,962 (17.3%) | 514 (0.4%)<br>12,232 (9.3%) | 115 (0.5%)<br>2,705 (11.1%) | 1,635 (0.4%)<br>61,265 (15.9%) | 205 (0.7%)<br>5,766 (19.9%) | 2,860 (0.4%)<br>99,441 (14.8%) | 424 (0.6%)<br>11,433 (16.2%) | -0.03<br>-0.04 |
| occurrence of Diabetic Neuropathy Copy; ft (%) | 23,944 (10.8%) | 2,302 (11.3%) | 12,232 (9.3%) | 2,/05 (11.1%) | 01,205 (15.3%) | 3,700 (19.9%) | 33,441 (14.8%) | 11,433 (10.2%) | -0.04 |

| Occurrence of diabetic nephropathy with ICD10 Copy; n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (%) | 23,516 (15.2%) | 1,648 (9.6%) | 8,598 (6.5%) | 1,283 (5.3%) | 37,114 (9.6%) | 2,340 (8.1%) | 69,228 (10.3%) | 5,271 (7.5%) | 0.10 |
| Hypoglycemia ; n (%) | 2,683 (1.7%) | 357 (2.1%) | 2,848 (2.2%) | 594 (2.4%) | 7,156 (1.9%) | 660 (2.3%) | 12,687 (1.9%) | 1,611 (2.3%) | -0.03 |
| Hyperglycemia; n (%) | 5,729 (3.7%) | 582 (3.4%) | 3,944 (3.0%) | 627 (2.6%) | 15,025 (3.9%) | 1,020 (3.5%) | 24,698 (3.7%) | 2,229 (3.2%) | 0.03 |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 8,950 (5.8%) | 552 (3.2%) | 4,904 (3.7%) | 534 (2.2%) | 25,824 (6.7%) | 1,227 (4.2%) | 39,678 (5.9%) | 2,313 (3.3%) | 0.12 |
| Diabetic ketoacidosis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 00 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome | 0 (0.0%) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 0 (0.070) | 000 (0.0%) | 00 (0.070) | |
| (HONK); n (%) | 677 (0.4%) | 76 (0.4%) | 472 (0.4%) | 73 (0.3%) | 1,573 (0.4%) | 144 (0.5%) | 2,722 (0.4%) | 293 (0.4%) | 0.00 |
| Diabetes with peripheral circulatory disorders with ICD- | | | | | | | | | |
| 10 Copy; n (%) | 10,012 (6.5%) | 787 (4.6%) | 3,656 (2.8%) | 613 (2.5%) | 24,561 (6.4%) | 1,804 (6.2%) | 38,229 (5.7%) | 3,204 (4.5%) | 0.05 |
| Diabetic Foot; n (%) | 2,746 (1.8%) | 225 (1.3%) | 1,770 (1.3%) | 267 (1.1%) | 8,551 (2.2%) | 561 (1.9%) | 13,067 (1.9%) | 1,053 (1.5%) | 0.03 |
| Gangrene ; n (%) | 196 (0.1%) | 21 (0.1%) | 140 (0.1%) | 5 (0.0%) | 528 (0.1%) | 19 (0.1%) | 864 (0.1%) | 45 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 771 (0.5%) | 46 (0.3%) | 205 (0.2%) | 24 (0.1%) | 1,708 (0.4%) | 84 (0.3%) | 2,684 (0.4%) | 154 (0.2%) | 0.04 |
| Osteomyelitis; n (%) | 575 (0.4%) | 43 (0.3%) | 368 (0.3%) | 45 (0.2%) | 1,347 (0.3%) | 74 (0.3%) | 2,290 (0.3%) | 162 (0.2%) | 0.02 |
| Skin infections; n (%) | 7,163 (4.6%) | 798 (4.7%) | 5,853 (4.4%) | 994 (4.1%) | 21,559 (5.6%) | 1,617 (5.6%) | 34,575 (5.1%) | 3,409 (4.8%) | 0.01 |
| Erectile dysfunction; n (%) | 4,013 (2.6%) | 591 (3.4%) | 3,090 (2.3%) | 691 (2.8%) | 7,642 (2.0%) | 868 (3.0%) | 14,745 (2.2%) | 2,150 (3.1%) | -0.06 |
| Diabetes with unspecified complication; n (%) | 7,328 (4.7%) | 839 (4.9%) | 4,931 (3.7%) | 1,046 (4.3%) | 16,772 (4.4%) | 1,530 (5.3%) | 29,031 (4.3%) | 3,415 (4.8%) | -0.02 |
| Diabetes mellitus without mention of complications; n<br>(%) | 131,414 (84.8%) | 14,605 (85.1%) | 120,351 (91.1%) | 22,432 (92.2%) | 355,860 (92.3%) | 26,575 (91.7%) | 607,625 (90.4%) | 63,612 (90.3%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims within | 131,414 (04.070) | 14,003 (83.178) | 120,331 (31.176) | 22,432 (32.270) | 333,800 (32.3%) | 20,373 (31.7%) | 007,023 (30.478) | 03,012 (30.370) | 0.00 |
| 365 days; n (%) | 140,329 (90.6%) | 15,738 (91.7%) | 111,054 (84.1%) | 21,293 (87.6%) | 364,169 (94.5%) | 27,766 (95.8%) | 615,552 (91.6%) | 64,797 (92.0%) | -0.01 |
| Hyperlipidemia; n (%) | 111,115 (71.7%) | 13,329 (77.7%) | 89,589 (67.8%) | 18,477 (76.0%) | 293,228 (76.1%) | 23,958 (82.7%) | 493,932 (73.5%) | 55,764 (79.1%) | -0.13 |
| Edema; n (%) | 8,922 (5.8%) | 767 (4.5%) | 4,785 (3.6%) | 772 (3.2%) | 31,716 (8.2%) | 2,111 (7.3%) | 45,423 (6.8%) | 3,650 (5.2%) | 0.07 |
| Renal Dysfunction (non-diabetic); n (%) | 31,030 (20.0%) | 1,617 (9.4%) | 13,265 (10.0%) | 1,233 (5.1%) | 75,670 (19.6%) | 3,535 (12.2%) | 119,965 (17.8%) | 6,385 (9.1%) | 0.26 |
| Occurrence of acute renal disease ; n (%) | 3,885 (2.5%) | 136 (0.8%) | 1,944 (1.5%) | 95 (0.4%) | 10,543 (2.7%) | 322 (1.1%) | 16,372 (2.4%) | 553 (0.8%) | 0.13 |
| Occurrence of chronic renal insufficiency; n (%) | 26,302 (17.0%) | 1,333 (7.8%) | 9,757 (7.4%) | 892 (3.7%) | 63,348 (16.4%) | 2,891 (10.0%) | 99,407 (14.8%) | 5,116 (7.3%) | 0.24 |
| Chronic kidney disease ; n (%) | 25,400 (16.4%) | 1,244 (7.3%) | 9,238 (7.0%) | 765 (3.1%) | 60,327 (15.7%) | 2,654 (9.2%) | 94,965 (14.1%) | 4,663 (6.6%) | 0.25 |
| CKD Stage 3-4; n (%) | 17,724 (11.4%) | 638 (3.7%) | 6,019 (4.6%) | 375 (1.5%) | 42,095 (10.9%) | 1,536 (5.3%) | 65,838 (9.8%) | 2,549 (3.6%) | 0.25 |
| Occurrence of hypertensive nephropathy; n (%) | 11,901 (7.7%) | 539 (3.1%) | 4,074 (3.1%) | 305 (1.3%) | 25,957 (6.7%) | 1,009 (3.5%) | 41,932 (6.2%) | 1,853 (2.6%) | 0.18 |
| Occurrence of miscellaneous renal insufficiency ; n (%) | 6,270 (4.0%) | 315 (1.8%) | 3,464 (2.6%) | 373 (1.5%) | 20,943 (5.4%) | 1,032 (3.6%) | 30,677 (4.6%) | 1,720 (2.4%) | 0.12 |
| Glaucoma or cataracts ; n (%) | 29,202 (18.9%) | 2,865 (16.7%) | 18,976 (14.4%) | 3,293 (13.5%) | 96,718 (25.1%) | 7,893 (27.2%) | 144,896 (21.6%) | 14,051 (19.9%) | 0.04 |
| Cellulitis or abscess of toe; n (%) | 1,798 (1.2%) | 152 (0.9%) | 980 (0.7%) | 137 (0.6%) | 4,579 (1.2%) | 308 (1.1%) | 7,357 (1.1%) | 597 (0.8%) | 0.03 |
| Foot ulcer; n (%) | 2,634 (1.7%) | 213 (1.2%) | 1,736 (1.3%) | 264 (1.1%) | 8,482 (2.2%) | 558 (1.9%) | 12,852 (1.9%) | 1,035 (1.5%) | 0.03 |
| Bladder stones; n (%) | 170 (0.1%) | 13 (0.1%) | 132 (0.1%) | 16 (0.1%) | 548 (0.1%) | 37 (0.1%) | 850 (0.1%) | 66 (0.1%) | 0.00<br>0.01 |
| Kidney stones; n (%) Urinary tract infections (UTIs); n (%) | 2,807 (1.8%)<br>11,361 (7.3%) | 261 (1.5%)<br>883 (5.1%) | 2,375 (1.8%)<br>6,545 (5.0%) | 433 (1.8%)<br>963 (4.0%) | 8,275 (2.1%)<br>41,611 (10.8%) | 659 (2.3%)<br>2,560 (8.8%) | 13,457 (2.0%)<br>59,517 (8.9%) | 1,353 (1.9%)<br>4,406 (6.3%) | 0.01 |
| Dipstick urinalysis; n (%) | 49,794 (32.1%) | 5,364 (31.3%) | 37,552 (28.4%) | 7,447 (30.6%) | 135,533 (35.2%) | 10,690 (36.9%) | 222,879 (33.1%) | 23,501 (33.4%) | -0.01 |
| Non-dipstick urinalysis; n (%) | 64,593 (41.7%) | 7,874 (45.9%) | 44,790 (33.9%) | 10,311 (42.4%) | 151,194 (39.2%) | 13,426 (46.3%) | 260,577 (38.8%) | 31,611 (44.9%) | -0.12 |
| Urine function test; n (%) | 2,926 (1.9%) | 230 (1.3%) | 2,192 (1.7%) | 317 (1.3%) | 10,601 (2.8%) | 809 (2.8%) | 15,719 (2.3%) | 1,356 (1.9%) | 0.03 |
| Cytology; n (%) | 733 (0.5%) | 74 (0.4%) | 752 (0.6%) | 124 (0.5%) | 2,588 (0.7%) | 202 (0.7%) | 4,073 (0.6%) | 400 (0.6%) | 0.00 |
| Cystoscopy; n (%) | 1,397 (0.9%) | 110 (0.6%) | 1,137 (0.9%) | 161 (0.7%) | 4,335 (1.1%) | 295 (1.0%) | 6,869 (1.0%) | 566 (0.8%) | 0.02 |
| Other Covariates | ,, | , | , . ( , | . ( , | ,, | , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Osteoarthritis; n (%) | 18,548 (12.0%) | 1,772 (10.3%) | 10,553 (8.0%) | 1,694 (7.0%) | 64,696 (16.8%) | 4,889 (16.9%) | 93,797 (14.0%) | 8,355 (11.9%) | 0.06 |
| Other arthritis, arthropathies and musculoskeletal pain; n | | | | | | | | | |
| (%) | 43,333 (28.0%) | 4,698 (27.4%) | 31,686 (24.0%) | 5,758 (23.7%) | 134,642 (34.9%) | 10,271 (35.4%) | 209,661 (31.2%) | 20,727 (29.4%) | 0.04 |
| Dorsopathies; n (%) | 27,300 (17.6%) | 3,034 (17.7%) | 19,269 (14.6%) | 3,723 (15.3%) | 80,976 (21.0%) | 6,590 (22.7%) | 127,545 (19.0%) | 13,347 (18.9%) | 0.00 |
| Fractures; n (%) | 3,317 (2.1%) | 299 (1.7%) | 2,317 (1.8%) | 355 (1.5%) | 11,160 (2.9%) | 681 (2.3%) | 16,794 (2.5%) | 1,335 (1.9%) | 0.04 |
| Falls; n (%) | 4,393 (2.8%) | 292 (1.7%) | 1,273 (1.0%) | 126 (0.5%) | 13,534 (3.5%) | 651 (2.2%) | 19,200 (2.9%) | 1,069 (1.5%) | 0.10 |
| Osteoporosis; n (%) | 6,177 (4.0%) | 446 (2.6%) | 2,182 (1.7%) | 323 (1.3%) | 23,320 (6.1%) | 1,802 (6.2%) | 31,679 (4.7%) | 2,571 (3.6%) | 0.06<br>0.01 |
| Hyperthyroidism; n (%) | 881 (0.6%) | 92 (0.5%) | 541 (0.4%) | 104 (0.4%) | 2,984 (0.8%) | 244 (0.8%) | 4,406 (0.7%) | 440 (0.6%) | -0.03 |
| Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) | 21,624 (14.0%)<br>4,419 (2.9%) | 2,517 (14.7%)<br>666 (3.9%) | 13,319 (10.1%)<br>3,264 (2.5%) | 2,893 (11.9%)<br>897 (3.7%) | 44,004 (11.4%)<br>12,341 (3.2%) | 3,638 (12.6%)<br>1,310 (4.5%) | 78,947 (11.7%)<br>20,024 (3.0%) | 9,048 (12.8%)<br>2,873 (4.1%) | -0.03 |
| Depression; n (%) | 10,169 (6.6%) | 1,264 (7.4%) | 7,134 (5.4%) | 1,503 (6.2%) | 32,440 (8.4%) | 2,562 (8.8%) | 49,743 (7.4%) | 5,329 (7.6%) | -0.06 |
| Anxiety; n (%) | 9,789 (6.3%) | 1,176 (6.9%) | 5,860 (4.4%) | 1,146 (4.7%) | 26,959 (7.0%) | 2,045 (7.1%) | 42,608 (6.3%) | 4,367 (6.2%) | 0.00 |
| Sleep_Disorder; n (%) | 7,808 (5.0%) | 1,334 (7.8%) | 9,758 (7.4%) | 2,822 (11.6%) | 24,586 (6.4%) | 2,463 (8.5%) | 42,152 (6.3%) | 6,619 (9.4%) | -0.12 |
| Dementia; n (%) | 4,899 (3.2%) | 163 (1.0%) | 2,106 (1.6%) | 124 (0.5%) | 23,566 (6.1%) | 942 (3.2%) | 30,571 (4.5%) | 1,229 (1.7%) | 0.16 |
| Delirium; n (%) | 1,146 (0.7%) | 47 (0.3%) | 567 (0.4%) | 36 (0.1%) | 4,774 (1.2%) | 187 (0.6%) | 6,487 (1.0%) | 270 (0.4%) | 0.07 |
| Psychosis; n (%) | 1,233 (0.8%) | 77 (0.4%) | 619 (0.5%) | 46 (0.2%) | 5,761 (1.5%) | 258 (0.9%) | 7,613 (1.1%) | 381 (0.5%) | 0.07 |
| Obesity; n (%) | 29,896 (19.3%) | 4,631 (27.0%) | 18,364 (13.9%) | 4,643 (19.1%) | 48,909 (12.7%) | 5,747 (19.8%) | 97,169 (14.5%) | 15,021 (21.3%) | -0.18 |
| Overweight; n (%) | 8,442 (5.5%) | 854 (5.0%) | 2,983 (2.3%) | 553 (2.3%) | 12,502 (3.2%) | 1,070 (3.7%) | 23,927 (3.6%) | 2,477 (3.5%) | 0.01 |
| Smoking; n (%) | 14,958 (9.7%) | 1,412 (8.2%) | 7,989 (6.1%) | 1,213 (5.0%) | 44,623 (11.6%) | 3,182 (11.0%) | 67,570 (10.0%) | 5,807 (8.2%) | 0.06 |
| Alcohol abuse or dependence; n (%) | 56 (0.0%) | 0 (0.0%) | 37 (0.0%) | 6 (0.0%) | ** | ** | ** | ** | ** |
| Drug abuse or dependence; n (%) | 63 (0.0%) | 7 (0.0%) | 25 (0.0%) | 4 (0.0%) | ** | ** | ** | ** | ** |
| COPD; n (%) | 11,438 (7.4%) | 842 (4.9%) | 5,445 (4.1%) | 667 (2.7%) | 35,836 (9.3%) | 2,375 (8.2%) | 52,719 (7.8%) | 3,884 (5.5%) | 0.09 |

| Asthma; n (%) | 6,705 (4.3%) | 826 (4.8%) | 4,598 (3.5%) | 883 (3.6%) | 18,875 (4.9%) | 1,554 (5.4%) | 30,178 (4.5%) | 3,263 (4.6%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 12,320 (8.0%) | 2,043 (11.9%) | 11,112 (8.4%) | 3,033 (12.5%) | 23,357 (6.1%) | 2,710 (9.3%) | 46,789 (7.0%) | 7,786 (11.1%) | -0.14 |
| Pneumonia; n (%) | 2,800 (1.8%) | 193 (1.1%) | 1,979 (1.5%) | 213 (0.9%) | 9,582 (2.5%) | 478 (1.6%) | 14,361 (2.1%) | 884 (1.3%) | 0.06 |
| Imaging; n (%) | 70 (0.0%) | 3 (0.0%) | 34 (0.0%) | 3 (0.0%) | 173 (0.0%) | 12 (0.0%) | 277 (0.0%) | 18 (0.0%) | #DIV/0! |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 589 (0.4%) | 64 (0.4%) | 395 (0.3%) | 78 (0.3%) | 1,594 (0.4%) | 198 (0.7%) | 2,578 (0.4%) | 340 (0.5%) | -0.01 |
| DM Medications - Glitazones; n (%) | 10,422 (6.7%) | 1,544 (9.0%) | 8,718 (6.6%) | 2,208 (9.1%) | 24,517 (6.4%) | 2,742 (9.5%) | 43,657 (6.5%) | 6,494 (9.2%) | -0.10 |
| | 19,589 (12.6%) | 5,087 (29.7%) | 15,413 (11.7%) | 7,310 (30.1%) | 53,691 (13.9%) | 10,058 (34.7%) | 88,693 (13.2%) | 22,455 (31.9%) | -0.16 |
| DM Medications - Insulin; n (%) | | | | | | | | | |
| DM Medications - Meglitinides; n (%) | 924 (0.6%) | 247 (1.4%) | 1,054 (0.8%) | 491 (2.0%) | 3,952 (1.0%) | 817 (2.8%) | 5,930 (0.9%) | 1,555 (2.2%) | -0.11 |
| DM Medications - Metformin; n (%) | 108,309 (69.9%) | 13,385 (78.0%) | 96,831 (73.3%) | 19,082 (78.5%) | 254,527 (66.0%) | 21,505 (74.2%) | 459,667 (68.4%) | 53,972 (76.6%) | -0.18 |
| Concomitant initiation or current use of DPP4i Copy; n | | | | | | | | | |
| (%) | 17,486 (11.3%) | 3,345 (19.5%) | 21,174 (16.0%) | 5,938 (24.4%) | 51,735 (13.4%) | 7,439 (25.7%) | 90,395 (13.4%) | 16,722 (23.7%) | -0.27 |
| Concomitant initiation or current use of AGIs; n (%) | 425 (0.3%) | 45 (0.3%) | 286 (0.2%) | 39 (0.2%) | 1,174 (0.3%) | 139 (0.5%) | 1,885 (0.3%) | 223 (0.3%) | 0.00 |
| Concomitant initiation or current use of Glitazones; n (%) | 8,576 (5.5%) | 1,175 (6.8%) | 7,176 (5.4%) | 1,639 (6.7%) | 20,067 (5.2%) | 2,075 (7.2%) | 35,819 (5.3%) | 4,889 (6.9%) | -0.07 |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 4,299 (2.8%) | 2,107 (12.3%) | 4,901 (3.7%) | 3,223 (13.3%) | 7,426 (1.9%) | 2,835 (9.8%) | 16,626 (2.5%) | 8,165 (11.6%) | -0.36 |
| Concomitant initiation or current use of Insulin; n (%) | 13,776 (8.9%) | 3,869 (22.6%) | 11,356 (8.6%) | 5,709 (23.5%) | 39,091 (10.1%) | 8,072 (27.8%) | 64,223 (9.6%) | 17,650 (25.1%) | -0.42 |
| Concomitant initiation or current use of Meglitinides; n | , , , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | ., ( , | , , | .,. , | , , , , | ,, | |
| (%) | 613 (0.4%) | 171 (1.0%) | 711 (0.5%) | 321 (1.3%) | 2,576 (0.7%) | 581 (2.0%) | 3,900 (0.6%) | 1,073 (1.5%) | -0.09 |
| (70) | 015 (0.175) | 171 (1.070) | 711 (0.570) | 521 (1.570) | 2,570 (0.770) | 301 (2.070) | 3,300 (0.070) | 1,075 (1.570) | 0.03 |
| Concomitant initiation or current use of Metformin; n (%) | 92,596 (59.8%) | 11,270 (65.7%) | 83,076 (62.9%) | 16,009 (65.8%) | 217,493 (56.4%) | 18,170 (62.7%) | 393,165 (58.5%) | 45,449 (64.5%) | -0.12 |
| Past use of DPP4i Copy; n (%) | 6,565 (4.2%) | 1,159 (6.8%) | 5,963 (4.5%) | 1,809 (7.4%) | 17,310 (4.5%) | 2,138 (7.4%) | 29,838 (4.4%) | 5,106 (7.2%) | -0.12 |
| Past use of AGIs Copy; n (%) | 164 (0.1%) | 19 (0.1%) | 109 (0.1%) | 39 (0.2%) | 420 (0.1%) | 59 (0.2%) | 693 (0.1%) | 117 (0.2%) | -0.03 |
| Past use of Glitazones Copy; n (%) | 1,846 (1.2%) | 369 (2.2%) | 1,543 (1.2%) | 569 (2.3%) | 4,450 (1.2%) | 667 (2.3%) | 7,839 (1.2%) | 1,605 (2.3%) | -0.08 |
| Past use of GLP-1 RA Copy; n (%) | 2,375 (1.5%) | 888 (5.2%) | 2,076 (1.6%) | 1,436 (5.9%) | 4,256 (1.1%) | 1,234 (4.3%) | 8,707 (1.3%) | 3,558 (5.0%) | -0.21 |
| Past use of Insulin Copy; n (%) | 5,813 (3.8%) | 1,218 (7.1%) | 4,057 (3.1%) | 1,601 (6.6%) | 14,604 (3.8%) | 1,987 (6.9%) | 24,474 (3.6%) | 4,806 (6.8%) | -0.14 |
| Past use of Meglitinides Copy; n (%) | 311 (0.2%) | 76 (0.4%) | 343 (0.3%) | 170 (0.7%) | 1,376 (0.4%) | 236 (0.8%) | 2,030 (0.3%) | 482 (0.7%) | -0.06 |
| Past use of metformin (final) Copy; n (%) | 15,713 (10.1%) | 2,115 (12.3%) | 13,756 (10.4%) | 3,073 (12.6%) | 37,034 (9.6%) | 3,335 (11.5%) | 66,503 (9.9%) | 8,523 (12.1%) | -0.07 |
| Other Medications | , , , , | , - ( , | -, ( , | -,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | -/ ( | |
| Use of ACE inhibitors; n (%) | 84,706 (54.7%) | 8,925 (52.0%) | 72,224 (54.7%) | 12,297 (50.6%) | 197,008 (51.1%) | 13,650 (47.1%) | 353,938 (52.6%) | 34,872 (49.5%) | 0.06 |
| Use of ARBs; n (%) | 47,885 (30.9%) | 6,552 (38.2%) | 42,148 (31.9%) | 9,717 (40.0%) | 119,221 (30.9%) | 11,500 (39.7%) | 209,254 (31.1%) | 27,769 (39.4%) | -0.17 |
| * * * | | | | | | | | | |
| Use of Loop Diuretics ; n (%) | 19,348 (12.5%) | 1,498 (8.7%) | 12,373 (9.4%) | 1,847 (7.6%) | 68,480 (17.8%) | 4,431 (15.3%) | 100,201 (14.9%) | 7,776 (11.0%) | 0.12 |
| Use of other diuretics; n (%) | 4,344 (2.8%) | 466 (2.7%) | 3,400 (2.6%) | 615 (2.5%) | 13,410 (3.5%) | 985 (3.4%) | 21,154 (3.1%) | 2,066 (2.9%) | 0.01 |
| Use of nitrates-United; n (%) | 7,132 (4.6%) | 547 (3.2%) | 4,935 (3.7%) | 735 (3.0%) | 27,238 (7.1%) | 1,788 (6.2%) | 39,305 (5.8%) | 3,070 (4.4%) | 0.06 |
| Use of other hypertension drugs; n (%) | 11,822 (7.6%) | 853 (5.0%) | 8,348 (6.3%) | 1,083 (4.5%) | 34,116 (8.9%) | 2,082 (7.2%) | 54,286 (8.1%) | 4,018 (5.7%) | 0.09 |
| Use of digoxin; n (%) | 2,388 (1.5%) | 178 (1.0%) | 1,809 (1.4%) | 225 (0.9%) | 11,438 (3.0%) | 609 (2.1%) | 15,635 (2.3%) | 1,012 (1.4%) | 0.07 |
| Use of Anti-arrhythmics; n (%) | 1,811 (1.2%) | 148 (0.9%) | 1,428 (1.1%) | 195 (0.8%) | 7,241 (1.9%) | 442 (1.5%) | 10,480 (1.6%) | 785 (1.1%) | 0.04 |
| Use of COPD/asthma meds; n (%) | 18,661 (12.0%) | 2,398 (14.0%) | 16,481 (12.5%) | 3,563 (14.7%) | 54,930 (14.3%) | 5,018 (17.3%) | 90,072 (13.4%) | 10,979 (15.6%) | -0.06 |
| Use of statins; n (%) | 106,155 (68.5%) | 12,492 (72.8%) | 85,402 (64.7%) | 17,004 (69.9%) | 267,482 (69.4%) | 22,004 (75.9%) | 459,039 (68.3%) | 51,500 (73.1%) | -0.11 |
| Use of other lipid-lowering drugs; n (%) | 14,959 (9.7%) | 2,353 (13.7%) | 15,699 (11.9%) | 3,931 (16.2%) | 42,819 (11.1%) | 4,445 (15.3%) | 73,477 (10.9%) | 10,729 (15.2%) | -0.13 |
| Use of antiplatelet agents; n (%) | 16,208 (10.5%) | 1,683 (9.8%) | 13,697 (10.4%) | 2,526 (10.4%) | 50,943 (13.2%) | 4,302 (14.8%) | 80,848 (12.0%) | 8,511 (12.1%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | () | () | | |
| Apixaban, Warfarin); n (%) | 9,071 (5.9%) | 726 (4.2%) | 6,372 (4.8%) | 810 (3.3%) | 35,017 (9.1%) | 2,235 (7.7%) | 50,460 (7.5%) | 3,771 (5.4%) | 0.09 |
| Use of heparin and other low-molecular weight heparins; | | | | | | | | | |
| n (%) | 309 (0.2%) | 16 (0.1%) | 7 (0.0%) | 0 (0.0%) | 1,042 (0.3%) | 70 (0.2%) | 1,358 (0.2%) | 086 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 21,661 (14.0%) | 2,844 (16.6%) | 19,311 (14.6%) | 3,992 (16.4%) | 53,840 (14.0%) | 4,711 (16.3%) | 94,812 (14.1%) | 11,547 (16.4%) | -0.06 |
| Use of oral corticosteroids; n (%) | 18,506 (11.9%) | 2,069 (12.1%) | 15,049 (11.4%) | 2,725 (11.2%) | 53,287 (13.8%) | 4,148 (14.3%) | 86,842 (12.9%) | 8,942 (12.7%) | 0.01 |
| Use of bisphosphonate (United); n (%) | 3,267 (2.1%) | 202 (1.2%) | 1,232 (0.9%) | 166 (0.7%) | 10,720 (2.8%) | 820 (2.8%) | 15,219 (2.3%) | 1,188 (1.7%) | 0.04 |
| Use of opioids; n (%) | 28,673 (18.5%) | 3,296 (19.2%) | 25,050 (19.0%) | 4,773 (19.6%) | 77,313 (20.1%) | 5,898 (20.3%) | 131,036 (19.5%) | 13,967 (19.8%) | -0.01 |
| Use of antidepressants; n (%) | 30,934 (20.0%) | 4,117 (24.0%) | 24,343 (18.4%) | 5,483 (22.5%) | 84,498 (21.9%) | 7,501 (25.9%) | 139,775 (20.8%) | 17,101 (24.3%) | -0.08 |
| Use of antipsychotics; n (%) | 2,865 (1.8%) | 313 (1.8%) | 1,708 (1.3%) | 306 (1.3%) | 10,029 (2.6%) | 710 (2.4%) | 14,602 (2.2%) | 1,329 (1.9%) | 0.02 |
| Use of anticonvulsants; n (%) | 20,628 (13.3%) | 2,395 (14.0%) | 12,316 (9.3%) | 2,631 (10.8%) | 53,496 (13.9%) | 4,560 (15.7%) | 86,440 (12.9%) | 9,586 (13.6%) | -0.02 |
| Use of lithium; n (%) | 183 (0.1%) | 23 (0.1%) | 171 (0.1%) | 13 (0.1%) | 395 (0.1%) | 27 (0.1%) | 749 (0.1%) | 063 (0.1%) | 0.00 |
| Use of Benzos; n (%) | 12,618 (8.1%) | 1,545 (9.0%) | 10,457 (7.9%) | 2,066 (8.5%) | 37,940 (9.8%) | 2,876 (9.9%) | 61,015 (9.1%) | 6,487 (9.2%) | 0.00 |
| Use of anxiolytics/hypnotics; n (%) | 6,385 (4.1%) | 938 (5.5%) | 6,064 (4.6%) | 1,394 (5.7%) | 17,827 (4.6%) | 1,653 (5.7%) | 30,276 (4.5%) | 3,985 (5.7%) | -0.05 |
| Use of dementia meds; n (%) | 3,210 (2.1%) | 113 (0.7%) | 1,591 (1.2%) | 88 (0.4%) | 15,947 (4.1%) | 791 (2.7%) | 20,748 (3.1%) | 992 (1.4%) | 0.11 |
| Use of antiparkinsonian meds; n (%) | 2,966 (1.9%) | 338 (2.0%) | 1,934 (1.5%) | 385 (1.6%) | 10,222 (2.7%) | 859 (3.0%) | 15,122 (2.2%) | 1,582 (2.2%) | 0.00 |
| Any use of pramlintide; n (%) | 3 (0.0%) | 28 (0.2%) | 22 (0.0%) | 43 (0.2%) | 22 (0.0%) | 35 (0.1%) | 047 (0.0%) | 106 (0.2%) | -0.06 |
| Any use of 1st generation sulfonylureas; n (%) | 18 (0.0%) | 2 (0.0%) | 57 (0.0%) | 1 (0.0%) | ** | ** | ** | ** | ** |
| Entresto (sacubitril/valsartan); n (%) | 182 (0.1%) | 8 (0.0%) | 45 (0.0%) | 6 (0.0%) | ** | ** | ** | ** | ** |
| Initiation as monotherapy Copy; n (%) | 16,688 (10.8%) | 1,198 (7.0%) | 12,296 (9.3%) | 1,306 (5.4%) | 39,187 (10.2%) | 1,233 (4.3%) | 68,171 (10.1%) | 3,737 (5.3%) | 0.18 |
| Labs | , | , | . , , | | | | 286,926 | 41,472 | |
| Lab values- HbA1c (%) ; n (%) | 60,079 (38.8%) | 7,406 (43.2%) | 8,994 (6.8%) | 1,531 (6.3%) | N/A | N/A | 69,073 (24.1%) | 8,937 (21.5%) | 0.06 |
| Lab values-HbA1c (%) (within 3 months); n (%) | 46,986 (30.3%) | 6,068 (35.4%) | 7,101 (5.4%) | 1,306 (5.4%) | N/A | N/A | 54,087 (18.9%) | 7,374 (17.8%) | 0.03 |
| Lab values- HbA1c (%) (within 3 months); n (%) Lab values- HbA1c (%) (within 6 months); n (%) | 60,079 (38.8%) | 7,406 (43.2%) | 8,994 (6.8%) | 1,531 (6.3%) | N/A<br>N/A | N/A<br>N/A | 69,073 (24.1%) | 8,937 (21.5%) | 0.03 |
| Lab values- HDMLC (/0) (WILLIIII O HIUHLIS) , II (/0) | 00,073 (30.070) | 7,400 (43.2%) | 0,224 (0.0%) | 1,551 (0.5%) | N/A | IN/A | 03,013 (24.170) | 0,33/ (21.370) | 0.00 |

| Lab values- BNP; n (%) | 984 (0.6%) | 101 (0.6%) | 131 (0.1%) | 14 (0.1%) | N/A | N/A | 1,115 (0.4%) | 115 (0.3%) | 0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP (within 3 months); n (%) | 593 (0.4%) | 65 (0.4%) | 79 (0.1%) | 9 (0.0%) | N/A | N/A | 672 (0.2%) | 074 (0.2%) | 0.00 |
| Lab values- BNP (within 6 months); n (%) | 984 (0.6%) | 101 (0.6%) | 131 (0.1%) | 14 (0.1%) | N/A | N/A | 1,115 (0.4%) | 115 (0.3%) | 0.02 |
| Lab values- BUN (mg/dl); n (%) | 59,127 (38.2%) | 7,320 (42.7%) | 7,741 (5.9%) | 1,426 (5.9%) | N/A | N/A | 66,868 (23.3%) | 8,746 (21.1%) | 0.05 |
| | | | | | • | - | | | 0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 45,566 (29.4%) | 5,834 (34.0%) | 5,886 (4.5%) | 1,167 (4.8%) | N/A | N/A | 51,452 (17.9%) | 7,001 (16.9%) | |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 59,127 (38.2%) | 7,320 (42.7%) | 7,741 (5.9%) | 1,426 (5.9%) | N/A | N/A | 66,868 (23.3%) | 8,746 (21.1%) | 0.05 |
| Lab values- Creatinine (mg/dl); n (%) | 60,630 (39.1%) | 7,582 (44.2%) | 8,186 (6.2%) | 1,576 (6.5%) | N/A | N/A | 68,816 (24.0%) | 9,158 (22.1%) | 0.05 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 46,724 (30.2%) | 6,043 (35.2%) | 6,236 (4.7%) | 1,301 (5.3%) | N/A | N/A | 52,960 (18.5%) | 7,344 (17.7%) | 0.02 |
| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 60,630 (39.1%) | 7,582 (44.2%) | 8,186 (6.2%) | 1,576 (6.5%) | N/A | N/A | 68,816 (24.0%) | 9,158 (22.1%) | 0.05 |
| Lab values- HDL level (mg/dl); n (%) | 50,020 (32.3%) | 6,461 (37.7%) | 7,994 (6.1%) | 1,439 (5.9%) | N/A | N/A | 58,014 (20.2%) | 7,900 (19.0%) | 0.03 |
| (g/// (/ | , (, | 2,102 (011111) | ,,,,,, | _, (, | .,, | | // | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 36,675 (23.7%) | 4,910 (28.6%) | 5,881 (4.5%) | 1,126 (4.6%) | N/A | N/A | 42,556 (14.8%) | 6,036 (14.6%) | 0.01 |
| Lab values-TIDE level (Hig/GI) (WICHIII 3 HIGHCHS), II (76) | 30,073 (23.7%) | 4,510 (28.0%) | 3,881 (4.3%) | 1,120 (4.0%) | IN/A | IV/A | 42,330 (14.870) | 0,030 (14.0%) | 0.01 |
| 1.1 | 50,000 (00,00) | 6 464 (27 70) | 7.004 (6.40() | 4 420 (5 00() | 21/2 | | 50.044(20.20() | 7 000 (40 00() | 0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 50,020 (32.3%) | 6,461 (37.7%) | 7,994 (6.1%) | 1,439 (5.9%) | N/A | N/A | 58,014 (20.2%) | 7,900 (19.0%) | |
| Lab values- LDL level (mg/dl); n (%) | 51,820 (33.5%) | 6,667 (38.9%) | 8,382 (6.3%) | 1,463 (6.0%) | N/A | N/A | 60,202 (21.0%) | 8,130 (19.6%) | 0.03 |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 37,965 (24.5%) | 5,085 (29.6%) | 6,157 (4.7%) | 1,149 (4.7%) | N/A | N/A | 44,122 (15.4%) | 6,234 (15.0%) | 0.01 |
| Lab values-LDL level (mg/dl) (within 6 months); n (%) | 51,820 (33.5%) | 6,667 (38.9%) | 8,382 (6.3%) | 1,463 (6.0%) | N/A | N/A | 60,202 (21.0%) | 8,130 (19.6%) | 0.03 |
| Lab values- NT-proBNP; n (%) | 153 (0.1%) | 9 (0.1%) | 12 (0.0%) | 0 (0.0%) | N/A | N/A | 165 (0.1%) | 9 (0.0%) | 0.04 |
| Lab values- NT-proBNP (within 3 months); n (%) | 95 (0.1%) | 5 (0.0%) | 6 (0.0%) | 0 (0.0%) | N/A | N/A | 101 (0.0%) | 5 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | | | | | | | | | |
| | 153 (0.1%) | 9 (0.1%) | 12 (0.0%) | 0 (0.0%) | N/A | N/A | 165 (0.1%) | 9 (0.0%) | |
| Lab values-Total cholesterol (mg/dl); n (%) | 50,792 (32.8%) | 6,592 (38.4%) | 7,701 (5.8%) | 1,444 (5.9%) | N/A | N/A | 58,493 (20.4%) | 8,036 (19.4%) | 0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 37,250 (24.0%) | 5,024 (29.3%) | 5,639 (4.3%) | 1,134 (4.7%) | N/A | N/A | 42,889 (14.9%) | 6,158 (14.8%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 50,792 (32.8%) | 6,592 (38.4%) | 7,701 (5.8%) | 1,444 (5.9%) | N/A | N/A | 58,493 (20.4%) | 8,036 (19.4%) | 0.03 |
| Lab values-Triglyceride level (mg/dl); n (%) | 50,177 (32.4%) | 6,549 (38.2%) | 7,861 (6.0%) | 1,423 (5.9%) | N/A | N/A | 58,038 (20.2%) | 7,972 (19.2%) | 0.03 |
| Lab values- Triglyceride level (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 36,827 (23.8%) | 4,987 (29.1%) | 5,788 (4.4%) | 1,120 (4.6%) | N/A | N/A | 42,615 (14.9%) | 6,107 (14.7%) | 0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n | 30,027 (23.070) | 1,507 (25.270) | 3,700 (11.75) | 1,120 (110,0) | | , | 12,013 (111370) | 0,107 (11.770) | 0.01 |
| (%) | 50,177 (32.4%) | 6,549 (38.2%) | 7,861 (6.0%) | 1,423 (5.9%) | N/A | N/A | 58,038 (20.2%) | 7,972 (19.2%) | 0.03 |
| | 30,177 (32.4%) | 0,349 (38.2%) | 7,861 (6.0%) | 1,423 (5.9%) | N/A | IN/A | 30,030 (20.2%) | 7,972 (19.2%) | 0.03 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 59,675 | 7,362 | 8,091 | 1,482 | N/A | N/A | 67,766 | 8,844 | |
| mean (sd) | 8.19 (1.84) | 8.51 (1.76) | 8.39 (1.91) | 8.53 (1.75) | N/A | N/A | 8.21 (1.85) | 8.51 (1.76) | -0.17 |
| median [IQR] | 7.75 [6.93, 9.00] | 8.10 [7.25, 9.47] | 7.95 [7.00, 9.30] | 8.10 [7.30, 9.40] | N/A | N/A | 7.77 (1.85) | 8.10 (1.76) | -0.18 |
| Missing; n (%) | 95,211 (61.5%) | 9,792 (57.1%) | 123,949 (93.9%) | 22,836 (93.9%) | N/A | N/A | 219,160 (76.4%) | 32,628 (78.7%) | -0.06 |
| Lab result number- BNP mean | 984 | 101 | 131 | 14 | N/A | N/A | 1,115 | 115 | |
| mean (sd) | 184.36 (301.56) | 69.43 (79.37) | 262.73 (698.20) | 535.59 (1,297.93) | N/A | N/A | 193.57 (370.65) | 126.18 (448.51) | 0.16 |
| median [IQR] | 77.10 [29.92, 204.97] | 41.30 [18.65, 86.70] | 61.00 [30.00, 216.00] | 55.50 [16.65, 170.65] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 153,902 (99.4%) | 17,053 (99.4%) | 131,909 (99.9%) | 24,304 (99.9%) | N/A | N/A | 285,811 (99.6%) | 41,357 (99.7%) | -0.02 |
| | | | | | | | | | -0.02 |
| Lab result number- BUN (mg/dl) mean | 59,127 | 7,320 | 7,741 | 1,426 | N/A | N/A | 66,868 | 8,746 | |
| mean (sd) | 18.65 (8.00) | 16.63 (5.60) | 1,108.21 (12,786.12) | 2,280.99 (18,384.49) | N/A | N/A | 144.78 (4350.21) | 385.82 (7422.14) | -0.04 |
| median [IQR] | 17.00 [13.50, 22.00] | 16.00 [13.00, 19.00] | 16.00 [13.00, 20.00] | 16.00 [13.00, 19.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 95,759 (61.8%) | 9,834 (57.3%) | 124,299 (94.1%) | 22,892 (94.1%) | N/A | N/A | 220,058 (76.7%) | 32,726 (78.9%) | -0.05 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to | | | | | | | | | |
| 15 included) | 60,232 | 7,531 | 7,231 | 1,439 | N/A | N/A | 67,463 | 8,970 | |
| mean (sd) | 1.04 (0.40) | 0.92 (0.24) | 1.00 (0.36) | 0.93 (0.23) | N/A | N/A | 1.04 (0.40) | 0.92 (0.24) | 0.36 |
| median [IQR] | 0.95 [0.79, 1.18] | 0.89 [0.76, 1.04] | 0.95 [0.79, 1.10] | 0.90 [0.76, 1.05] | N/A | N/A | 0.95 (0.40) | 0.89 (0.24) | 0.18 |
| Missing; n (%) | 94,654 (61.1%) | | 124,809 (94.5%) | | | N/A | , , | , , | -0.05 |
| | 94,034 (01.1%) | 9,623 (56.1%) | 124,809 (94.5%) | 22,879 (94.1%) | N/A | IN/A | 219,463 (76.5%) | 32,502 (78.4%) | -0.05 |
| Lab result number- HDL level (mg/dl) mean (only =<5000 | | | | | | | | | |
| included) | 50,020 | 6,461 | 7,944 | 1,422 | N/A | N/A | 57,964 | 7,883 | |
| mean (sd) | 46.42 (13.62) | 45.25 (13.20) | 44.50 (14.95) | 46.24 (105.86) | N/A | N/A | 46.16 (13.81) | 45.43 (46.52) | 0.02 |
| median [IQR] | 44.50 [37.00, 54.00] | 43.00 [36.00, 52.00] | 43.00 [36.00, 52.00] | 42.50 [35.00, 50.06] | N/A | N/A | 44.29 (13.81) | 42.91 (46.52) | 0.04 |
| Missing; n (%) | 104,866 (67.7%) | 10,693 (62.3%) | 124,096 (94.0%) | 22,896 (94.2%) | N/A | N/A | 228,962 (79.8%) | 33,589 (81.0%) | -0.03 |
| Lab result number- LDL level (mg/dl) mean (only =<5000 | | | | | | | | | |
| included) | 50,646 | 6,539 | 7,492 | 1,290 | N/A | N/A | 58,138 | 7,829 | |
| mean (sd) | 87.95 (39.92) | 84.31 (39.29) | 90.16 (42.99) | 86.14 (40.59) | N/A | N/A | 88.23 (40.33) | 84.61 (39.51) | 0.09 |
| median [IQR] | 85.00 [64.00, 111.00] | 82.00 [61.00, 106.00] | 89.00 [66.00, 115.00] | 85.00 [62.50, 110.50] | N/A | N/A | 85.52 (40.33) | 82.49 (39.51) | 0.08 |
| Missing; n (%) | 104,240 (67.3%) | 10,615 (61.9%) | 124,548 (94.3%) | 23,028 (94.7%) | N/A | N/A | 228,788 (79.7%) | 33,643 (81.1%) | -0.04 |
| Lab result number-Total cholesterol (mg/dl) mean (only | | | _ | | | | | | |
| =<5000 included) | 50,753 | 6,586 | 7,649 | 1,425 | N/A | N/A | 58,402 | 8,011 | |
| mean (sd) | 174.22 (46.76) | 172.48 (46.71) | 175.10 (52.79) | 171.47 (55.16) | N/A | N/A | 174.34 (47.59) | 172.30 (48.32) | 0.04 |
| median [IQR] | 168.00 [143.00, 199.00] | 166.50 [142.00, 195.50] | | 169.00 [143.00, 196.00] | N/A | N/A | 168.52 (47.59) | 166.94 (48.32) | 0.03 |
| Missing; n (%) | 104,133 (67.2%) | 10,568 (61.6%) | 124,391 (94.2%) | 22,893 (94.1%) | N/A | N/A | 228,524 (79.6%) | 33,461 (80.7%) | -0.03 |

| Lab result number-Triglyceride level (mg/dl) mean (only | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| =<5000 included) | 50,170 | 6,548 | 7,808 | 1,404 | N/A | N/A | 57,978 | 7,952 | |
| mean (sd) | 184.72 (150.34) | 197.99 (180.75) | 187.17 (163.73) | 195.06 (186.08) | N/A | N/A | 185.05 (152.21) | 197.47 (181.71) | -0.07 |
| median [IQR] | 151.00 [108.00, 216.00] | 157.75 [112.00, 227.00] | 150.00 [105.00, 219.25] | 158.75 [111.00, 227.00] | N/A | N/A | 150.87 (152.21) | 157.93 (181.71) | -0.04 |
| Missing; n (%) | 104,716 (67.6%) | 10,606 (61.8%) | 124,232 (94.1%) | 22,914 (94.2%) | N/A | N/A | 228,948 (79.8%) | 33,520 (80.8%) | -0.03 |
| Lab result number- Hemoglobin mean (only >0 included) | 40,207 | 4,846 | 5,256 | 907 | N/A | N/A | 45,463 | 5,753 | |
| mean (sd) | 13.52 (1.64) | 14.06 (1.55) | 9,789.51 (284,520.72) | 13,220.12 (332,411.46) | N/A | N/A | 1143.73 (96735.42) | 2096.09 (131949.02) | -0.01 |
| median [IQR] | 13.55 [12.45, 14.60] | 14.10 [13.00, 15.10] | 13.70 [12.60, 14.80] | 13.95 [12.90, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 114,679 (74.0%) | 12,308 (71.8%) | 126,784 (96.0%) | 23,411 (96.3%) | N/A | N/A | 241,463 (84.2%) | 35,719 (86.1%) | -0.05 |
| Lab result number- Serum sodium mean (only > 90 and < | | | | | | | | | |
| 190 included) | 58,728 | 7,403 | 7,402 | 1,411 | N/A | N/A | 66,130 | 8,814 | |
| mean (sd) | 139.42 (2.80) | 139.27 (2.61) | 138.86 (2.72) | 139.05 (2.40) | N/A | N/A | 139.36 (2.79) | 139.23 (2.58) | 0.05 |
| median [IQR] | 139.67 [138.00, 141.00] | 139.00 [138.00, 141.00] | | 139.00 [138.00, 140.67] | N/A | N/A | 139.60 (2.79) | 139.00 (2.58) | 0.22 |
| Missing; n (%) | 96,158 (62.1%) | 9,751 (56.8%) | 124,638 (94.4%) | 22,907 (94.2%) | N/A | N/A | 220,796 (77.0%) | 32,658 (78.7%) | -0.04 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 54,335 | 6,987 | 6,383 | 1,182 | N/A | N/A | 60,718 | 8,169 | |
| mean (sd) | 4.26 (0.31) | 4.31 (0.30) | 4.10 (0.73) | 4.17 (0.69) | N/A | N/A | 4.24 (0.38) | 4.29 (0.38) | -0.13 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 4.20 [4.00, 4.40] | 4.30 [4.00, 4.50] | N/A | N/A | 4.29 (0.38) | 4.30 (0.38) | -0.03 |
| Missing; n (%) | 100,551 (64.9%) | 10,167 (59.3%) | 125,657 (95.2%) | 23,136 (95.1%) | N/A | N/A | 226,208 (78.8%) | 33,303 (80.3%) | -0.04 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | |
| (only 10-1000 included) | 58,552 | 7,391 | 7,387 | 1,393 | N/A | N/A | 65,939 | 8,784 | |
| mean (sd) | 174.40 (73.35) | 178.35 (69.83) | 182.10 (77.32) | 175.89 (63.14) | N/A | N/A | 175.26 (73.81) | 177.96 (68.82) | -0.04 |
| median [IQR] | 156.00 [126.00, 203.00] | 162.00 [130.00, 211.00] | 162.00 [130.00, 215.00] | 163.00 [131.50, 208.00] | N/A | N/A | 156.67 (73.81) | 162.16 (68.82) | -0.08 |
| Missing; n (%) | 96,334 (62.2%) | 9,763 (56.9%) | 124,653 (94.4%) | 22,925 (94.3%) | N/A | N/A | 220,987 (77.0%) | 32,688 (78.8%) | -0.04 |
| Laboration and Debaggious areas (auto 4.7 included) | co 2co | 7.544 | 7.444 | 1 271 | N/A | N/A | 67.712 | 8,912 | |
| Lab result number- Potassium mean (only 1-7 included) | 60,268 | 7,541<br>4.44 (0.40) | 7,444 | 1,371 | N/A<br>N/A | N/A<br>N/A | 4.44 (0.44) | 4.43 (0.40) | 0.02 |
| mean (sd) | 4.46 (0.44)<br>4.45 [4.20, 4.70] | 4.40 [4.20, 4.70] | 4.32 (0.46)<br>4.30 [4.00, 4.60] | 4.36 (0.41)<br>4.38 [4.10, 4.60] | N/A<br>N/A | N/A<br>N/A | 4.44 (0.44) | 4.43 (0.40) | 0.02 |
| median [IQR] | | | | | · | N/A<br>N/A | , , | , , | -0.05 |
| Missing; n (%) | 94,618 (61.1%) | 9,613 (56.0%) | 124,596 (94.4%) | 22,947 (94.4%) | N/A | N/A | 219,214 (76.4%) | 32,560 (78.5%) | -0.05 |
| Comorbidity Scores<br>CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.48 (1.68) | 2.06 (1.28) | 1.84 (1.27) | 1.65 (0.97) | 2.61 (1.79) | 2.37 (1.51) | 2.43 (1.67) | 2.05 (1.29) | 0.25 |
| | 2.00 [1.00, 3.00] | , , | | | , , | 2.00 [1.00, 3.00] | , , | , , | 0.23 |
| median [IQR] | 2.00 [1.00, 5.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 3.00] | 1.80 (1.67) | 1.65 (1.29) | 0.10 |
| Frailty Score: Qualitative Version 365 days as Categories, | | | | | | | | | |
| 0; n (%) | 97,586 (63.0%) | 11,069 (64.5%) | 71,771 (54.4%) | 12,999 (53.5%) | 159,513 (41.4%) | 13,058 (45.0%) | 328,870 (48.9%) | 37,126 (52.7%) | -0.08 |
| 1 to 2; n (%) | 42,109 (27.2%) | 4,734 (27.6%) | 45,704 (34.6%) | 9,121 (37.5%) | 136,252 (35.4%) | 10,120 (34.9%) | 224,065 (33.3%) | 23,975 (34.0%) | -0.01 |
| 3 or more; n (%) | 15,191 (9.8%) | 1,351 (7.9%) | 14,565 (11.0%) | 2,198 (9.0%) | 89,667 (23.3%) | 5,809 (20.0%) | 119,423 (17.8%) | 9,358 (13.3%) | 0.12 |
| 5 of more, ir (76) | 13,131 (3.0%) | 1,551 (7.570) | 14,505 (11.0%) | 2,130 (3.0%) | 05,007 (25.570) | 3,003 (20.070) | 113,423 (17.070) | 3,330 (13.370) | 0.12 |
| Frailty Score: Empirical Version 365 days as Categories, | | | | | | | | | |
| <0.12908; n (%) | 43,729 (28.2%) | 5,999 (35.0%) | 38,804 (29.4%) | 8,113 (33.4%) | 51,925 (13.5%) | 4,669 (16.1%) | 134,458 (20.0%) | 18,781 (26.7%) | -0.16 |
| 0.12908 - 0.1631167; n (%) | 55,491 (35.8%) | 6,402 (37.3%) | 50,669 (38.4%) | 9,645 (39.7%) | 111,334 (28.9%) | 8,922 (30.8%) | 217,494 (32.3%) | 24,969 (35.4%) | -0.07 |
| >= 0.1631167; n (%) | 55,666 (35.9%) | 4,753 (27.7%) | 42,567 (32.2%) | 6,560 (27.0%) | 222,173 (57.6%) | 15,396 (53.1%) | 320,406 (47.7%) | 26,709 (37.9%) | 0.20 |
| Non-Frailty; n (%) | 86,446 (55.8%) | 9,990 (58.2%) | 65,874 (49.9%) | 13,103 (53.9%) | 20,611 (5.3%) | 1,336 (4.6%) | 172,931 (25.7%) | 24,429 (34.7%) | -0.20 |
| Frailty Score (mean): Qualitative Version 365 days, | | | | | | | | | |
| mean (sd) | 0.78 (1.42) | 0.67 (1.20) | 0.91 (1.42) | 0.83 (1.20) | 1.53 (1.95) | 1.32 (1.69) | 1.24 (1.74) | 0.99 (1.42) | 0.16 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.57 (1.74) | 0.41 (1.42) | 0.10 |
| Frailty Score (mean): Empirical Version 365 days, | | | | | | | | | |
| mean (sd) | 0.16 (0.05) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.04) | 0.19 (0.06) | 0.18 (0.05) | 0.18 (0.05) | 0.16 (0.04) | 0.44 |
| median [IQR] | 0.15 [0.13, 0.18] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.16] | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.20] | 0.16 (0.05) | 0.15 (0.04) | 0.22 |
| Healthcare Utilization | | | | | | | | | |
| Any hospitalization; n (%) | 7,615 (4.9%) | 403 (2.3%) | 6,017 (4.6%) | 501 (2.1%) | 27,334 (7.1%) | 1,128 (3.9%) | 40,966 (6.1%) | 2,032 (2.9%) | 0.15 |
| Any hospitalization within prior 30 days; n (%) | 2,663 (1.7%) | 63 (0.4%) | 2,107 (1.6%) | 77 (0.3%) | 9,168 (2.4%) | 186 (0.6%) | 13,938 (2.1%) | 326 (0.5%) | 0.14 |
| Any hospitalization during prior 31-180 days; n (%) | 5,232 (3.4%) | 341 (2.0%) | 4,082 (3.1%) | 428 (1.8%) | 19,390 (5.0%) | 964 (3.3%) | 28,704 (4.3%) | 1,733 (2.5%) | 0.10 |
| Endocrinologist Visit; n (%) | 10,283 (6.6%) | 2,944 (17.2%) | 9,029 (6.8%) | 4,320 (17.8%) | 32,210 (8.4%) | 5,395 (18.6%) | 51,522 (7.7%) | 12,659 (18.0%) | -0.31 |
| Endocrinologist Visit (30 days prior); n (%) | 6,054 (3.9%) | 2,159 (12.6%) | 5,613 (4.3%) | 3,385 (13.9%) | 18,533 (4.8%) | 3,825 (13.2%) | 30,200 (4.5%) | 9,369 (13.3%) | -0.31 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 7,255 (4.7%) | 2,095 (12.2%) | 6,203 (4.7%) | 3,089 (12.7%) | 24,236 (6.3%) | 4,125 (14.2%) | 37,694 (5.6%) | 9,309 (13.2%) | -0.26 |
| Internal medicine/family medicine visits; n (%) | 129,232 (83.4%) | 12,121 (70.7%) | 113,946 (86.3%) | 21,262 (87.4%) | 316,729 (82.2%) | 23,915 (82.5%) | 559,907 (83.3%) | 57,298 (81.3%) | 0.05 |
| Internal medicine/family medicine visits (30 days prior); | | | | | | | | | |
| n (%) | 95,398 (61.6%) | 8,775 (51.2%) | 85,543 (64.8%) | 16,208 (66.7%) | 220,852 (57.3%) | 17,395 (60.0%) | 401,793 (59.8%) | 42,378 (60.1%) | -0.01 |
| Internal medicine/family medicine visits (31 to 180 days | | | | | | | | | |
| prior); n (%) | 107,756 (69.6%) | 10,414 (60.7%) | 89,803 (68.0%) | 17,894 (73.6%) | 266,263 (69.1%) | 21,172 (73.0%) | 463,822 (69.0%) | 49,480 (70.2%) | -0.03 |
| Cardiologist visit; n (%) | 35,417 (22.9%) | 3,293 (19.2%) | 21,785 (16.5%) | 4,133 (17.0%) | 114,927 (29.8%) | 8,307 (28.7%) | 172,129 (25.6%) | 15,733 (22.3%) | 0.08 |
| Number of Cardiologist visits (30 days prior); n (%) | 12,163 (7.9%) | 1,041 (6.1%) | 7,375 (5.6%) | 1,236 (5.1%) | 38,495 (10.0%) | 2,576 (8.9%) | 58,033 (8.6%) | 4,853 (6.9%) | 0.06 |

| Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) | 29,585 (19.1%)<br>39,699 (25.6%)<br>4,705 (3.0%)<br>0 (0.0%) | 2,777 (16.2%)<br>3,920 (22.9%)<br>608 (3.5%)<br>0 (0.0%) | 18,012 (13.6%)<br>32,047 (24.3%)<br>4,168 (3.2%)<br>0 (0.0%) | 3,495 (14.4%)<br>5,731 (23.6%)<br>1,037 (4.3%)<br>0 (0.0%) | 98,325 (25.5%)<br>114,568 (29.7%)<br>11,116 (2.9%)<br>0 (0.0%) | 7,192 (24.8%)<br>8,455 (29.2%)<br>960 (3.3%)<br>0 (0.0%) | 145,922 (21.7%)<br>186,314 (27.7%)<br>19,989 (3.0%)<br>000 (0.0%) | 13,464 (19.1%)<br>18,106 (25.7%)<br>2,605 (3.7%)<br>000 (0.0%) | 0.06<br>0.05<br>-0.04<br>#DIV/0! |
|---|---|---|---|---|---|---|---|---|---|
| Naive new user v8 Copy; n (%) N antidiabetic drugs at index date Copy | 33,568 (21.7%) | 1,869 (10.9%) | 27,156 (20.6%) | 2,032 (8.4%) | 74,547 (19.3%) | 1,975 (6.8%) | 135,271 (20.1%) | 5,876 (8.3%) | 0.34 |
| mean (sd) | 1.89 (0.73) | 2.29 (0.88) | 1.98 (0.76) | 2.35 (0.90) | 1.88 (0.74) | 2.36 (0.89) | 1.90 (0.74) | 2.34 (0.89) | -0.54 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [2.00, 3.00] | 2.00 [1.00, 2.00] | 2.00 [2.00, 3.00] | 2.00 [1.00, 2.00] | 2.00 [2.00, 3.00] | 2.00 (0.74) | 2.00 (0.89) | 0.00 |
| number of different/distinct medication prescriptions | | | | | | | | _ | |
| mean (sd)<br>median [IQR] | 9.15 (4.15)<br>8.00 [6.00, 11.00] | 10.03 (4.47)<br>9.00 [7.00, 12.00] | 8.64 (3.92)<br>8.00 [6.00, 11.00] | 9.85 (4.23)<br>9.00 [7.00, 12.00] | 9.16 (3.98)<br>9.00 [6.00, 11.00] 1 | 10.48 (4.44) | 9.06 (4.01)<br>8.57 (4.01) | 10.15 (4.38)<br>9.41 (4.38) | -0.26<br>-0.20 |
| Number of Hospitalizations | 8.00 [6.00, 11.00] | 9.00 [7.00, 12.00] | 8.00 [6.00, 11.00] | 9.00 [7.00, 12.00] | 9.00 [6.00, 11.00] | 10.00 [7.00, 13.00] | 8.37 (4.01) | 9.41 (4.56) | -0.20 |
| mean (sd) | 0.06 (0.27) | 0.03 (0.17) | 0.05 (0.24) | 0.02 (0.16) | 0.08 (0.34) | 0.04 (0.23) | 0.07 (0.31) | 0.03 (0.19) | 0.16 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.31) | 0.00 (0.19) | 0.00 |
| Number of hospital days<br>mean (sd) | 0.29 (2.03) | 0.11 (0.96) | 0.26 (1.78) | 0.10 (0.87) | 0.51 (3.04) | 0.23 (1.86) | 0.41 (2.62) | 0.16 (1.38) | 0.12 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 [0.00, 0.00] | 0.00 (2.62) | 0.00 (1.38) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.32 (0.96) | 0.21 (0.76) | 0.10 (0.93) | 0.04 (0.54) | 0.43 (1.16) | 0.31 (1.07) | 0.34 (1.07) | 0.19 (0.84) | 0.16 |
| median [IQR] Number of Office visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.07) | 0.00 (0.84) | 0.00 |
| mean (sd) | 3.95 (3.11) | 4.28 (3.09) | 3.80 (3.07) | 4.27 (3.11) | 4.45 (3.52) | 5.10 (3.63) | 4.21 (3.34) | 4.61 (3.33) | -0.12 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 6.00] | 4.00 [3.00, 7.00] | 3.57 (3.34) | 3.41 (3.33) | 0.05 |
| Number of Endocrinologist visits | 0.29 (1.68) | 0.94 (3.31) | 0.28 (1.62) | 0.98 (3.45) | 0.44 (2.45) | 1.25 (4.77) | 0.37 (2.15) | 1.08 (4.02) | -0.22 |
| mean (sd)<br>median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , , | 0.00 [0.00, 0.00] | 0.00 (2.15) | 0.00 (4.02) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | , | , | |
| mean (sd) | 8.28 (11.20) | 6.97 (10.95) | 5.99 (7.55) | 6.47 (7.65) | 6.87 (9.22) | 7.76 (10.04) | 7.02 (9.42) | 7.12 (9.53) | -0.01 |
| median [IQR] Number of Cardiologist visits | 5.00 [2.00, 11.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 8.00] | 4.00 [2.00, 9.00] | 4.00 [1.00, 9.00] | 5.00 [2.00, 10.00] | 4.23 (9.42) | 4.41 (9.53) | -0.02 |
| mean (sd) | 0.96 (2.84) | 0.76 (2.44) | 0.63 (2.23) | 0.63 (2.15) | 1.40 (3.79) | 1.35 (3.65) | 1.15 (3.33) | 0.96 (2.92) | 0.06 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , , | 0.00 [0.00, 1.00] | 0.00 (3.33) | 0.00 (2.92) | 0.00 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd)<br>median [IQR] | 0.45 (1.12)<br>0.00 [0.00, 1.00] | 0.35 (0.86)<br>0.00 [0.00, 0.00] | 0.40 (0.93)<br>0.00 [0.00, 0.00] | 0.35 (0.83)<br>0.00 [0.00, 0.00] | 0.55 (1.15) | 0.50 (1.07)<br>0.00 [0.00, 1.00] | 0.50 (1.10)<br>0.00 (1.10) | 0.41 (0.94)<br>0.00 (0.94) | 0.09<br>0.00 |
| Number of HbA1c tests ordered | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.10) | 0.00 (0.54) | 0.00 |
| mean (sd) | 1.20 (0.86) | 1.36 (0.88) | 1.00 (0.85) | 1.30 (0.86) | 1.30 (0.82) | 1.56 (0.82) | 1.22 (0.84) | 1.42 (0.85) | -0.24 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 (0.84) | 1.41 (0.85) | -0.49 |
| Number of glucose tests orderedmean (sd) | 0.39 (2.19) | 0.44 (1.71) | 0.32 (1.15) | 0.40 (1.03) | 0.34 (0.93) | 0.48 (1.14) | 0.35 (1.36) | 0.44 (1.27) | -0.07 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , , | 0.00 (1.36) | 0.00 (1.27) | 0.00 |
| Number of lipid tests ordered | | | | | | | | _ | |
| mean (sd) | 0.92 (0.89) | 1.07 (0.96) | 0.83 (1.13) | 1.07 (1.14) | 0.93 (0.78) | 1.13 (0.84) | 0.91 (0.88) | 1.09 (0.98) | -0.19<br>0.00 |
| median [IQR] Number of creatinine tests ordered | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 (0.88) | 1.00 (0.98) | 0.00 |
| mean (sd) | 0.04 (0.27) | 0.03 (0.21) | 0.06 (0.33) | 0.04 (0.23) | 0.07 (0.34) | 0.07 (0.32) | 0.06 (0.32) | 0.05 (0.27) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.32) | 0.00 (0.27) | 0.00 |
| Number of BUN tests orderedmean (sd) | 0.02 (0.20) | 0.02 (0.16) | 0.03 (0.23) | 0.02 (0.17) | 0.04 (0.28) | 0.04 (0.26) | 0.03 (0.25) | 0.03 (0.21) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.02 (0.16) | 0.00 [0.00, 0.00] | 0.02 (0.17) | , , | 0.00 [0.00, 0.00] | 0.03 (0.25) | 0.03 (0.21) | 0.00 |
| Number of tests for microal buminuria | | | | | | | , | , | |
| mean (sd) | 0.77 (1.14) | 0.85 (1.19) | 0.58 (0.99) | 0.76 (1.12) | 0.44 (0.67) | 0.54 (0.73) | 0.54 (0.87) | 0.69 (1.00) | -0.16 |
| median [IQR] Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level Copy | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.87) | 0.00 (1.00) | 0.00 |
| mean (sd) | 6.00 (6.67) | 5.41 (6.00) | 2.52 (4.05) | 2.02 (3.24) | 5.62 (7.42) | 5.82 (6.93) | 5.10 (6.71) | 4.41 (5.67) | 0.11 |
| median [IQR] | 5.00 [0.00, 9.00] | 5.00 [0.00, 8.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 3.44 (6.71) | 2.86 (5.67) | 0.09 |
| Use of thiazide; n (%) | 21,636 (14.0%) | 2,104 (12.3%) | 17,561 (13.3%) | 2,846 (11.7%) | 59,136 (15.3%) | 4,124 (14.2%) | 98,333 (14.6%) | 9,074 (12.9%) | 0.05 |
| Use of beta blockers; n (%) | 64,047 (41.4%) | 6,162 (35.9%) | 49,659 (37.6%) | 8,563 (35.2%) | 190,922 (49.5%) | 13,995 (48.3%) | 304,628 (45.3%) | 28,720 (40.8%) | 0.09 |
| Use of calcium channel blockers; n (%) | 51,925 (33.5%) | 4,913 (28.6%) | 41,303 (31.3%) | 6,991 (28.7%) | 139,264 (36.1%) | 9,858 (34.0%) | 232,492 (34.6%) | 21,762 (30.9%) | 0.08 |

| | Optu | ım | Market | Scan | Medio | care | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference- 2nd<br>Generation SUs | Eveneure Connellif:- | Reference- 2nd<br>Generation SUs | Evenouse Connelled!- | Reference- 2nd<br>Generation SUs | Evnoguro Conseliflo-i | Reference- 2nd<br>Generation SUs | Evnosuro Conadifloria | St. Dif |
| Number of patients | 16740 | Exposure-Canagliflozin<br>16740 | 23265 | Exposure-Canagliflozin<br>23265 | 28845 | Exposure-Canagliflozin<br>28845 | 68,850 | Exposure-Canagliflozin<br>68,850 | 3t. DIT |
| Age | 10740 | 10740 | 23203 | 23203 | 20043 | 20043 | 00,030 | 00,030 | |
| mean (sd) | 62.01 (8.13) | 62.11 (7.84) | 59.18 (6.78) | 59.28 (6.44) | 70.96 (5.29) | 71.04 (5.27) | 64.80 (6.58) | 64.89 (6.37) | -0.03 |
| median [IQR] | 61.00 [55.00, 68.00] | 61.00 [56.00, 68.00] | 58.00 [54.00, 63.00] | 59.00 [54.00, 63.00] | 70.00 [67.00, 74.00] | 70.00 [67.00, 74.00] | 63.76 (6.58) | 64.09 (6.37) | -0.05 |
| Age categories | 01.00 [55.00, 00.00] | 01.00 [50.00, 00.00] | 30.00 [34.00, 03.00] | 33.00 [34.00, 03.00] | 70.00 [07.00, 74.00] | 70.00 [07.00, 74.00] | 03.70 (0.30) | 04.03 (0.37) | 0.0. |
| 18 - 54; n (%) | 3,698 (22.1%) | 3,224 (19.3%) | 6,341 (27.3%) | 5,909 (25.4%) | 0 (0.0%) | 0 (0.0%) | 10,039 (14.6%) | 9,133 (13.3%) | 0.04 |
| 55 - 64; n (%) | 6,485 (38.7%) | 7,238 (43.2%) | 13,228 (56.9%) | 13,588 (58.4%) | 355 (1.2%) | 326 (1.1%) | 20,068 (29.1%) | 21,152 (30.7%) | -0.03 |
| 65 - 74; n (%) | 5,339 (31.9%) | 5,124 (30.6%) | 2,904 (12.5%) | 3,121 (13.4%) | 22,248 (77.1%) | 22,245 (77.1%) | 30,491 (44.3%) | 30,490 (44.3%) | 0.00 |
| >= 75; n (%) | 1,218 (7.3%) | 1,154 (6.9%) | 792 (3.4%) | 647 (2.8%) | 6,242 (21.6%) | 6,274 (21.8%) | 8,252 (12.0%) | 8,075 (11.7%) | 0.01 |
| Gender | | | | | | | | | |
| Males; n (%) | 9,326 (55.7%) | 9,329 (55.7%) | 12,867 (55.3%) | 12,977 (55.8%) | 14,338 (49.7%) | 14,294 (49.6%) | 36,531 (53.1%) | 36,600 (53.2%) | 0.00 |
| Females; n (%) | 7,414 (44.3%) | 7,411 (44.3%) | 10,398 (44.7%) | 10,288 (44.2%) | 14,507 (50.3%) | 14,551 (50.4%) | 32,319 (46.9%) | 32,250 (46.8%) | 0.00 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 23,182 (80.4%) | 23,167 (80.3%) | 23,182 (80.4%) | 23,167 (80.3%) | 0.00 |
| Black; n (%) | N/A | N/A | N/A | N/A | 2,305 (8.0%) | 2,349 (8.1%) | 2,305 (8.0%) | 2,349 (8.1%) | 0.00 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 1,028 (3.6%) | 1,033 (3.6%) | 1,028 (3.6%) | 1,033 (3.6%) | 0.00 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 989 (3.4%) | 979 (3.4%) | 989 (3.4%) | 979 (3.4%) | 0.00 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 117 (0.4%) | 116 (0.4%) | 117 (0.4%) | 116 (0.4%) | 0.00 |
| Other/Unknown; n (%) Region (lumping missing&other category with West) | N/A | N/A | N/A | N/A | 1,224 (4.2%) | 1,201 (4.2%) | 1,224 (4.2%) | 1,201 (4.2%) | 0.00 |
| Northeast; n (%) | 1,493 (8.9%) | 1,442 (8.6%) | 4,400 (18.9%) | 4,366 (18.8%) | 5,438 (18.9%) | 5,436 (18.8%) | 11,331 (16.5%) | 11,244 (16.3%) | 0.01 |
| South; n (%) | 8,914 (53.2%) | 8,950 (53.5%) | 4,094 (17.6%) | 4,131 (17.8%) | 12,680 (44.0%) | 12,557 (43.5%) | 25,688 (37.3%) | 25,638 (37.2%) | 0.00 |
| Midwest; n (%) | 3,472 (20.7%) | 3,479 (20.8%) | 12,357 (53.1%) | 12,331 (53.0%) | 5,681 (19.7%) | 5,860 (20.3%) | 21,510 (31.2%) | 21,670 (31.5%) | -0.0 |
| West; n (%) | 2,861 (17.1%) | 2,869 (17.1%) | 2,142 (9.2%) | 2,164 (9.3%) | 5,046 (17.5%) | 4,992 (17.3%) | 10,049 (14.6%) | 10,025 (14.6%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | 272 (1.2%) | 273 (1.2%) | N/A | N/A | 272 (1.2%) | 273 (1.2%) | 0.00 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 2,400 (14.3%) | 2,439 (14.6%) | 2,833 (12.2%) | 2,838 (12.2%) | 7,091 (24.6%) | 7,225 (25.0%) | 12,324 (17.9%) | 12,502 (18.2%) | -0.0 |
| Acute MI; n (%) | 46 (0.3%) | 38 (0.2%) | 62 (0.3%) | 56 (0.2%) | 111 (0.4%) | 100 (0.3%) | 219 (0.3%) | 194 (0.3%) | 0.00 |
| ACS/unstable angina; n (%) | 75 (0.4%) | 74 (0.4%) | 84 (0.4%) | 78 (0.3%) | 146 (0.5%) | 147 (0.5%) | 305 (0.4%) | 299 (0.4%) | 0.00 |
| Old MI; n (%) | 266 (1.6%) | 282 (1.7%) | 167 (0.7%) | 191 (0.8%) | 701 (2.4%) | 697 (2.4%) | 1,134 (1.6%) | 1,170 (1.7%) | -0.0 |
| Stable angina; n (%) | 331 (2.0%) | 344 (2.1%) | 327 (1.4%) | 308 (1.3%) | 849 (2.9%) | 855 (3.0%) | 1,507 (2.2%) | 1,507 (2.2%) | 0.00 |
| Coronary atherosclerosis and other forms of chronic | 2 200 (12 50/) | 2 244 (42 00/) | 2 (70 (11 50/) | 2 (00 (11 50)) | C 012 (22 C0/) | C 010 (24 08/) | 44 754 (47 40/) | 11.010/17.20() | -0.03 |
| ischemic heart disease; n (%) Other atherosclerosis with ICD10 Copy; n (%) | 2,260 (13.5%)<br>66 (0.4%) | 2,311 (13.8%)<br>71 (0.4%) | 2,679 (11.5%)<br>89 (0.4%) | 2,680 (11.5%)<br>130 (0.6%) | 6,812 (23.6%)<br>271 (0.9%) | 6,919 (24.0%)<br>336 (1.2%) | 11,751 (17.1%)<br>426 (0.6%) | 11,910 (17.3%)<br>537 (0.8%) | -0.03 |
| Previous cardiac procedure (CABG or PTCA or Stent); | bb (U.4%) | 71 (0.4%) | 89 (0.4%) | 130 (0.6%) | 271 (0.9%) | 336 (1.2%) | 426 (0.6%) | 537 (0.8%) | -0.02 |
| n (%) | 26 (0.2%) | 17 (0.1%) | 27 (0.1%) | 31 (0.1%) | 51 (0.2%) | 52 (0.2%) | 104 (0.2%) | 100 (0.1%) | 0.03 |
| History of CABG or PTCA; n (%) | 502 (3.0%) | 496 (3.0%) | 344 (1.5%) | 326 (1.4%) | 1,690 (5.9%) | 1,666 (5.8%) | 2,536 (3.7%) | 2,488 (3.6%) | 0.01 |
| Any stroke; n (%) | 447 (2.7%) | 446 (2.7%) | 432 (1.9%) | 464 (2.0%) | 1,546 (5.4%) | 1,579 (5.5%) | 2,425 (3.5%) | 2,489 (3.6%) | -0.0 |
| Ischemic stroke (w and w/o mention of cerebral | , , | ., | . , , | , , , , | , ( , | , ( , | , - ( , | ,, | |
| infarction); n (%) | 441 (2.6%) | 443 (2.6%) | 432 (1.9%) | 459 (2.0%) | 1,544 (5.4%) | 1,571 (5.4%) | 2,417 (3.5%) | 2,473 (3.6%) | -0.03 |
| Hemorrhagic stroke; n (%) | 6 (0.0%) | 5 (0.0%) | 1 (0.0%) | 6 (0.0%) | ** | ** | ** | ** | * |
| TIA; n (%) | 55 (0.3%) | 52 (0.3%) | 51 (0.2%) | 44 (0.2%) | 171 (0.6%) | 152 (0.5%) | 277 (0.4%) | 248 (0.4%) | 0.00 |
| Other cerebrovascular disease; n (%) | 121 (0.7%) | 109 (0.7%) | 104 (0.4%) | 96 (0.4%) | 314 (1.1%) | 331 (1.1%) | 539 (0.8%) | 536 (0.8%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) | 95 (0.6%) | 75 (0.4%) | 39 (0.2%) | 49 (0.2%) | 224 (0.8%) | 244 (0.8%) | 358 (0.5%) | 368 (0.5%) | 0.00 |
| Cerebrovascular procedure; n (%) | 6 (0.0%) | 5 (0.0%) | 2 (0.0%) | 4 (0.0%) | 13 (0.0%) | 17 (0.1%) | 021 (0.0%) | 026 (0.0%) | #DIV/0 |
| Heart failure (CHF); n (%) | 626 (3.7%) | 624 (3.7%) | 463 (2.0%) | 463 (2.0%) | 1,993 (6.9%) | 1,994 (6.9%) | 3,082 (4.5%) | 3,081 (4.5%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n | | | | | | 2 | | 0.00= (5.00) | |
| (%) | 705 (4.2%) | 715 (4.3%) | 610 (2.6%) | 610 (2.6%) | 2,231 (7.7%) | 2,292 (7.9%) | 3,546 (5.2%) | 3,617 (5.3%) | 0.00 |
| Atrial fibrillation; n (%) | 703 (4.2%) | 724 (4.3%) | 745 (3.2%) | 745 (3.2%) | 2,434 (8.4%) | 2,409 (8.4%) | 3,882 (5.6%) | 3,878 (5.6%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 873 (5.2%) | 880 (5.3%) | 744 (3.2%) | 784 (3.4%) | 2,760 (9.6%) | 2,761 (9.6%) | 4,377 (6.4%) | 4,425 (6.4%) | 0.00 |
| Cardiac conduction disorders; n (%) Other CVD; n (%) | 231 (1.4%)<br>975 (5.8%) | 224 (1.3%)<br>995 (5.9%) | 223 (1.0%)<br>1,144 (4.9%) | 206 (0.9%)<br>1,136 (4.9%) | 815 (2.8%)<br>3,065 (10.6%) | 751 (2.6%)<br>3,147 (10.9%) | 1,269 (1.8%)<br>5,184 (7.5%) | 1,181 (1.7%)<br>5,278 (7.7%) | -0.01 |
| Diabetes-related complications | 3/3(3.8%) | 330 (3.5%) | 1,144 (4.9%) | 1,130 (4.9%) | 3,003 (10.6%) | 5,147 (10.9%) | 3,104 (7.5%) | 3,210 (1.170) | -0.0. |
| Diabetic retinopathy; n (%) | 893 (5.3%) | 950 (5.7%) | 894 (3.8%) | 931 (4.0%) | 2,088 (7.2%) | 2,176 (7.5%) | 3,875 (5.6%) | 4,057 (5.9%) | -0.03 |
| Diabetes with other ophthalmic manifestations; n | 053 (3.3%) | 330 (3.7%) | 054 (3.0%) | 331 (4.0%) | 2,000 (7.2%) | 2,170 (7.370) | 3,073 (3.0%) | (0/C.C) 1CO,F | -0.0. |
| (%) | 89 (0.5%) | 98 (0.6%) | 544 (2.3%) | 556 (2.4%) | 829 (2.9%) | 817 (2.8%) | 1,462 (2.1%) | 1,471 (2.1%) | 0.00 |
| Retinal detachment, vitreous hemorrhage, | ( | ( | - ( 2/-/ | , | (/-/ | - , / | | . , , | |
| vitrectomy; n (%) | 65 (0.4%) | 60 (0.4%) | 62 (0.3%) | 60 (0.3%) | 133 (0.5%) | 118 (0.4%) | 260 (0.4%) | 238 (0.3%) | 0.02 |
| Retinal laser coagulation therapy; n (%) | 102 (0.6%) | 102 (0.6%) | 106 (0.5%) | 109 (0.5%) | 182 (0.6%) | 202 (0.7%) | 390 (0.6%) | 413 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy Copy; n (%) | 2,833 (16.9%) | 2,850 (17.0%) | 2,441 (10.5%) | 2,499 (10.7%) | 5,678 (19.7%) | 5,713 (19.8%) | 10,952 (15.9%) | 11,062 (16.1%) | -0.03 |

| Occurrence of diabetic nephropathy with ICD10 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Copy; n (%) | 1,592 (9.5%) | 1,610 (9.6%) | 1,235 (5.3%) | 1,208 (5.2%) | 2,370 (8.2%) | 2,334 (8.1%) | 5,197 (7.5%) | 5,152 (7.5%) | 0.00 |
| Hypoglycemia; n (%) | 359 (2.1%) | 342 (2.0%) | 487 (2.1%) | 533 (2.3%) | 633 (2.2%) | 656 (2.3%) | 1,479 (2.1%) | 1,531 (2.2%) | -0.01 |
| Hyperglycemia; n (%) | 581 (3.5%) | 578 (3.5%) | 638 (2.7%) | 616 (2.6%) | 1,019 (3.5%) | 1,016 (3.5%) | 2,238 (3.3%) | 2,210 (3.2%) | 0.01 |
| Disorders of fluid electrolyte and acid-base balance; n | | | | | | | | | |
| (%) | 569 (3.4%) | 541 (3.2%) | 496 (2.1%) | 515 (2.2%) | 1,213 (4.2%) | 1,221 (4.2%) | 2,278 (3.3%) | 2,277 (3.3%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome<br>(HONK); n (%) | 89 (0.5%) | 74 (0.4%) | 74 (0.3%) | 71 (0.3%) | 149 (0.5%) | 141 (0.5%) | 212 (0 59/) | 286 (0.4%) | 0.01 |
| Diabetes with peripheral circulatory disorders with | 09 (0.5%) | 74 (0.4%) | 74 (0.5%) | 71 (0.5%) | 149 (0.5%) | 141 (0.5%) | 312 (0.5%) | 200 (0.4%) | 0.01 |
| ICD-10 Copy; n (%) | 789 (4.7%) | 773 (4.6%) | 548 (2.4%) | 565 (2.4%) | 1,805 (6.3%) | 1,788 (6.2%) | 3,142 (4.6%) | 3,126 (4.5%) | 0.00 |
| Diabetic Foot; n (%) | 230 (1.4%) | 217 (1.3%) | 237 (1.0%) | 258 (1.1%) | 555 (1.9%) | 559 (1.9%) | 1,022 (1.5%) | 1,034 (1.5%) | 0.00 |
| Gangrene ; n (%) | 14 (0.1%) | 20 (0.1%) | 17 (0.1%) | 5 (0.0%) | 28 (0.1%) | 19 (0.1%) | 059 (0.1%) | 044 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 40 (0.2%) | 46 (0.3%) | 21 (0.1%) | 24 (0.1%) | 87 (0.3%) | 84 (0.3%) | 148 (0.2%) | 154 (0.2%) | 0.00 |
| Osteomyelitis; n (%) | 50 (0.3%) | 41 (0.2%) | 56 (0.2%) | 45 (0.2%) | 77 (0.3%) | 74 (0.3%) | 183 (0.3%) | 160 (0.2%) | 0.02 |
| Skin infections; n (%) | 812 (4.9%) | 778 (4.6%) | 925 (4.0%) | 943 (4.1%) | 1,598 (5.5%) | 1,605 (5.6%) | 3,335 (4.8%) | 3,326 (4.8%) | 0.00 |
| Erectile dysfunction; n (%) | 587 (3.5%) | 575 (3.4%) | 686 (2.9%) | 655 (2.8%) | 830 (2.9%) | 860 (3.0%) | 2,103 (3.1%) | 2,090 (3.0%) | 0.01 |
| Diabetes with unspecified complication; n (%) | 836 (5.0%) | 814 (4.9%) | 988 (4.2%) | 990 (4.3%) | 1,526 (5.3%) | 1,517 (5.3%) | 3,350 (4.9%) | 3,321 (4.8%) | 0.00 |
| Diabetes mellitus without mention of complications; | | | | | | | | | |
| n (%) | 14,237 (85.0%) | 14,249 (85.1%) | 21,402 (92.0%) | 21,452 (92.2%) | 26,407 (91.5%) | 26,443 (91.7%) | 62,046 (90.1%) | 62,144 (90.3%) | -0.01 |
| Hypertension: 1 inpatient or 2 outpatient claims | | | | | | | | | |
| within 365 days; n (%) | 15,348 (91.7%) | 15,341 (91.6%) | 20,375 (87.6%) | 20,341 (87.4%) | 27,592 (95.7%) | 27,624 (95.8%) | 63,315 (92.0%) | 63,306 (91.9%) | 0.00 |
| Hyperlipidemia; n (%) | 12,921 (77.2%) | 12,951 (77.4%) | 17,546 (75.4%) | 17,573 (75.5%) | 23,820 (82.6%) | 23,824 (82.6%) | 54,287 (78.8%) | 54,348 (78.9%) | 0.00 |
| Edema; n (%) | 721 (4.3%)<br>1,611 (9.6%) | 741 (4.4%) | 728 (3.1%) | 727 (3.1%) | 2,166 (7.5%) | 2,095 (7.3%) | 3,615 (5.3%) | 3,563 (5.2%)<br>6,323 (9.2%) | 0.00<br>0.01 |
| Renal Dysfunction (non-diabetic); n (%) | 1,611 (9.6%) | 1,605 (9.6%)<br>135 (0.8%) | 1,291 (5.5%)<br>89 (0.4%) | 1,199 (5.2%)<br>92 (0.4%) | 3,614 (12.5%) | 3,519 (12.2%)<br>320 (1.1%) | 6,516 (9.5%)<br>535 (0.8%) | 547 (0.8%) | 0.00 |
| Occurrence of acute renal disease; n (%) Occurrence of chronic renal insufficiency; n (%) | 1,286 (7.7%) | 1,321 (7.9%) | 910 (3.9%) | 861 (3.7%) | 300 (1.0%)<br>2,943 (10.2%) | 2,882 (10.0%) | 5,139 (7.5%) | 5,064 (7.4%) | 0.00 |
| Chronic kidney disease ; n (%) | 1,211 (7.2%) | 1,235 (7.4%) | 834 (3.6%) | 743 (3.2%) | 2,753 (9.5%) | 2,646 (9.2%) | 4,798 (7.0%) | 4,624 (6.7%) | 0.01 |
| CKD Stage 3-4; n (%) | 628 (3.8%) | 635 (3.8%) | 398 (1.7%) | 370 (1.6%) | 1,538 (5.3%) | 1,534 (5.3%) | 2,564 (3.7%) | 2,539 (3.7%) | 0.00 |
| Occurrence of hypertensive nephropathy; n (%) | 553 (3.3%) | 537 (3.2%) | 283 (1.2%) | 295 (1.3%) | 990 (3.4%) | 1,006 (3.5%) | 1,826 (2.7%) | 1,838 (2.7%) | 0.00 |
| Occurrence of miscellaneous renal insufficiency ; n | 000 (0.07.) | () | () | | ( | _,,,,, | _,=== (= ,-, | _,, | |
| (%) | 318 (1.9%) | 314 (1.9%) | 375 (1.6%) | 368 (1.6%) | 1,003 (3.5%) | 1,026 (3.6%) | 1,696 (2.5%) | 1,708 (2.5%) | 0.00 |
| Glaucoma or cataracts ; n (%) | 2,814 (16.8%) | 2,806 (16.8%) | 3,187 (13.7%) | 3,120 (13.4%) | 7,913 (27.4%) | 7,842 (27.2%) | 13,914 (20.2%) | 13,768 (20.0%) | 0.00 |
| Cellulitis or abscess of toe; n (%) | 176 (1.1%) | 146 (0.9%) | 129 (0.6%) | 132 (0.6%) | 332 (1.2%) | 306 (1.1%) | 637 (0.9%) | 584 (0.8%) | 0.01 |
| Foot ulcer; n (%) | 217 (1.3%) | 205 (1.2%) | 233 (1.0%) | 255 (1.1%) | 542 (1.9%) | 556 (1.9%) | 992 (1.4%) | 1,016 (1.5%) | -0.01 |
| Bladder stones; n (%) | 11 (0.1%) | 12 (0.1%) | 24 (0.1%) | 16 (0.1%) | 41 (0.1%) | 37 (0.1%) | 076 (0.1%) | 065 (0.1%) | 0.00 |
| Kidney stones; n (%) | 267 (1.6%) | 256 (1.5%) | 428 (1.8%) | 414 (1.8%) | 667 (2.3%) | 653 (2.3%) | 1,362 (2.0%) | 1,323 (1.9%) | 0.01 |
| Urinary tract infections (UTIs); n (%) | 850 (5.1%) | 871 (5.2%) | 926 (4.0%) | 923 (4.0%) | 2,574 (8.9%) | 2,543 (8.8%) | 4,350 (6.3%) | 4,337 (6.3%) | 0.00 |
| Dipstick urinalysis; n (%) | 5,198 (31.1%) | 5,250 (31.4%) | 7,224 (31.1%) | 7,104 (30.5%) | 10,370 (36.0%) | 10,618 (36.8%) | 22,792 (33.1%) | 22,972 (33.4%) | -0.01 |
| Non-dipstick urinalysis; n (%) | 7,491 (44.7%) | 7,645 (45.7%) | 9,491 (40.8%) | 9,736 (41.8%) | 13,163 (45.6%) | 13,338 (46.2%) | 30,145 (43.8%) | 30,719 (44.6%) | -0.02 |
| Urine function test; n (%) | 275 (1.6%) | 224 (1.3%) | 362 (1.6%) | 304 (1.3%) | 893 (3.1%) | 797 (2.8%) | 1,530 (2.2%) | 1,325 (1.9%) | 0.02 |
| Cytology; n (%) | 76 (0.5%) | 72 (0.4%) | 136 (0.6%) | 118 (0.5%) | 208 (0.7%) | 200 (0.7%) | 420 (0.6%) | 390 (0.6%) | 0.00 |
| Cystoscopy; n (%) | 120 (0.7%) | 107 (0.6%) | 202 (0.9%) | 156 (0.7%) | 298 (1.0%) | 292 (1.0%) | 620 (0.9%) | 555 (0.8%) | 0.01 |
| Other Covariates Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 1,728 (10.3%) | 1,733 (10.4%) | 1,617 (7.0%) | 1,622 (7.0%) | 4,923 (17.1%) | 4,854 (16.8%) | 8,268 (12.0%) | 8,209 (11.9%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | 1,728 (10.378) | 1,733 (10.476) | 1,017 (7.078) | 1,022 (7.076) | 4,923 (17.170) | 4,834 (10.878) | 8,208 (12.078) | 8,203 (11.370) | 0.00 |
| pain; n (%) | 4,582 (27.4%) | 4,572 (27.3%) | 5,474 (23.5%) | 5,476 (23.5%) | 10,139 (35.1%) | 10,202 (35.4%) | 20,195 (29.3%) | 20,250 (29.4%) | 0.00 |
| Dorsopathies; n (%) | 3,062 (18.3%) | 2,956 (17.7%) | 3,524 (15.1%) | 3,554 (15.3%) | 6,484 (22.5%) | 6,550 (22.7%) | 13,070 (19.0%) | 13,060 (19.0%) | 0.00 |
| Fractures; n (%) | 284 (1.7%) | 289 (1.7%) | 333 (1.4%) | 333 (1.4%) | 677 (2.3%) | 677 (2.3%) | 1,294 (1.9%) | 1,299 (1.9%) | 0.00 |
| Falls; n (%) | 318 (1.9%) | 286 (1.7%) | 106 (0.5%) | 120 (0.5%) | 630 (2.2%) | 648 (2.2%) | 1,054 (1.5%) | 1,054 (1.5%) | 0.00 |
| Osteoporosis; n (%) | 453 (2.7%) | 444 (2.7%) | 326 (1.4%) | 303 (1.3%) | 1,765 (6.1%) | 1,786 (6.2%) | 2,544 (3.7%) | 2,533 (3.7%) | 0.00 |
| Hyperthyroidism; n (%) | 121 (0.7%) | 87 (0.5%) | 117 (0.5%) | 97 (0.4%) | 251 (0.9%) | 242 (0.8%) | 489 (0.7%) | 426 (0.6%) | 0.01 |
| Hypothyroidism ; n (%) | 2,426 (14.5%) | 2,438 (14.6%) | 2,825 (12.1%) | 2,723 (11.7%) | 3,638 (12.6%) | 3,615 (12.5%) | 8,889 (12.9%) | 8,776 (12.7%) | 0.01 |
| Other disorders of thyroid gland; n (%) | 664 (4.0%) | 631 (3.8%) | 840 (3.6%) | 824 (3.5%) | 1,287 (4.5%) | 1,291 (4.5%) | 2,791 (4.1%) | 2,746 (4.0%) | 0.01 |
| Depression; n (%) | 1,229 (7.3%) | 1,217 (7.3%) | 1,471 (6.3%) | 1,423 (6.1%) | 2,574 (8.9%) | 2,543 (8.8%) | 5,274 (7.7%) | 5,183 (7.5%) | 0.01 |
| Anxiety; n (%) | 1,167 (7.0%) | 1,136 (6.8%) | 1,084 (4.7%) | 1,088 (4.7%) | 2,123 (7.4%) | 2,036 (7.1%) | 4,374 (6.4%) | 4,260 (6.2%) | 0.01 |
| Sleep_Disorder; n (%) | 1,227 (7.3%) | 1,260 (7.5%) | 2,580 (11.1%) | 2,582 (11.1%) | 2,379 (8.2%) | 2,430 (8.4%) | 6,186 (9.0%) | 6,272 (9.1%) | 0.00 |
| Dementia; n (%) | 155 (0.9%) | 162 (1.0%) | 112 (0.5%) | 120 (0.5%) | 902 (3.1%) | 938 (3.3%) | 1,169 (1.7%) | 1,220 (1.8%) | -0.01 |
| Delirium; n (%) | 39 (0.2%) | 46 (0.3%) | 36 (0.2%) | 35 (0.2%) | 179 (0.6%) | 186 (0.6%) | 254 (0.4%) | 267 (0.4%) | 0.00 |
| Psychosis; n (%) | 65 (0.4%) | 77 (0.5%) | 32 (0.1%) | 44 (0.2%) | 223 (0.8%) | 257 (0.9%) | 320 (0.5%) | 378 (0.5%) | 0.00 |
| Obesity; n (%) | 4,419 (26.4%) | 4,456 (26.6%) | 4,267 (18.3%) | 4,308 (18.5%) | 5,666 (19.6%) | 5,680 (19.7%) | 14,352 (20.8%) | 14,444 (21.0%) | 0.00 |
| Overweight; n (%) Smoking; n (%) | 838 (5.0%)<br>1,399 (8.4%) | 841 (5.0%)<br>1,383 (8.3%) | 537 (2.3%)<br>1,206 (5.2%) | 530 (2.3%)<br>1,169 (5.0%) | 1,065 (3.7%)<br>3,129 (10.8%) | 1,063 (3.7%) | 2,440 (3.5%)<br>5,734 (8.3%) | 2,434 (3.5%)<br>5,717 (8.3%) | 0.00<br>0.00 |
| Smoking; n (%) Alcohol abuse or dependence; n (%) | 1,399 (8.4%)<br>5 (0.0%) | 1,383 (8.3%)<br>0 (0.0%) | 1,206 (5.2%)<br>7 (0.0%) | 1,169 (5.0%)<br>6 (0.0%) | 3,129 (10.8%) | 3,165 (11.0%)<br>** | 5,/34 (8.3%) | 5,/1/ (8.3%) | 0.00 |
| Drug abuse or dependence; n (%) | 3 (0.0%) | 7 (0.0%) | 4 (0.0%) | 4 (0.0%) | ** | ** | ** | ** | ** |
| COPD; n (%) | 851 (5.1%) | 834 (5.0%) | 633 (2.7%) | 643 (2.8%) | 2,322 (8.0%) | 2,360 (8.2%) | 3,806 (5.5%) | 3,837 (5.6%) | 0.00 |
| | 032 (3.270) | 33. (3.070) | 000 (2.770) | 0.5(2.5/0) | 2,522 (5.570) | 2,555 (5.270) | 5,000 (5.570) | 3,037 (3.070) | 3.00 |

| Asthma; n (%) | 846 (5.1%) | 794 (4.7%) | 817 (3.5%) | 834 (3.6%) | 1,494 (5.2%) | 1,542 (5.3%) | 3,157 (4.6%) | 3,170 (4.6%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 1,899 (11.3%) | 1,960 (11.7%) | 2,788 (12.0%) | 2,804 (12.1%) | 2,661 (9.2%) | 2,680 (9.3%) | 7,348 (10.7%) | 7,444 (10.8%) | 0.00 |
| Pneumonia; n (%) | 181 (1.1%) | 190 (1.1%) | 187 (0.8%) | 208 (0.9%) | 471 (1.6%) | 474 (1.6%) | 839 (1.2%) | 872 (1.3%) | -0.01 |
| Imaging; n (%) | 2 (0.0%) | 3 (0.0%) | 3 (0.0%) | 3 (0.0%) | 15 (0.1%) | 12 (0.0%) | 20 (0.0%) | 18 (0.0%) | #DIV/0! |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 61 (0.4%) | 63 (0.4%) | 72 (0.3%) | 73 (0.3%) | 180 (0.6%) | 197 (0.7%) | 313 (0.5%) | 333 (0.5%) | 0.00 |
| DM Medications - Glitazones; n (%) | 1,570 (9.4%) | 1,478 (8.8%) | 2,106 (9.1%) | 2,058 (8.8%) | 2,732 (9.5%) | 2,715 (9.4%) | 6,408 (9.3%) | 6,251 (9.1%) | 0.01 |
| DM Medications - Insulin; n (%) | 4,643 (27.7%) | 4,731 (28.3%) | 6,185 (26.6%) | 6,447 (27.7%) | 9,686 (33.6%) | 9,923 (34.4%) | 20,514 (29.8%) | 21,101 (30.6%) | -0.02 |
| DM Medications - Meglitinides; n (%) | 227 (1.4%) | 223 (1.3%) | 418 (1.8%) | 421 (1.8%) | 744 (2.6%) | 791 (2.7%) | 1,389 (2.0%) | 1,435 (2.1%) | -0.01 |
| DM Medications - Metformin; n (%) | 13,035 (77.9%) | 13,035 (77.9%) | 18,359 (78.9%) | 18,245 (78.4%) | 21,390 (74.2%) | 21,384 (74.1%) | 52,784 (76.7%) | 52,664 (76.5%) | 0.00 |
| Concomitant initiation or current use of DPP4i Copy; | | | | | | | | | |
| n (%) | 3,291 (19.7%) | 3,255 (19.4%) | 5,946 (25.6%) | 5,704 (24.5%) | 7,563 (26.2%) | 7,384 (25.6%) | 16,800 (24.4%) | 16,343 (23.7%) | 0.02 |
| Concomitant initiation or current use of AGIs; n (%) | 40 (0.2%) | 45 (0.3%) | 44 (0.2%) | 36 (0.2%) | 124 (0.4%) | 139 (0.5%) | 208 (0.3%) | 220 (0.3%) | 0.00 |
| Concomitant initiation or current use of Glitazones; | 4 220 (7 20/) | 1 122 (6 00/) | 1,583 (6.8%) | 1 544 (C CO/) | 2.064 (7.49/) | 2.000 (7.10/) | 4.074 (7.40/) | 4 727 (C 00/) | 0.01 |
| n (%) Concomitant initiation or current use of GLP-1 RA; n | 1,230 (7.3%) | 1,133 (6.8%) | 1,363 (0.6%) | 1,544 (6.6%) | 2,061 (7.1%) | 2,060 (7.1%) | 4,874 (7.1%) | 4,737 (6.9%) | 0.01 |
| (%) | 1,791 (10.7%) | 1,857 (11.1%) | 2,706 (11.6%) | 2,734 (11.8%) | 2,458 (8.5%) | 2,727 (9.5%) | 6,955 (10.1%) | 7,318 (10.6%) | -0.02 |
| Concomitant initiation or current use of Insulin; n | 1,731 (10.778) | 1,037 (11.170) | 2,700 (11.0%) | 2,734 (11.670) | 2,438 (8.378) | 2,727 (3.370) | 0,933 (10.170) | 7,318 (10.0%) | -0.02 |
| (%) | 3,487 (20.8%) | 3,579 (21.4%) | 4,765 (20.5%) | 4,982 (21.4%) | 7,619 (26.4%) | 7,943 (27.5%) | 15,871 (23.1%) | 16,504 (24.0%) | -0.02 |
| Concomitant initiation or current use of | 5,107 (20.070) | 3,373 (22.170) | 1,705 (20.5%) | 1,502 (21.170) | 7,015 (20.170) | 7,5 15 (27.570) | 15,071 (25.170) | 10,50 1 (2 1.070) | 0.02 |
| Meglitinides; n (%) | 130 (0.8%) | 155 (0.9%) | 241 (1.0%) | 289 (1.2%) | 526 (1.8%) | 563 (2.0%) | 897 (1.3%) | 1,007 (1.5%) | -0.02 |
| Concomitant initiation or current use of Metformin; | , | , | ,, | | , | , | . , | ,, | |
| n (%) | 10,980 (65.6%) | 10,982 (65.6%) | 15,378 (66.1%) | 15,321 (65.9%) | 18,049 (62.6%) | 18,065 (62.6%) | 44,407 (64.5%) | 44,368 (64.4%) | 0.00 |
| Past use of DPP4i Copy; n (%) | 1,151 (6.9%) | 1,121 (6.7%) | 1,783 (7.7%) | 1,697 (7.3%) | 2,213 (7.7%) | 2,127 (7.4%) | 5,147 (7.5%) | 4,945 (7.2%) | 0.01 |
| Past use of AGIs Copy; n (%) | 21 (0.1%) | 18 (0.1%) | 28 (0.1%) | 37 (0.2%) | 56 (0.2%) | 58 (0.2%) | 105 (0.2%) | 113 (0.2%) | 0.00 |
| Past use of Glitazones Copy; n (%) | 340 (2.0%) | 345 (2.1%) | 523 (2.2%) | 514 (2.2%) | 671 (2.3%) | 655 (2.3%) | 1,534 (2.2%) | 1,514 (2.2%) | 0.00 |
| Past use of GLP-1 RA Copy; n (%) | 823 (4.9%) | 826 (4.9%) | 1,206 (5.2%) | 1,219 (5.2%) | 1,172 (4.1%) | 1,224 (4.2%) | 3,201 (4.6%) | 3,269 (4.7%) | 0.00 |
| Past use of Insulin Copy; n (%) | 1,156 (6.9%) | 1,152 (6.9%) | 1,420 (6.1%) | 1,465 (6.3%) | 2,067 (7.2%) | 1,981 (6.9%) | 4,643 (6.7%) | 4,598 (6.7%) | 0.00 |
| Past use of Meglitinides Copy; n (%) | 97 (0.6%) | 68 (0.4%) | 177 (0.8%) | 132 (0.6%) | 218 (0.8%) | 228 (0.8%) | 492 (0.7%) | 428 (0.6%) | 0.01 |
| Past use of metformin (final) Copy; n (%) | 2,055 (12.3%) | 2,053 (12.3%) | 2,981 (12.8%) | 2,924 (12.6%) | 3,341 (11.6%) | 3,319 (11.5%) | 8,377 (12.2%) | 8,296 (12.0%) | 0.01 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 8,762 (52.3%) | 8,727 (52.1%) | 11,715 (50.4%) | 11,848 (50.9%) | 13,662 (47.4%) | 13,602 (47.2%) | 34,139 (49.6%) | 34,177 (49.6%) | 0.00 |
| Use of ARBs; n (%) | 6,316 (37.7%) | 6,365 (38.0%) | 9,235 (39.7%) | 9,169 (39.4%) | 11,406 (39.5%) | 11,415 (39.6%) | 26,957 (39.2%) | 26,949 (39.1%) | 0.00 |
| Use of Loop Diuretics ; n (%) | 1,436 (8.6%) | 1,463 (8.7%) | 1,706 (7.3%) | 1,750 (7.5%) | 4,396 (15.2%) | 4,395 (15.2%) | 7,538 (10.9%) | 7,608 (11.1%) | -0.01 |
| Use of other diuretics; n (%) | 460 (2.7%) | 456 (2.7%) | 595 (2.6%) | 579 (2.5%) | 975 (3.4%) | 981 (3.4%) | 2,030 (2.9%) | 2,016 (2.9%) | 0.00 |
| Use of nitrates-United; n (%) | 570 (3.4%) | 543 (3.2%) | 673 (2.9%) | 696 (3.0%) | 1,759 (6.1%) | 1,776 (6.2%) | 3,002 (4.4%) | 3,015 (4.4%) | 0.00 |
| Use of other hypertension drugs; n (%) | 836 (5.0%) | 841 (5.0%) | 1,023 (4.4%) | 1,042 (4.5%) | 2,103 (7.3%) | 2,069 (7.2%) | 3,962 (5.8%) | 3,952 (5.7%) | 0.00 |
| Use of digoxin; n (%) | 160 (1.0%) | 175 (1.0%) | 214 (0.9%) | 221 (0.9%) | 654 (2.3%) | 606 (2.1%) | 1,028 (1.5%) | 1,002 (1.5%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 147 (0.9%) | 146 (0.9%) | 189 (0.8%) | 190 (0.8%) | 433 (1.5%) | 440 (1.5%) | 769 (1.1%) | 776 (1.1%) | 0.00 |
| Use of COPD/asthma meds; n (%) | 2,395 (14.3%) | 2,326 (13.9%) | 3,399 (14.6%) | 3,371 (14.5%) | 4,932 (17.1%) | 4,962 (17.2%) | 10,726 (15.6%) | 10,659 (15.5%) | 0.00 |
| Use of statins; n (%) | 12,032 (71.9%) | 12,150 (72.6%) | 16,087 (69.1%) | 16,153 (69.4%) | 21,847 (75.7%) | 21,876 (75.8%) | 49,966 (72.6%) | 50,179 (72.9%) | -0.01 |
| Use of other lipid-lowering drugs; n (%) | 2,203 (13.2%) | 2,259 (13.5%) | 3,621 (15.6%) | 3,669 (15.8%) | 4,378 (15.2%) | 4,409 (15.3%) | 10,202 (14.8%) | 10,337 (15.0%) | -0.01 |
| Use of antiplatelet agents; n (%) | 1,646 (9.8%) | 1,642 (9.8%) | 2,383 (10.2%) | 2,401 (10.3%) | 4,209 (14.6%) | 4,265 (14.8%) | 8,238 (12.0%) | 8,308 (12.1%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | | | | |
| Apixaban, Warfarin); n (%) | 711 (4.2%) | 713 (4.3%) | 774 (3.3%) | 785 (3.4%) | 2,191 (7.6%) | 2,225 (7.7%) | 3,676 (5.3%) | 3,723 (5.4%) | 0.00 |
| Use of heparin and other low-molecular weight | 47 (0 40() | 45 (0.40() | 0 (0 00/) | 0 (0 00() | 62 (0.20() | 50 (0.20() | 000 (0.40() | 005 (0.40() | 0.00 |
| heparins; n (%) | 17 (0.1%) | 16 (0.1%) | 0 (0.0%)<br>3,777 (16.2%) | 0 (0.0%)<br>3,810 (16.4%) | 63 (0.2%) | 69 (0.2%) | 080 (0.1%) | 085 (0.1%) | 0.00 |
| Use of NSAIDs; n (%) | 2,804 (16.8%)<br>2,110 (12.6%) | 2,766 (16.5%)<br>2,010 (12.0%) | 2,618 (11.3%) | 2,588 (11.1%) | 4,635 (16.1%) | 4,674 (16.2%)<br>4,125 (14.3%) | 11,216 (16.3%)<br>8,864 (12.9%) | 11,250 (16.3%) | 0.00 |
| Use of oral corticosteroids; n (%) Use of bisphosphonate (United); n (%) | 2,110 (12.6%) | 2,010 (12.0%) | 2,618 (11.3%)<br>164 (0.7%) | 2,588 (11.1%)<br>155 (0.7%) | 4,136 (14.3%)<br>811 (2.8%) | 4,125 (14.3%)<br>819 (2.8%) | 1,184 (1.7%) | 8,723 (12.7%)<br>1,176 (1.7%) | 0.00 |
| Use of opioids; n (%) | 3,250 (19.4%) | 3,204 (19.1%) | 4,506 (19.4%) | 4,557 (19.6%) | 5,860 (20.3%) | 5,864 (20.3%) | 13,616 (19.8%) | 13,625 (19.8%) | 0.00 |
| Use of antidepressants; n (%) | 3,994 (23.9%) | 3,963 (23.7%) | 5,150 (22.1%) | 5,158 (22.2%) | 7,507 (26.0%) | 7,437 (25.8%) | 16,651 (24.2%) | 16,558 (24.0%) | 0.00 |
| Use of antipsychotics; n (%) | 300 (1.8%) | 303 (1.8%) | 281 (1.2%) | 287 (1.2%) | 678 (2.4%) | 701 (2.4%) | 1,259 (1.8%) | 1,291 (1.9%) | -0.01 |
| Use of anticonvulsants; n (%) | 2,436 (14.6%) | 2,322 (13.9%) | 2,448 (10.5%) | 2,480 (10.7%) | 4,502 (15.6%) | 4,524 (15.7%) | 9,386 (13.6%) | 9,326 (13.5%) | 0.00 |
| Use of lithium; n (%) | 15 (0.1%) | 20 (0.1%) | 33 (0.1%) | 11 (0.0%) | 38 (0.1%) | 27 (0.1%) | 086 (0.1%) | 058 (0.1%) | 0.00 |
| Use of Benzos; n (%) | 1,504 (9.0%) | 1,501 (9.0%) | 1,957 (8.4%) | 1,972 (8.5%) | 2,903 (10.1%) | 2,856 (9.9%) | 6,364 (9.2%) | 6,329 (9.2%) | 0.00 |
| Use of anxiolytics/hypnotics; n (%) | 932 (5.6%) | 906 (5.4%) | 1,304 (5.6%) | 1,324 (5.7%) | 1,707 (5.9%) | 1,632 (5.7%) | 3,943 (5.7%) | 3,862 (5.6%) | 0.00 |
| Use of dementia meds; n (%) | 104 (0.6%) | 112 (0.7%) | 82 (0.4%) | 88 (0.4%) | 760 (2.6%) | 785 (2.7%) | 946 (1.4%) | 985 (1.4%) | 0.00 |
| Use of antiparkinsonian meds; n (%) | 322 (1.9%) | 325 (1.9%) | 374 (1.6%) | 362 (1.6%) | 830 (2.9%) | 852 (3.0%) | 1,526 (2.2%) | 1,539 (2.2%) | 0.00 |
| Any use of pramlintide; n (%) | 0 (0.0%) | 28 (0.2%) | 10 (0.0%) | 41 (0.2%) | ** | ** | ** | ** | ** |
| Any use of 1st generation sulfonylureas; n (%) | 1 (0.0%) | 2 (0.0%) | 6 (0.0%) | 1 (0.0%) | ** | ** | ** | ** | ** |
| Entresto (sacubitril/valsartan); n (%) | 15 (0.1%) | 8 (0.0%) | 10 (0.0%) | 6 (0.0%) | ** | ** | ** | ** | ** |
| Initiation as monotherapy Copy; n (%) | 1,194 (7.1%) | 1,198 (7.2%) | 1,283 (5.5%) | 1,306 (5.6%) | 1,205 (4.2%) | 1,233 (4.3%) | 3,682 (5.3%) | 3,737 (5.4%) | 0.00 |
| Labs | , () | , - = (- := := / | , -= (=:=:-) | , = (=====) | , -= (::=:=/ | , -= (::=::) | 40,005 | 40,005 | 2.30 |
| Lab values- HbA1c (%); n (%) | 7,105 (42.4%) | 7,211 (43.1%) | 1,740 (7.5%) | 1,440 (6.2%) | N/A | N/A | 8,845 (22.1%) | 8,651 (21.6%) | 0.01 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 5,645 (33.7%) | 5,910 (35.3%) | 1,376 (5.9%) | 1,224 (5.3%) | N/A | N/A | 7,021 (17.6%) | 7,134 (17.8%) | -0.01 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 7,105 (42.4%) | 7,211 (43.1%) | 1,740 (7.5%) | 1,440 (6.2%) | N/A | N/A | 8,845 (22.1%) | 8,651 (21.6%) | 0.01 |
| | , | , | , | , | • | • | , | , | |

| Lab values- BNP; n (%) | 73 (0.4%) | 99 (0.6%) | 14 (0.1%) | 13 (0.1%) | N/A | N/A | 087 (0.2%) | 112 (0.3%) | -0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP (within 3 months); n (%) | 42 (0.3%) | 64 (0.4%) | 8 (0.0%) | 9 (0.0%) | N/A | N/A | 050 (0.1%) | 073 (0.2%) | -0.03 |
| Lab values- BNP (within 6 months); n (%) | 73 (0.4%) | 99 (0.6%) | 14 (0.1%) | 13 (0.1%) | N/A | N/A | 087 (0.2%) | 112 (0.3%) | -0.02 |
| Lab values- BUN (mg/dl); n (%) | 6,923 (41.4%) | 7,113 (42.5%) | 1,610 (6.9%) | 1,347 (5.8%) | N/A | N/A | 8,533 (21.3%) | 8,460 (21.1%) | 0.00 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 5,349 (32.0%) | 5,668 (33.9%) | 1,229 (5.3%) | 1,095 (4.7%) | N/A | N/A | 6,578 (16.4%) | 6,763 (16.9%) | -0.01 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 6,923 (41.4%) | 7,113 (42.5%) | 1,610 (6.9%) | 1,347 (5.8%) | N/A | N/A | 8,533 (21.3%) | 8,460 (21.1%) | 0.00 |
| Lab values- Creatinine (mg/dl); n (%) | 7,103 (42.4%) | 7,370 (44.0%) | 1,719 (7.4%) | 1,488 (6.4%) | N/A | N/A | 8,822 (22.1%) | 8,858 (22.1%) | 0.00 |
| Lab values- Creatinine (mg/dl) (within 3 months); n | 7,103 (42.4%) | 7,370 (44.0%) | 1,719 (7.478) | 1,488 (0.4%) | 14/4 | N/A | 0,022 (22.170) | 0,030 (22.170) | 0.00 |
| | 5 404 (22 00) | 5.072 (25.40() | 4 224 (5 70() | 4 224 (5 20() | 21/2 | 21/2 | C 005 (47 00() | 7.002 (4.7.70/) | 2.22 |
| (%) | 5,484 (32.8%) | 5,872 (35.1%) | 1,321 (5.7%) | 1,221 (5.2%) | N/A | N/A | 6,805 (17.0%) | 7,093 (17.7%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 6 months) ; n | | | | | | | | | |
| (%) | 7,103 (42.4%) | | 1,719 (7.4%) | 1,488 (6.4%) | N/A | N/A | 8,822 (22.1%) | 8,858 (22.1%) | 0.00 |
| Lab values- HDL level (mg/dl); n (%) | 6,063 (36.2%) | 6,278 (37.5%) | 1,611 (6.9%) | 1,358 (5.8%) | N/A | N/A | 7,674 (19.2%) | 7,636 (19.1%) | 0.00 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 4,499 (26.9%) | 4,780 (28.6%) | 1,182 (5.1%) | 1,058 (4.5%) | N/A | N/A | 5,681 (14.2%) | 5,838 (14.6%) | -0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 6,063 (36.2%) | 6,278 (37.5%) | 1,611 (6.9%) | 1,358 (5.8%) | N/A | N/A | 7,674 (19.2%) | 7,636 (19.1%) | 0.00 |
| Lab values- LDL level (mg/dl); n (%) | 6,280 (37.5%) | 6,482 (38.7%) | 1,663 (7.1%) | 1,379 (5.9%) | N/A | N/A | 7,943 (19.9%) | 7,861 (19.7%) | 0.01 |
| === · | 0,200 (011071) | 5,102 (001111) | _,,,,, | =,0:0 (0:0::) | .,,. | , | ., (, | .,(==:::-) | |
| Lab values-LDL level (mg/dl) (within 3 months); n (%) | 4,650 (27.8%) | 4,954 (29.6%) | 1,216 (5.2%) | 1,078 (4.6%) | N/A | N/A | 5,866 (14.7%) | 6,032 (15.1%) | -0.01 |
| Lab values EDETever (IIIg/ai/ (Within 5 Honelis/ ) II (70) | 4,030 (27.0%) | 4,554 (25.0%) | 1,210 (3.270) | 1,070 (4.070) | 14/5 | 14/4 | 3,000 (14.770) | 0,032 (13.170) | 0.01 |
| 1.1 1 1.1 1 (11) (11) (11) | 6 200 (27 50() | 6 402 (20 70) | 4 662 (7 40() | 4 270 (5 00() | 21/2 | 21/2 | 7.042 (40.00() | 7.004 (40.70() | 2.24 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 6,280 (37.5%) | 6,482 (38.7%) | 1,663 (7.1%) | 1,379 (5.9%) | N/A | N/A | 7,943 (19.9%) | 7,861 (19.7%) | 0.01 |
| Lab values- NT-proBNP; n (%) | 13 (0.1%) | 9 (0.1%) | 4 (0.0%) | 0 (0.0%) | N/A | N/A | 17 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 3 months); n (%) | 9 (0.1%) | 5 (0.0%) | 2 (0.0%) | 0 (0.0%) | N/A | N/A | 11 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 13 (0.1%) | 9 (0.1%) | 4 (0.0%) | 0 (0.0%) | N/A | N/A | 17 (0.0%) | 9 (0.0%) | - |
| Lab values-Total cholesterol (mg/dl); n (%) | 6,193 (37.0%) | 6,409 (38.3%) | 1,610 (6.9%) | 1,363 (5.9%) | N/A | N/A | 7,803 (19.5%) | 7,772 (19.4%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 4,591 (27.4%) | 4,894 (29.2%) | 1,183 (5.1%) | 1,066 (4.6%) | N/A | N/A | 5,774 (14.4%) | 5,960 (14.9%) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 6 | ,,,,,,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | _,, | =,000 (, | .,,. | , | ÷/···(=·····/ | -, (= ·····-) | |
| months); n (%) | 6,193 (37.0%) | 6,409 (38.3%) | 1,610 (6.9%) | 1,363 (5.9%) | N/A | N/A | 7,803 (19.5%) | 7,772 (19.4%) | 0.00 |
| Lab values- Triglyceride level (mg/dl); n (%) | 6,139 (36.7%) | 6,366 (38.0%) | 1,598 (6.9%) | 1,343 (5.8%) | N/A | N/A | 7,737 (19.3%) | 7,772 (19.4%) | 0.00 |
| | 0,139 (30.7%) | 0,300 (38.0%) | 1,598 (6.9%) | 1,343 (3.6%) | N/A | N/A | 7,757 (19.5%) | 7,709 (19.5%) | 0.00 |
| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 4,554 (27.2%) | 4,857 (29.0%) | 1,177 (5.1%) | 1,053 (4.5%) | N/A | N/A | 5,731 (14.3%) | 5,910 (14.8%) | -0.01 |
| Lab values- Triglyceride level (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 6,139 (36.7%) | 6,366 (38.0%) | 1,598 (6.9%) | 1,343 (5.8%) | N/A | N/A | 7,737 (19.3%) | 7,709 (19.3%) | 0.00 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 7,067 | 7,168 | 1,685 | 1,391 | N/A | N/A | 8,752 | 8,559 | |
| mean (sd) | 8.55 (1.87) | 8.50 (1.76) | 8.59 (1.89) | 8.53 (1.77) | N/A | N/A | 8.56 (1.87) | 8.50 (1.76) | 0.03 |
| median [IQR] | 8.10 [7.20, 9.60] | 8.10 [7.25, 9.43] | 8.10 [7.30, 9.50] | 8.10 [7.25, 9.40] | N/A | N/A | 8.10 (1.87) | 8.10 (1.76) | 0.00 |
| Missing; n (%) | 9,673 (57.8%) | | 21,580 (92.8%) | 21,874 (94.0%) | N/A | N/A | 31,253 (78.1%) | 31,446 (78.6%) | -0.01 |
| Lab result number- BNP mean | 73 | 99 | 14 | 13 | N/A | N/A | 87 | 112 | |
| mean (sd) | 105.60 (266.26) | 68.61 (79.50) | 110.61 (177.08) | 575.59 (1,341.91) | N/A | N/A | 106.41 (256.16) | 127.46 (451.58) | -0.06 |
| | | | | | | N/A | #VALUE! | | |
| median [IQR] | 43.00 [18.05, 97.15] | 40.40 [17.00, 86.10] | 45.00 [17.75, 119.62] | 56.00 [20.00, 194.30] | N/A | | | #VALUE! | #VALUE! |
| Missing; n (%) | 16,667 (99.6%) | 16,641 (99.4%) | 23,251 (99.9%) | 23,252 (99.9%) | N/A | N/A | 39,918 (99.8%) | 39,893 (99.7%) | 0.02 |
| Lab result number- BUN (mg/dl) mean | 6,923 | 7,113 | 1,610 | 1,347 | N/A | N/A | 8,533 | 8,460 | |
| mean (sd) | 16.86 (6.32) | 16.65 (5.62) | 988.41 (11,243.54) | 2,413.80 (18,907.89) | N/A | N/A | 200.17 (4883.23) | 398.32 (7543.23) | -0.03 |
| median [IQR] | 16.00 [13.00, 19.50] | 16.00 [13.00, 19.00] | 15.83 [13.00, 19.00] | 16.00 [13.00, 19.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 9,817 (58.6%) | 9,627 (57.5%) | 21,655 (93.1%) | 21,918 (94.2%) | N/A | N/A | 31,472 (78.7%) | 31,545 (78.9%) | 0.00 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | |
| to 15 included) | 7,065 | 7,319 | 1,572 | 1,354 | N/A | N/A | 8,637 | 8,673 | |
| mean (sd) | 0.95 (0.29) | | 0.95 (0.28) | 0.92 (0.23) | N/A | N/A | 0.95 (0.29) | 0.92 (0.24) | 0.11 |
| median [IQR] | 0.90 [0.76, 1.07] | 0.89 [0.76, 1.04] | 0.91 [0.76, 1.06] | 0.89 [0.76, 1.05] | N/A | N/A | 0.90 (0.29) | 0.89 (0.24) | 0.04 |
| | | | | | | · | | , , | |
| Missing; n (%) | 9,675 (57.8%) | 9,421 (56.3%) | 21,693 (93.2%) | 21,911 (94.2%) | N/A | N/A | 31,368 (78.4%) | 31,332 (78.3%) | 0.00 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | |
| =<5000 included) | 6,063 | 6,278 | 1,600 | 1,341 | N/A | N/A | 7,663 | 7,619 | |
| mean (sd) | 44.91 (13.29) | 45.34 (13.17) | 44.01 (13.95) | 46.54 (108.97) | N/A | N/A | 44.72 (13.43) | 45.55 (47.25) | -0.02 |
| median [IQR] | 43.00 [36.00, 52.00] | 43.50 [36.28, 52.00] | 43.00 [36.00, 51.00] | 43.00 [35.00, 50.75] | N/A | N/A | 43.00 (13.43) | 43.41 (47.25) | -0.01 |
| Missing; n (%) | 10,677 (63.8%) | 10,462 (62.5%) | 21,665 (93.1%) | 21,924 (94.2%) | N/A | N/A | 32,342 (80.8%) | 32,386 (81.0%) | -0.01 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | |
| =<5000 included) | 6,127 | 6,357 | 1,464 | 1,218 | N/A | N/A | 7,591 | 7,575 | |
| mean (sd) | 85.82 (40.64) | 84.61 (39.33) | 89.35 (41.61) | 86.98 (40.52) | N/A | N/A | 86.50 (40.83) | 84.99 (39.53) | 0.04 |
| median [IQR] | 84.00 [62.00, 109.00] | 82.00 [61.00, 107.00] | 88.25 [65.00, 113.50] | 85.88 [63.00, 112.00] | N/A | N/A | 84.82 (40.83) | 82.62 (39.53) | 0.05 |
| Missing; n (%) | 10,613 (63.4%) | 10,383 (62.0%) | 21,801 (93.7%) | 22,047 (94.8%) | N/A | N/A | 32,414 (81.0%) | 32,430 (81.1%) | 0.00 |
| | 10,013 (03.4%) | 10,363 (02.0%) | 21,001 (33.770) | 22,047 (34.070) | N/A | IN/M | 32,414 (01.070) | 32,430 (01.170) | 0.00 |
| Lab result number-Total cholesterol (mg/dl) mean | 6.400 | C 400 | 4.507 | 4.244 | | h. /a | 7.787 | 7.747 | |
| (only =<5000 included) | 6,190 | 6,403 | 1,597 | 1,344 | N/A | N/A | * * | 7,747 | |
| mean (sd) | 174.42 (47.37) | 172.68 (46.78) | 175.05 (50.49) | 172.22 (55.71) | N/A | N/A | 174.55 (48.03) | 172.60 (48.45) | 0.04 |
| median [IQR] | 169.00 [143.00, 199.00] | | | | N/A | N/A | 169.41 (48.03) | 167.52 (48.45) | 0.04 |
| Missing; n (%) | 10,550 (63.0%) | 10,337 (61.8%) | 21,668 (93.1%) | 21,921 (94.2%) | N/A | N/A | 32,218 (80.5%) | 32,258 (80.6%) | 0.00 |

| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only =<5000 included) | 6,138 | 6,365 | 1,585 | 1,324 | N/A | N/A | 7,723 | 7,689 | |
| mean (sd) | 199.03 (170.61) | 197.06 (178.97) | 193.72 (167.75) | 195.36 (188.68) | N/A | N/A | 197.94 (170.04) | 196.77 (180.69) | 0.01 |
| median [IQR] | 159.00 [111.00, 231.00] | 157.33 [112.00, 226.00] | 155.00 [109.00, 223.75] | 160.00 [112.00, 227.00] | N/A | N/A | 158.18 (170.04) | 157.79 (180.69) | 0.00 |
| Missing; n (%) | 10,602 (63.3%) | 10,375 (62.0%) | 21,680 (93.2%) | 21,941 (94.3%) | N/A | N/A | 32,282 (80.7%) | 32,316 (80.8%) | 0.00 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | |
| included) | 4,465 | 4,725 | 1,110 | 856 | N/A | N/A | 5,575 | 5,581 | |
| mean (sd) | 13.82 (1.54) | 14.06 (1.56) | 10,214.28 (300,385.23) | 14,006.95 (342,165.79) | N/A | N/A | 2044.76 (134010.49) | 2160.25 (133961.62) | 0.00 |
| median [IQR] | 13.83 [12.80, 14.80] | 14.10 [13.00, 15.10] | 13.80 [12.80, 14.70] | 14.00 [12.90, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 12,275 (73.3%) | 12,015 (71.8%) | 22,155 (95.2%) | 22,409 (96.3%) | N/A | N/A | 34,430 (86.1%) | 34,424 (86.0%) | 0.00 |
| Lab result number- Serum sodium mean (only > 90 and < 190 included) | 6,917 | 7,194 | 1,610 | 1,327 | N/A | N/A | 8,527 | 8,521 | |
| mean (sd) | 139.22 (2.73) | 139.28 (2.62) | 138.81 (2.80) | 139.05 (2.41) | N/A | N/A | 139.14 (2.74) | 139.24 (2.59) | -0.04 |
| median [IQR] | 139.00 [137.67, 141.00] | 139.00 [138.00, 141.00] | 139.00 [137.00, 140.50] | 139.00 [138.00, 140.67] | N/A | N/A | 139.00 (2.74) | 139.00 (2.59) | 0.00 |
| Missing; n (%) | 9,823 (58.7%) | 9,546 (57.0%) | 21,655 (93.1%) | 21,938 (94.3%) | N/A | N/A | 31,478 (78.7%) | 31,484 (78.7%) | 0.00 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 6,438 | 6,794 | 1,399 | 1,117 | N/A | N/A | 7,837 | 7,911 | |
| mean (sd) | 4.29 (0.30) | 4.30 (0.30) | 4.19 (0.62) | 4.16 (0.70) | N/A | N/A | 4.27 (0.38) | 4.28 (0.38) | -0.03 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 4.30 [4.00, 4.50] | 4.30 [4.00, 4.50] | N/A | N/A | 4.30 (0.38) | 4.30 (0.38) | 0.00 |
| Missing; n (%) | 10,302 (61.5%) | 9,946 (59.4%) | 21,866 (94.0%) | 22,148 (95.2%) | N/A | N/A | 32,168 (80.4%) | 32,094 (80.2%) | 0.01 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | |
| (only 10-1000 included) | 6,905 | 7,185 | 1,588 | 1,309 | N/A | N/A | 8,493 | 8,494 | 2.05 |
| mean (sd) | 182.23 (74.88)<br>164.00 [130.45, 217.00] | 178.16 (69.58)<br>162.00 [130.00, 211.00] | 182.28 (74.67)<br>164.25 [131.00, 214.75] | 176.56 (63.34)<br>163.00 [132.00, 209.00] | N/A<br>N/A | N/A<br>N/A | 182.24 (74.85)<br>164.05 (74.85) | 177.91 (68.66) | 0.06<br>0.03 |
| median [IQR]<br>Missing; n (%) | 9,835 (58.8%) | 9,555 (57.1%) | 21,677 (93.2%) | 21,956 (94.4%) | N/A | N/A | 31,512 (78.8%) | 162.15 (68.66)<br>31,511 (78.8%) | 0.03 |
| Lab result number- Potassium mean (only 1-7 | 9,033 (30.0%) | 9,555 (57.1%) | 21,077 (93.2%) | 21,930 (94.4%) | N/A | IN/A | 31,312 (76.6%) | 31,311 (70.0%) | 0.00 |
| included) | 7,074 | 7,329 | 1,561 | 1,293 | N/A | N/A | 8,635 | 8,622 | |
| mean (sd) | 4.45 (0.40) | 4.44 (0.40) | 4.37 (0.43) | 4.36 (0.41) | N/A | N/A | 4.44 (0.41) | 4.43 (0.40) | 0.02 |
| median [IQR] | 4.40 [4.20, 4.70] | 4.40 [4.20, 4.70] | 4.35 [4.05, 4.60] | 4.35 [4.10, 4.60] | N/A | N/A | 4.39 (0.41) | 4.39 (0.40) | 0.00 |
| Missing; n (%) | 9,666 (57.7%) | 9,411 (56.2%) | 21,704 (93.3%) | 21,972 (94.4%) | N/A | N/A | 31,370 (78.4%) | 31,383 (78.4%) | 0.00 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.07 (1.27) | 2.07 (1.28) | 1.65 (0.99) | 1.65 (0.98) | 2.36 (1.50) | 2.37 (1.51) | 2.05 (1.29) | 2.05 (1.30) | 0.00 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.66 (1.29) | 1.66 (1.30) | 0.00 |
| Frailty Score: Qualitative Version 365 days as | | | | | | | | | |
| Categories, | 40.070 (65.60() | 40.027 (64.70) | 42 720 (54 70) | 42 400 (52 70/) | 42.474.(45.70() | 42.040 (45.40() | 25 000 (52 50) | 26 252 (52 20) | 0.00 |
| 0; n (%)<br>1 to 2; n (%) | 10,978 (65.6%)<br>4,527 (27.0%) | 10,837 (64.7%)<br>4,585 (27.4%) | 12,728 (54.7%)<br>8,508 (36.6%) | 12,498 (53.7%)<br>8,680 (37.3%) | 13,174 (45.7%)<br>10,071 (34.9%) | 13,018 (45.1%)<br>10,062 (34.9%) | 36,880 (53.6%)<br>23,106 (33.6%) | 36,353 (52.8%)<br>23,327 (33.9%) | 0.02<br>-0.01 |
| 1 to 2; n (%)<br>3 or more; n (%) | 1,235 (7.4%) | 1,318 (7.9%) | 2,029 (8.7%) | 2,087 (9.0%) | 5,600 (19.4%) | 5,765 (20.0%) | 8,864 (12.9%) | 9,170 (13.3%) | -0.01 |
| Frailty Score: Empirical Version 365 days as | 1,233 (7.470) | 1,310 (7.370) | 2,023 (8.776) | 2,087 (3.076) | 3,000 (13.470) | 3,703 (20.0%) | 8,804 (12.576) | 3,170 (13.370) | -0.01 |
| Categories, | | | | | | | | | |
| <0.12908; n (%) | 5,736 (34.3%) | 5,863 (35.0%) | 7,903 (34.0%) | 7,780 (33.4%) | 4,472 (15.5%) | 4,654 (16.1%) | 18,111 (26.3%) | 18,297 (26.6%) | -0.01 |
| 0.12908 - 0.1631167; n (%) | 6,275 (37.5%) | 6,241 (37.3%) | 9,182 (39.5%) | 9,210 (39.6%) | 9,121 (31.6%) | 8,892 (30.8%) | 24,578 (35.7%) | 24,343 (35.4%) | 0.01 |
| >= 0.1631167; n (%) | 4,729 (28.2%) | 4,636 (27.7%) | 6,180 (26.6%) | 6,275 (27.0%) | 15,252 (52.9%) | 15,299 (53.0%) | 26,161 (38.0%) | 26,210 (38.1%) | 0.00 |
| Non-Frailty; n (%) | 9,549 (57.0%) | 9,735 (58.2%) | 12,416 (53.4%) | 12,489 (53.7%) | 1,626 (5.6%) | 1,331 (4.6%) | 23,591 (34.3%) | 23,555 (34.2%) | 0.00 |
| Frailty Score (mean): Qualitative Version 365 days, | | | | | | | | | |
| mean (sd) | 0.64 (1.16) | 0.67 (1.20) | 0.81 (1.19) | 0.83 (1.20) | 1.29 (1.69) | 1.31 (1.69) | 0.97 (1.42) | 0.99 (1.43) | -0.01<br>0.00 |
| median [IQR] Frailty Score (mean): Empirical Version 365 days, | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.42 (1.42) | 0.42 (1.43) | 0.00 |
| mean (sd) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.04) | 0.14 (0.04) | 0.18 (0.05) | 0.18 (0.05) | 0.16 (0.04) | 0.16 (0.04) | 0.00 |
| median [IQR] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.17] | 0.14 (0.04) | 0.14 [0.12, 0.16] | 0.17 [0.14, 0.20] | 0.17 [0.14, 0.20] | 0.15 (0.04) | 0.15 (0.04) | 0.00 |
| Healthcare Utilization | 0.1 (0.12, 0.17) | 0.11 (0.12, 0.17) | 0.11 (0.12, 0.10) | 0.1 (0.11, 0.10) | 0.17 [0.11, 0.20] | 0.17 [0.11, 0.20] | 0.13 (0.0 1) | 0.15 (0.0 1) | 0.00 |
| Any hospitalization; n (%) | 422 (2.5%) | 395 (2.4%) | 472 (2.0%) | 486 (2.1%) | 1,130 (3.9%) | 1,123 (3.9%) | 2,024 (2.9%) | 2,004 (2.9%) | 0.00 |
| Any hospitalization within prior 30 days; n (%) | 73 (0.4%) | 63 (0.4%) | 66 (0.3%) | 77 (0.3%) | 166 (0.6%) | 186 (0.6%) | 305 (0.4%) | 326 (0.5%) | -0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 352 (2.1%) | 333 (2.0%) | 411 (1.8%) | 413 (1.8%) | 985 (3.4%) | 959 (3.3%) | 1,748 (2.5%) | 1,705 (2.5%) | 0.00 |
| Endocrinologist Visit; n (%) | 2,703 (16.1%) | 2,677 (16.0%) | 3,720 (16.0%) | 3,721 (16.0%) | 5,251 (18.2%) | 5,303 (18.4%) | 11,674 (17.0%) | 11,701 (17.0%) | 0.00 |
| Endocrinologist Visit (30 days prior); n (%) | 1,886 (11.3%) | 1,922 (11.5%) | 2,696 (11.6%) | 2,851 (12.3%) | 3,533 (12.2%) | 3,750 (13.0%) | 8,115 (11.8%) | 8,523 (12.4%) | -0.02 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 1,914 (11.4%) | 1,900 (11.4%) | 2,567 (11.0%) | 2,647 (11.4%) | 3,948 (13.7%) | 4,050 (14.0%) | 8,429 (12.2%) | 8,597 (12.5%) | -0.01 |
| Internal medicine/family medicine visits; n (%) | 12,196 (72.9%) | 11,920 (71.2%) | 20,638 (88.7%) | 20,362 (87.5%) | 24,256 (84.1%) | 23,791 (82.5%) | 57,090 (82.9%) | 56,073 (81.4%) | 0.04 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | |
| prior); n (%) | 8,667 (51.8%) | 8,658 (51.7%) | 15,681 (67.4%) | 15,619 (67.1%) | 17,442 (60.5%) | 17,316 (60.0%) | 41,790 (60.7%) | 41,593 (60.4%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 days prior); n (%) | 10,237 (61.2%) | 10,229 (61.1%) | 17,149 (73.7%) | 17,062 (73.3%) | 21,118 (73.2%) | 21,055 (73.0%) | 48,504 (70.4%) | 48,346 (70.2%) | 0.00 |
| Cardiologist visit; n (%) | 3,197 (19.1%) | 3,226 (19.3%) | 3,866 (16.6%) | 3,917 (16.8%) | 8,193 (28.4%) | 8,255 (28.6%) | 15,256 (22.2%) | 15,398 (22.4%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 990 (5.9%) | 1,022 (6.1%) | 1,192 (5.1%) | 1,175 (5.1%) | 2,541 (8.8%) | 2,563 (8.9%) | 4,723 (6.9%) | 4,760 (6.9%) | 0.00 |
| 5 · | () | ,- ,, | , - () | , - \/ | | | , | | |

| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| n (%) | 2,698 (16.1%) | 2,721 (16.3%) | 3,272 (14.1%) | 3,308 (14.2%) | 7,110 (24.6%) | 7,144 (24.8%) | 13,080 (19.0%) | 13,173 (19.1%) | 0.00 |
| Electrocardiogram ; n (%) | 3,814 (22.8%) | 3,833 (22.9%) | 5,351 (23.0%) | 5,482 (23.6%) | 8,209 (28.5%) | 8,398 (29.1%) | 17,374 (25.2%) | 17,713 (25.7%) | -0.01 |
| Use of glucose test strips; n (%) | 578 (3.5%) | 584 (3.5%) | 926 (4.0%) | 953 (4.1%) | 932 (3.2%) | 953 (3.3%) | 2,436 (3.5%) | 2,490 (3.6%) | -0.01 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Naive new user v8 Copy; n (%) | 1,847 (11.0%) | 1,869 (11.2%) | 1,991 (8.6%) | 2,032 (8.7%) | 1,870 (6.5%) | 1,975 (6.8%) | 5,708 (8.3%) | 5,876 (8.5%) | -0.01 |
| N antidiabetic drugs at index date Copy | | | | | | | | | |
| mean (sd) | 2.26 (0.88) | 2.26 (0.86) | 2.32 (0.90) | 2.32 (0.88) | 2.33 (0.89) | 2.35 (0.88) | 2.31 (0.89) | 2.32 (0.88) | -0.01 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 (0.89) | 2.00 (0.88) | 0.00 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 9.99 (4.51) | 9.95 (4.43) | 9.68 (4.21) | 9.71 (4.16) | 10.40 (4.33) | 10.45 (4.40) | 10.06 (4.33) | 10.08 (4.33) | 0.00 |
| median [IQR] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 10.00 [7.00, 13.00] | 10.00 [7.00, 13.00] | 9.42 (4.33) | 9.42 (4.33) | 0.00 |
| Number of Hospitalizations | 0.02 (0.24) | 0.02 (0.47) | 0.03 (0.45) | 0.02 (0.46) | 0.04 (0.22) | 0.04 (0.22) | 0.00 (0.04) | 0.03 (0.40) | 2.22 |
| mean (sd) | 0.03 (0.24) | 0.03 (0.17) | 0.02 (0.15) | 0.02 (0.16) | 0.04 (0.23) | 0.04 (0.23) | 0.03 (0.21) | 0.03 (0.19) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.21) | 0.00 (0.19) | 0.00 |
| Number of hospital days | 0.13/1.00 | 0.13 (0.07) | 0.00 (0.01) | 0.10 (0.00) | 0.22 (4.50) | 0.22 (4.07) | 0.45 (4.33) | 0.16 (1.40) | -0.01 |
| mean (sd) | 0.12 (1.00) | 0.12 (0.97)<br>0.00 [0.00, 0.00] | 0.09 (0.81)<br>0.00 [0.00, 0.00] | 0.10 (0.88) | 0.22 (1.56)<br>0.00 [0.00, 0.00] | 0.23 (1.87)<br>0.00 [0.00, 0.00] | 0.15 (1.22)<br>0.00 (1.22) | 0.16 (1.40)<br>0.00 (1.40) | 0.00 |
| median [IQR] Number of Emergency Department (ED) visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.22) | 0.00 (1.40) | 0.00 |
| mean (sd) | 0.21 (0.72) | 0.21 (0.76) | 0.04 (0.74) | 0.04 (0.55) | 0.31 (0.95) | 0.31 (1.07) | 0.19 (0.83) | 0.19 (0.85) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.83) | 0.00 (0.85) | 0.00 |
| Number of Office visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.03) | 0.00 (0.03) | 0.00 |
| mean (sd) | 4.29 (3.42) | 4.24 (3.06) | 4.23 (3.30) | 4.21 (3.07) | 5.08 (3.83) | 5.08 (3.60) | 4.60 (3.56) | 4.58 (3.30) | 0.01 |
| median [IQR] | 3.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 7.00] | 4.00 [3.00, 7.00] | 3.42 (3.56) | 3.42 (3.30) | 0.00 |
| Number of Endocrinologist visits | | | | | | | (, | () | |
| mean (sd) | 0.77 (2.73) | 0.85 (3.12) | 0.72 (2.61) | 0.87 (3.27) | 1.08 (4.08) | 1.22 (4.66) | 0.88 (3.33) | 1.01 (3.88) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.33) | 0.00 (3.88) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | |
| mean (sd) | 7.13 (11.56) | 7.03 (10.98) | 6.26 (7.11) | 6.46 (7.42) | 7.46 (10.23) | 7.75 (9.99) | 6.97 (9.67) | 7.14 (9.47) | -0.02 |
| median [IQR] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 8.00] | 4.00 [2.00, 9.00] | 4.00 [2.00, 10.00] | 5.00 [2.00, 10.00] | 4.00 (9.67) | 4.42 (9.47) | -0.04 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 0.78 (2.61) | 0.76 (2.44) | 0.61 (2.04) | 0.63 (2.14) | 1.33 (3.71) | 1.35 (3.65) | 0.95 (2.97) | 0.96 (2.93) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (2.97) | 0.00 (2.93) | 0.00 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd) | 0.36 (0.86) | 0.36 (0.86) | 0.35 (0.82) | 0.35 (0.83) | 0.50 (1.05) | 0.50 (1.07) | 0.42 (0.93) | 0.42 (0.94) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.93) | 0.00 (0.94) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 1.36 (0.89) | 1.35 (0.87) | 1.28 (0.88) | 1.28 (0.85) | 1.56 (0.90) | 1.56 (0.82) | 1.42 (0.89) | 1.41 (0.84) | 0.01 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.42 (0.89) | 1.42 (0.84) | 0.00 |
| Number of glucose tests ordered | 0.42/4.07) | 0.42 (4.74) | 0.20 (1.62) | 0.20 (4.02) | 0.47 (1.24) | 0.47/1.11 | 0.43 (4.50) | 0.42 (4.26) | 0.00 |
| mean (sd)<br>median [IQR] | 0.43 (1.87)<br>0.00 [0.00, 0.00] | 0.43 (1.71)<br>0.00 [0.00, 0.00] | 0.39 (1.63)<br>0.00 [0.00, 0.00] | 0.39 (1.03)<br>0.00 [0.00, 0.00] | 0.47 (1.34)<br>0.00 [0.00, 0.00] | 0.47 (1.11)<br>0.00 [0.00, 0.00] | 0.43 (1.58)<br>0.00 (1.58) | 0.43 (1.26)<br>0.00 (1.26) | 0.00 |
| Number of lipid tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.38) | 0.00 (1.26) | 0.00 |
| mean (sd) | 1.06 (0.96) | 1.06 (0.94) | 1.06 (1.29) | 1.06 (1.13) | 1.13 (0.88) | 1.13 (0.83) | 1.09 (1.05) | 1.09 (0.97) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (1.05) | 1.00 (0.97) | 0.00 |
| Number of creatinine tests ordered | 1.00 (0.00, 2.00) | 1.00 [0.00, 2.00] | 1.00 (0.00) 1.00) | 1.00 (0.00, 2.00) | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (1.03) | 1.00 (0.57) | 0.00 |
| mean (sd) | 0.03 (0.22) | 0.03 (0.20) | 0.03 (0.23) | 0.04 (0.24) | 0.07 (0.34) | 0.07 (0.32) | 0.05 (0.28) | 0.05 (0.27) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.28) | 0.00 (0.27) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.02 (0.16) | 0.02 (0.16) | 0.02 (0.18) | 0.02 (0.18) | 0.04 (0.28) | 0.04 (0.26) | 0.03 (0.22) | 0.03 (0.21) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.22) | 0.00 (0.21) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | |
| mean (sd) | 0.84 (1.19) | 0.85 (1.18) | 0.74 (1.11) | 0.74 (1.10) | 0.53 (0.73) | 0.54 (0.73) | 0.68 (0.99) | 0.68 (0.99) | 0.00 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.99) | 0.00 (0.99) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | |
| digit level Copy | | | | | | | | | |
| mean (sd) | 5.56 (5.86) | 5.43 (6.00) | 2.09 (3.20) | 2.05 (3.27) | 5.91 (6.84) | 5.82 (6.92) | 4.53 (5.60) | 4.45 (5.69) | 0.01 |
| median [IQR] | 5.00 [0.00, 8.00] | 5.00 [0.00, 8.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 4.00 [0.00, 9.00] | 4.00 [0.00, 9.00] | 2.89 (5.60) | 2.89 (5.69) | 0.00 |
| Use of this ride in (9/) | 2.040 (4.2.20/) | 2.060 (42.30/) | 2 702 (42 00/) | 2 727 /44 00/1 | 4 135 (14 30/) | 4 100 (1 4 30/) | 0.047 (43.00/) | 0 007 /43 00/1 | 0.00 |
| Use of thiazide; n (%) Use of beta blockers; n (%) | 2,040 (12.2%)<br>6,033 (36.0%) | 2,060 (12.3%)<br>6,038 (36.1%) | 2,782 (12.0%)<br>8,159 (35.1%) | 2,737 (11.8%)<br>8,198 (35.2%) | 4,125 (14.3%)<br>13,867 (48.1%) | 4,100 (14.2%)<br>13,913 (48.2%) | 8,947 (13.0%)<br>28,059 (40.8%) | 8,897 (12.9%)<br>28,149 (40.9%) | 0.00 |
| Use of calcium channel blockers; n (%) | 4,836 (28.9%) | 4,820 (28.8%) | 6,641 (28.5%) | 6,697 (28.8%) | 9,762 (33.8%) | 9,796 (34.0%) | 21,239 (30.8%) | 21,313 (31.0%) | 0.00 |
| ose or earciam channel brockers, ii (/o) | 7,030 (20.370) | 7,020 (20.070) | 0,071 (20.370) | 0,037 (20.070) | 3,102 (33.070) | 5,750 (34.070) | 21,233 (30.070) | 21,313 (31.070) | 0.00 |